CLINICAL TRIAL: NCT02709486
Title: A PHASE 3 RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED, MULTICENTER STUDY OF THE ANALGESIC EFFICACY AND SAFETY OF THE SUBCUTANEOUS ADMINISTRATION OF TANEZUMAB IN SUBJECTS WITH OSTEOARTHRITIS OF THE HIP OR KNEE
Brief Title: Study of the Analgesic Efficacy and Safety of Subcutaneous Tanezumab in Subjects With Osteoarthritis of the Hip or Knee.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A4091057; 2013-004508-21 (EudraCT Number); OA 6-MONTH EU STUDY (Other: Alias Study Number)
Record Dates: First submitted 2016-02-26; First posted 2016-03-16 (Estimated); Results first posted 2019-06-26 (Actual); Last update posted 2019-06-26 (Actual); Status verified 2019-06

CONDITIONS: Osteoarthritis, Hip; Osteoarthritis, Knee
Keywords: Osteoarthritis, pain, tanezumab.
MeSH Terms: conditions — Osteoarthritis, Hip; Osteoarthritis, Knee; Osteoarthritis; Pain | interventions — tanezumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Low dose (Experimental): Investigational product
  Interventions: Drug: Tanezumab
- High dose (Experimental): Investigational product
  Interventions: Drug: Tanezumab
- Placebo (Placebo Comparator): Investigational product
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tanezumab — 2.5 mg
  Arms: Low dose
Drug: Tanezumab — 5 mg
  Arms: High dose
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Tanezumab is a monoclonal antibody that binds to and inhibits the actions of nerve growth factor (NGF). The Nerve Growth Factor Inhibitor (NGFI) class may offer an important breakthrough in the treatment of chronic pain and is under clinical investigation for the treatment of pain associated with osteoarthritis or other chronic pain conditions.

The primary objective of this study is to demonstrate superior efficacy of tanezumab 5 mg and 2.5 mg administered subcutaneously (SC) every 8 weeks versus placebo at Week 24 in subjects with osteoarthritis of the knee or hip. The 2.5 mg dose was shown to provide efficacy benefits with a favorable safety profile when administered intravenously in previous Phase 3 clinical trials. The 5 mg dose is expected to provide added efficacy benefit over the 2.5 mg dose based on data from previous studies.

DETAILED DESCRIPTION:
This is a randomized, double blind, placebo controlled, parallel group multicenter Phase 3 study of the efficacy and safety of tanezumab when administered by SC injection for 24 weeks compared to placebo in subjects with osteoarthritis of the knee or hip. A total of approximately 810 subjects will be randomized to 1 of 3 treatment groups in a 1:1:1 ratio (ie, 270/group). The randomization will be stratified by index joint (hip or knee), and most severe Kellgren-Lawrence grade (of any knee or hip joint) at study entry (grade 2, 3 or 4). Subjects will receive up to three SC doses of one of the following treatments at an 8-week interval between each injection:

1. tanezumab 2.5 mg;
2. tanezumab 5 mg;
3. Placebo to match tanezumab. The study is designed with a total (post-randomization) duration of 48 weeks and will consist of three periods: Screening (up to 37 days), Double-blind Treatment (24 weeks) and Safety Follow-up (24 weeks). The Screening Period (beginning up to 37 days prior to Randomization) includes a Washout Period (lasting a minimum of 2 days for all prohibited pain medications), if required, and an Initial Pain Assessment Period (the 7 days prior to Randomization/Baseline).

Week 24 is the landmark analysis in this study. Subjects who do not complete the Double-blind Treatment period will enter and complete the 24-week Early-termination follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of osteoarthritis of the index hip or knee based on American College of Rheumatology criteria with Kellgren Lawrence x-ray Grade of at least 2 as diagnosed by the Central Reader
* A history of insufficient pain relief from acetaminophen along with a history of insufficient pain relief from, inability to tolerate or contraindication to taking NSAIDs, and tramadol or opioid treatments.
* WOMAC Pain subscale score of at least 5 in the index hip or knee at Screening.
* Be willing to discontinue all non study pain medications for osteoarthritis and not use prohibited pain medications throughout the duration of the study.
* Female subjects of childbearing potential must agree to comply with protocol specified contraceptive requirements.

Exclusion Criteria:

* Subjects exceeding protocol defined BMI or body weight limits.
* History of other diseases specified in the protocol (e.g. inflammatory joint diseases, crystalline diseases such as gout or pseudogout) that may involve the index joint and that could interfere with efficacy assessments.
* Radiographic evidence of protocol specified bone or joint conditions in any screening radiograph as determined by the central radiology reviewer.
* A history of osteonecrosis or osteoporotic fracture.
* History of significant trauma or surgery to a knee, hip or shoulder within the previous year.
* Planned surgical procedure during the duration of the study.
* Presence of conditions (e.g. fibromyalgia, radiculopathy) associated with moderate to severe pain that may confound assessments or self evaluation of osteoarthritis pain.
* Signs or symptoms of carpal tunnel syndrome in the year prior to Screening.
* Considered unfit for surgery based upon American Society of Anesthesiologists physical classification system for surgery grading, or subjects who would not be willing to undergo joint replacement surgery if required.
* History of intolerance or hypersensitivity to acetaminophen or any of its excipients or existence of a medical condition or use of concomitant medication for which the use of acetaminophen is contraindicated.
* Use of prohibited medications without the appropriate washout period prior to Screening or Initial Pain Assessment Period.
* History of cancer within 5 years of Screening, except for cutaneous basal cell or squamous cell cancer resolved by excision.
* Subjects with signs and symptoms of clinically significant cardiac disease as described in the protocol.
* Diagnosis of a transient ischemic attack in the 6 months prior to Screening, diagnosis of stroke with residual deficits that would preclude completion of required study activities.
* History, diagnosis, or signs and symptoms of clinically significant neurological disease such as but not limited to peripheral or autonomic neuropathy.
* History, diagnosis, signs or symptoms of any clinically significant psychiatric disorder.
* History of known alcohol, analgesic or drug abuse within 2 years of Screening.
* Previous exposure to exogenous NGF or to an anti-NGF antibody.
* History of allergic or anaphylactic reaction to a therapeutic or diagnostic monoclonal antibody or IgG fusion protein.
* Poorly controlled hypertension as defined in the protocol or taking an antihypertensive that has not been stable for at least 1 month prior to Screening.
* Evidence of protocol defined orthostatic hypotension at Screening.
* Disqualifying score on the Survey of Autonomic Symptoms questionnaire at Screening.
* Screening AST, ALT, serum creatinine or HbA1c values that exceed protocol defined limits.
* Presence of drugs of abuse in screening urine toxicology panel.
* Positive hepatitis B, hepatitis C or HIV test results indicative of current infection.
* Participation in other investigational drug studies within protocol defined time limits.
* Pregnant, breastfeeding or female subjects of childbearing potential who are unwilling or unable to follow protocol required contraceptive requirements.
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that in the judgment of the investigator, would make the subject inappropriate for entry into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 849 (Actual)
Dates: Start 2016-03-02 (Actual); Primary Completion 2018-06-08 (Actual); Study Completion 2018-11-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (147):
- Austria (2):
  - Nuhr Medical Center, Senftenberg
  - Rheuma Zentrum Favoriten, Vienna
- Bulgaria (16):
  - Medical Center BLAGOEVGRAD 2009, EOOD, Blagoevgrad
  - DCC St. Pantaleimon OOD, Pleven
  - Medical Center " Health for all" EOOD, Plovdiv
  - UMHAT Kaspela, Plovdiv
  - "Medical Center Teodora" EOOD, Rousse
  - Multiprofile Hospital for Active Treatment-Silistra AD, Silistra
  - "Medical Center- Smolyan" OOD, Smolyan
  - NMTH 'Tsar Boris III". Clinic of Internal Diseases, Sofia
  - Multiprofile hospital for active treatment - "Lyulin" EAD, Sofia
  - Diagnostic Consultative Center XIV- Sofia EOOD, Sofia
  - Medical Center-Avicena EOOD, Sofia
  - UMHAT Sveti Ivan Rilski - EAD, Sofia
  - UMHAT "Sofiamed" OOD, Block 2, Sofia
  - "Medical Center - Dr. Hayvazov" EOOD, Sofia
  - UMHAT "Prof. Dr. Stoyan Kirkovich" AD, Stara Zagora
  - Multiprofile Hospital for active treatment "SVETA PETKA" AD, Vidin
- Finland (2):
  - Dextra Oy/Pihlajalinna Ite Kuopio, Kuopio
  - Oulu Deaconess Institute, Oulu
- France (7):
  - Hôpital Edouard Herriot, Lyon
  - Unite Clinique Therapeutique des Maladies Osteoarticulaires, Montpellier
  - CHR Orleans La Source, Orléans
  - Hopital Lariboisiere, Paris
  - Hopital Saint-Antoine, Paris
  - Hôpital Cochin, Paris
  - Hopital Cochin, Paris
- Germany (6):
  - Praxis Dr. Kronung, Offenbach, Hesse
  - Rheumapraxis, Aachen
  - Rheumazentrum Prof. Dr. med Gunther Neeck, Bad Doberan
  - Kerckhoff Klinik GmbH, Bad Nauheim
  - Charite Universitaetsmedizin Berlin, Berlin
  - CIRI GmbH, Frankfurt am Main
- Hungary (6):
  - Bekes Megyei Központi Korhaz Dr Rethy Pal Tagkorhaz, Reumatologia Szakrendeles, Békéscsaba
  - Clinexpert Egeszsegugyi Szolgaltato es Kereskedelmi Kft., Budapest
  - Obudai Egeszsegugyi Centrum Kft, Budapest
  - Qualiclinic Kft., Budapest
  - Jutrix Kft, Kecskemét
  - Tolna Megyei Balassa Janos Korhaz, Ortopediai osztaly, Szekszárd
- Italy (13):
  - Farmacia AOUC Settore Sperimentazione Farmaci, Florence, FI
  - Istituto Clinico Humanitas Unita Operativa di Medicina Generale e Reumatologia -, Rozzano, Milan
  - Azienda Ospedaliera-Universitaria S.Orsola-Malpighi, Bologna
  - Farmacia Clinica Puggioli, Bologna
  - AZ OSPEDALIERO - UNIVERSITARIA CAREGGI-SOD Reumatologia - Dip. Medicina Sperimentale e Clinica, Florence
  - Dipartmento di diagnostica per immagini, Florence
  - AOU Maggiore della Carita di Novara - S.C. Medicina Fisica e Riabilitativa, Novara
  - Dipartimento Immagini Radiologia, Novara
  - Farmacia Ospedaliera, Novara
  - Azienda Ospedaliero-Universitaria E Policlinico Umberto I, Rome
  - Azienda Ospedaliera Universitaria Senese - UOC Reumatologia,, Siena
  - U.O.C. Farmacia - Gestione medicinali per la sperimentazione clinica, Siena
  - Ospedale Civile Maggiore Borgo Trento, Verona
- Japan (30):
  - Sato Orthopedic Clinic, Ichikawa, Chiba
  - Kamagaya General Hospital, Kamagaya, Chiba
  - Fukuoka Mirai Hospital, Higashi-ku,Fukuoka, Fukuoka
  - Shinkokura Hospital, Kitakyushu, Fukuoka
  - Obase Hospital, Miyako-gun, Fukuoka
  - Takagi Hospital, Ōkawa, Fukuoka
  - Himeno Hospital, Yamegun, Fukuoka
  - Takahashi Orthopedics Clinic, Chitose, Hokkaido
  - Hakodate Central General Hospital, Hakodate, Hokkaido
  - Hakodate Ohmura Orthopedic Hospital, Hakodate, Hokkaido
  - Obihiro Orthopaedic Hospital, Obihiro, Hokkaido
  - Okubo Hospital, Akashi, Hyōgo
  - Kobe Kaisei Hospital, Kobe, Hyōgo
  - Kobe Konan Yamate clinic, Kobe, Hyōgo
  - National Hospital Organization Sagamihara National Hospital, Sagamihara, Kanagawa
  - Medical Corporation Association Sankikai, Yokohama Shinmidori General Hospital, Yokohama, Kanagawa
  - Marunouchi Hospital, Matsumoto, Nagano
  - National Hospital Organization Nagasaki Medical Center, Ōmura, Nagasaki
  - Sobajima Clinic/Orthopedics, Higashiosaka, Osaka
  - National Hospital Organization Osaka Minami Medical Center, Kawachi-Nagano, Osaka
  - Hamamatsu Medical Center, Hamamatsu, Shizuoka
  - National Hospital Organization Utsunomiya national Hospital, Utsunomiya, Tochigi
  - Sonodakai Joint Replacement Center Hospital, Adachi-ku, Tokyo
  - Kitasato University Kitasato Institute Hospital, Minato-ku, Tokyo
  - Ohimachi Orthopaedic Clinic, Shinagawa-ku, Tokyo
  - Akita City Hospital, Akita
  - Kyushu Central Hospital, Fukuoka
  - Hiroshima Clinic, Hiroshima
  - Jujo Takeda Rehabilitation Hospital, Kyoto
  - Nagayoshi General Hospital, Osaka
- Poland (9):
  - NZOZ OSTEO-MEDIC s.c. A. Racewicz, J. Supronik, Bialystok
  - ClinicMed Daniluk, Nowak Społka Jawna, Bialystok
  - Centrum Kliniczno - Badawcze J. Brzezicki, B. Gornikiewicz - Brzezicka Lekarze Spolka Partnerska, Elblag
  - Centrum Medyczne Pratia Gdynia, Gdynia
  - Centrum Medyczne Pratia Krakow, Krakow
  - Malopolskie Centrum Medyczne S.C, Krakow
  - Centrum Terapii Wspolczesnej J.M Jasnorzewska, Lodz
  - MTZ Clinical Research Sp. z o.o., Warsaw
  - REUMATIKA - Centrum Reumatologii NZOZ, Warsaw
- Portugal (3):
  - Hospital Conde de Bertiandos, Ponte de Lima, Viana do Castelo District
  - Centro Hospitalar Lisboa Ocidental, E.P.E., Hospital Egas Moniz, Lisbon
  - Hospital Egas Moniz, Lisbon
- Romania (6):
  - SC Duo Medical SRL, Bucharest, Sector 1
  - Centrul Medical SANA S.R.L., Bucharest, Sector 1
  - Spitalul Judetean de Urgenta Bacau, Bacau
  - Spitalul Clinic "Sf. Maria", Bucharest
  - Spitalul Clinic Judetean de Urgenta Sf. Apostol Andrei Constanta, Constanța
  - Spitalul Clinic Judetean de Urgenta Sibiu, Sibiu
- Slovakia (8):
  - AB-BA ambulancia s.r.o., Bratislava
  - ROMJAN s.r.o., Bratislava
  - Kompan, s.r.o, Dolny Kubín
  - ALGMED s.r.o., Košice
  - Reum. hapi s.r.o., Nové Mesto nad Váhom
  - Medipa s.r.o., Piešťany
  - MUDr. Viliam Cibik, PhD, s.r.o., Pruské
  - Reumex s.r.o, Rimavská Sobota
- Spain (21):
  - Hospital La Esperanza, Santiago de Compostela, A Coruna
  - Corporacio Sanitaria Parc Tauli de Sabadell, Sabadell, Barcelona
  - Corporació Sanitaria Parc Taulí de Sabadell, Sabadell, Barcelona
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - Hospital Universitario de Getafe, Getafe, Madrid
  - Complejo Hospital Universitario A Coruna (CHUAC), A Coruña
  - Hospital La Esperanza, A Coruña
  - Instituto de Ciencias Medicas, Alicante
  - Instituto de Ciencias Médicas, Alicante
  - Hospital del Mar, Barcelona
  - Hospital CIMA Sanitas, Barcelona
  - Hospital Universitario Reina Sofia., Córdoba
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital General Universitario de Guadalajara, Guadalajara
  - Hospital Universitario La Princesa Farmacia - Ensayos Clinicos, Madrid
  - Hospital Universitario La Princesa, Madrid
  - Hospital Universitario La Paz Servicio de Farmacia, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Regional Universitario de Malaga. Farmacia del Hospital Civil, Málaga
  - Hospital Regional Universitario de Malaga, Málaga
  - Hospital Infanta Luisa, Seville
- Sweden (8):
  - Ladulaas Kliniska Studier, Borås
  - CTC (Clinical Trial Center), Sahlgrenska University Hospital, Gothenburg
  - ProbarE i Lund AB, Lund
  - PharmaSite, Malmo
  - Avdelningen for kliniska provningar, S-huset, Örebro
  - ProbarE, Stockholm
  - Karolinska Trial Alliance, Fas 1, Stockholm
  - Karolinska Trial Alliance, KTA., Stockholm
- United Kingdom (10):
  - The Alverton Practice, Penzance, Cornwall
  - Brannel Surgery, St Austell, Cornwall
  - Knowle House Surgery, Plymouth, Devon
  - Western General Hospital, Edinburgh, Midlothian
  - Clinical Trials, Bradford on Avon Health Centre, Bradford-on-Avon
  - Health Centre, Bradford on Avon & Melksham Health Partnership, Bradford-on-Avon
  - Oxford University Hospitals NHS Foundation Trust, Headington, Oxford
  - St George's University Hospitals NHS Foundation Trust, London
  - Northumbria Healthcare NHS Foundation Trust, North Shields
  - Nuffield Department of Orthopaedics, Oxford

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Schnitzer TJ, Conaghan PG, Berenbaum F, Abraham L, Cappelleri JC, Bushmakin AG, Viktrup L, Yang R, Brown MT. Effect size varies based on calculation method and may affect interpretation of treatment effect: an illustration using randomised clinical trials in osteoarthritis. Adv Rheumatol. 2024 Apr 22;64(1):31. doi: 10.1186/s42358-024-00358-y. PMID 38650049
- [Derived] Guermazi A, Roemer FW, Kompel AJ, Diaz LE, Crema MD, Brown MT, Hickman A, Pixton GC, Viktrup L, Fountaine RJ, Burr A, Sherlock SP, West CR. Inter-Reader Consistency and Exclusionary Findings During Radiographic Screening for Phase 3 Trials of Tanezumab in Patients With Osteoarthritis. Osteoarthr Imaging. 2022 Sep-Dec;2(3-4):100082. doi: 10.1016/j.ostima.2022.100082. Epub 2022 Nov 15. PMID 38343426
- [Derived] Carrino JA, McAlindon TE, Schnitzer TJ, Guermazi A, Hochberg MC, Conaghan PG, Brown MT, Burr A, Fountaine RJ, Pixton GC, Viktrup L, Verburg KM, West CR. Characterization of adverse joint outcomes in patients with osteoarthritis treated with subcutaneous tanezumab. Osteoarthritis Cartilage. 2023 Dec;31(12):1612-1626. doi: 10.1016/j.joca.2023.08.010. Epub 2023 Aug 29. PMID 37652258
- [Derived] Shoji S, Suzuki A, Nouri P, Cai CH, Gaitonde P, Marshall S. Prediction of relative change in free nerve growth factor following subcutaneous administration of tanezumab, a novel monoclonal antibody to nerve growth factor. CPT Pharmacometrics Syst Pharmacol. 2023 Sep;12(9):1358-1370. doi: 10.1002/psp4.13015. Epub 2023 Jul 31. PMID 37470295
- [Derived] Brown MT, Cornblath DR, Koltzenburg M, Gorson KC, Hickman A, Pixton GC, Gaitonde P, Viktrup L, West CR. Peripheral Nerve Safety of Nerve Growth Factor Inhibition by Tanezumab: Pooled Analyses of Phase III Clinical Studies in Over 5000 Patients with Osteoarthritis. Clin Drug Investig. 2023 Jul;43(7):551-563. doi: 10.1007/s40261-023-01286-3. Epub 2023 Jul 18. PMID 37460782
- [Derived] Colloca L, Dworkin RH, Farrar JT, Tive L, Yang J, Viktrup L, Dasic G, West CR, Whalen E, Brown MT, Gilbert SA, Verburg KM. Predicting Treatment Responses in Patients With Osteoarthritis: Results From Two Phase III Tanezumab Randomized Clinical Trials. Clin Pharmacol Ther. 2023 Apr;113(4):878-886. doi: 10.1002/cpt.2842. Epub 2023 Jan 31. PMID 36621827
- [Derived] Hunter DJ, Schnitzer TJ, Hall J, Semel D, Davignon I, Cappelleri JC, Bushmakin AG, Abraham L. Time to first and sustained improvement in WOMAC domains among patients with osteoarthritis receiving tanezumab. Osteoarthr Cartil Open. 2022 Jul 2;4(3):100294. doi: 10.1016/j.ocarto.2022.100294. eCollection 2022 Sep. PMID 36474952
- [Derived] Atkinson J, Edwards RA, Bonfanti G, Barroso J, Schnitzer TJ. A Two-Step, Trajectory-Focused, Analytics Approach to Attempt Prediction of Analgesic Response in Patients with Moderate-to-Severe Osteoarthritis. Adv Ther. 2023 Jan;40(1):252-264. doi: 10.1007/s12325-022-02336-6. Epub 2022 Oct 27. PMID 36301512
- [Derived] Mease P, Kuritzky L, Wright WL, Mallick-Searle T, Fountaine R, Yang R, Sadrarhami M, Faison W, Johnston E, Viktrup L. Efficacy and safety of tanezumab, NSAIDs, and placebo in patients with moderate to severe hip or knee osteoarthritis and a history of depression, anxiety, or insomnia: post-hoc analysis of phase 3 trials. Curr Med Res Opin. 2022 Nov;38(11):1909-1922. doi: 10.1080/03007995.2022.2113689. Epub 2022 Aug 28. PMID 35980115
- [Derived] Schnitzer TJ, Bonfanti G, Atkinson J, Donevan S, Viktrup L, Barroso J, Whalen E, Edwards RA. Characterizing 16-Week Responder Profiles Using Group-Based Trajectory Modeling in Over 4300 Clinical Trial Participants Receiving Pharmaceutical Treatment for Moderate to Severe Osteoarthritis. Adv Ther. 2022 Oct;39(10):4742-4756. doi: 10.1007/s12325-022-02290-3. Epub 2022 Aug 12. PMID 35960482
- [Derived] Conaghan PG, Dworkin RH, Schnitzer TJ, Berenbaum F, Bushmakin AG, Cappelleri JC, Viktrup L, Abraham L. WOMAC Meaningful Within-patient Change: Results From 3 Studies of Tanezumab in Patients With Moderate-to-severe Osteoarthritis of the Hip or Knee. J Rheumatol. 2022 Jun;49(6):615-621. doi: 10.3899/jrheum.210543. Epub 2022 Mar 1. PMID 35232805
- [Derived] Conaghan PG, Abraham L, Viktrup L, Cislo P. Impact of tanezumab on health status, non-work activities and work productivity in adults with moderate-to-severe osteoarthritis. BMC Musculoskelet Disord. 2022 Feb 1;23(1):106. doi: 10.1186/s12891-022-05029-x. PMID 35105318
- [Derived] Berenbaum F, Schnitzer T, Kivitz A, Viktrup L, Johnston E, Yang R, Whalen E, Tive L, Semel D. Gender, age, disease severity, body mass index and diabetes may not affect response to subcutaneous tanezumab in patients with osteoarthritis after 16 weeks of treatment. A subgroup analysis of placebo-controlled trials. Int J Clin Pract. 2021 Dec;75(12):e14975. doi: 10.1111/ijcp.14975. Epub 2021 Oct 21. PMID 34626502
- [Derived] Berenbaum F, Schnitzer TJ, Kivitz AJ, Viktrup L, Hickman A, Pixton G, Brown MT, Davignon I, West CR. General Safety and Tolerability of Subcutaneous Tanezumab for Osteoarthritis: A Pooled Analysis of Three Randomized, Placebo-Controlled Trials. Arthritis Care Res (Hoboken). 2022 Jun;74(6):918-928. doi: 10.1002/acr.24637. Epub 2022 Mar 25. PMID 33973384
- [Derived] Berenbaum F, Langford R, Perrot S, Miki K, Blanco FJ, Yamabe T, Isogawa N, Junor R, Carey W, Viktrup L, West CR, Brown MT, Verburg KM. Subcutaneous tanezumab for osteoarthritis: Is the early improvement in pain and function meaningful and sustained? Eur J Pain. 2021 Aug;25(7):1525-1539. doi: 10.1002/ejp.1764. Epub 2021 May 3. PMID 33728717
- [Derived] Berenbaum F, Blanco FJ, Guermazi A, Miki K, Yamabe T, Viktrup L, Junor R, Carey W, Brown MT, West CR, Verburg KM. Subcutaneous tanezumab for osteoarthritis of the hip or knee: efficacy and safety results from a 24-week randomised phase III study with a 24-week follow-up period. Ann Rheum Dis. 2020 Jun;79(6):800-810. doi: 10.1136/annrheumdis-2019-216296. Epub 2020 Mar 31. PMID 32234715
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4091057
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4091057&StudyName=A+Phase+3+Randomized%2C+Double-blind%2C+Placebo-controlled%2C+Multicenter+Study+Of+The+Analgesic+Efficacy+And+Safety+Of+The+Subcutaneous+Administration+Of+Tanezumab+In+Subjects+With+Osteoarthritis+Of+The+Hip+Or+Knee

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo matched to tanezumab (RN624 or PF-04383119) injection administered subcutaneously on Day 1 (Baseline), Week 8 and Week 16.
- Tanezumab 2.5 mg: Tanezumab (RN624 or PF-04383119) 2.5 mg injection administered subcutaneously on Day 1 (Baseline), Week 8 and Week 16.
- Tanezumab 5 mg: Tanezumab (RN624 or PF-04383119) 5 mg injection administered subcutaneously on Day 1 (Baseline), Week 8 and Week 16.
Period: Overall Study
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg
Started | 282 | 283 | 284
Completed | 238 | 249 | 239
Not Completed | 44 | 34 | 45
Not completed — Adverse Event | 2 | 5 | 3
Not completed — Death | 0 | 0 | 2
Not completed — Insufficient clinical response | 7 | 3 | 3
Not completed — Lost to Follow-up | 3 | 2 | 2
Not completed — Other | 0 | 2 | 3
Not completed — Withdrawal by Subject | 32 | 22 | 32

BASELINE CHARACTERISTICS:
Population: The safety population was defined as all participants treated with tanezumab or placebo subcutaneously.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg | Total
Number analyzed (Participants) | 282 | 283 | 284 | 849
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.24 (9.58) | 65.17 (8.39) | 65.23 (10.16) | 64.88 (9.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 196 | 198 | 193 | 587
  Male | 86 | 85 | 91 | 262
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19 | 19 | 10 | 48
  Not Hispanic or Latino | 263 | 264 | 274 | 801
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 247 | 245 | 248 | 740
  Black or African American | 0 | 0 | 0 | 0
  Asian | 34 | 38 | 34 | 106
  Other | 1 | 0 | 2 | 3
  Unknown | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale at Week 24
Description: WOMAC: Self-administered, disease-specific questionnaire which assesses clinically important, participant-relevant symptoms for pain, stiffness and physical function in participants with osteoarthritis (OA). The WOMAC pain subscale is a 5-item questionnaire used to assess the amount of pain experienced due to OA of index joint (knee or hip) during past 48 hours. It was calculated as the mean of scores from 5 individual questions scored on a numerical rating scale (NRS). Scores for each question and WOMAC Pain subscale score on NRS ranged from 0 (no pain) to 10 (extreme pain), where higher scores indicated higher pain.
Time Frame: Baseline, Week 24
Population: The intent to treat (ITT) population included all randomized participants who received at least one dose of subcutaneous (SC) study medication (either tanezumab or placebo).
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg
Number analyzed (Participants) | 282 | 283 | 284
units on a scale | -2.24 (0.17) | -2.70 (0.17) | -2.85 (0.17)
Statistical Analysis 1: Comparison: Placebo vs Tanezumab 2.5 mg; Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. Analysis of covariance (ANCOVA) model for imputed datasets included treatment, randomization stratification variables (index joint and highest Kellgren-Lawrence grade) as fixed effects, baseline WOMAC pain subscale and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority — Step-down testing procedure within each of the primary outcome measures was applied to maintain Type I error. Tanezumab 5 mg versus placebo was tested first and if found significant, then the testing was continued for Tanezumab 2.5 mg versus placebo. Tanezumab treatment group was declared as superior to placebo if the corresponding treatment contrast was significant over all 3 primary outcome measures; p = 0.0088, ANCOVA — Threshold for significance at 0.05 level; Least Square Mean Difference = -0.46, 95% CI 2-sided [-0.81 to -0.12], Standard Error of Mean 0.18
Statistical Analysis 2: Comparison: Placebo vs Tanezumab 5 mg; Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment, randomization stratification variables (index joint and highest Kellgren-Lawrence grade) as fixed effects, baseline WOMAC pain subscale and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority — A step-down testing procedure within each of the primary outcome measures was applied to maintain Type I error. Tanezumab 5 mg versus placebo was tested first and if found significant, then the testing was continued for Tanezumab 2.5 mg versus placebo. A tanezumab treatment group was declared as superior to placebo if the corresponding treatment contrast was significant over all 3 primary outcome measures; p = 0.0006, ANCOVA — Threshold for significance at 0.05 level; Least Square Mean Difference = -0.62, 95% CI 2-sided [-0.97 to -0.26], Standard Error of Mean 0.18

2. Primary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Physical Function Subscale at Week 24
Description: WOMAC: Self-administered, disease-specific questionnaire which assesses clinically important, participant-relevant symptoms for pain, stiffness and physical function in participants with OA. Physical function refers to participant's ability to move around and perform usual activities of daily living. The WOMAC physical function subscale is a 17-item questionnaire used to assess the degree of difficulty experienced due to OA in index joint (knee or hip) during past 48 hours. It was calculated as mean of the scores from 17 individual questions scored on a NRS. Scores for each question and WOMAC physical function subscale score on NRS ranged from 0 (no difficulty) to 10 (extreme difficulty), where higher scores indicated extreme difficulty/worse physical function.
Time Frame: Baseline, Week 24
Population: The intent to treat population included all randomized participants who received at least one dose of subcutaneous study medication (either tanezumab or placebo).
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg
Number analyzed (Participants) | 282 | 283 | 284
units on a scale | -2.11 (0.17) | -2.70 (0.17) | -2.82 (0.17)
Statistical Analysis 1: Comparison: Placebo vs Tanezumab 2.5 mg; Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment, randomization stratification variables (index joint and highest Kellgren-Lawrence grade) as fixed effects, baseline WOMAC physical function subscale and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.0008, ANCOVA — Threshold for significance at 0.05 level; Least Square Mean Difference = -0.59, 95% CI 2-sided [-0.93 to -0.24], Standard Error of Mean 0.18
Statistical Analysis 2: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < .0001, ANCOVA — Threshold for significance at 0.05 level; Least Square Mean Difference = -0.71, 95% CI 2-sided [-1.05 to -0.36], Standard Error of Mean 0.17

3. Primary Outcome: Change From Baseline in the Patient's Global Assessment (PGA) of Osteoarthritis at Week 24
Description: PGA of OA was assessed by asking a question from participants: "Considering all the ways your osteoarthritis in your knee or hip (index joint) affects you, how are you doing today?" Participants responded on a scale ranging from 1-5, where 1=very good (no symptom and no limitation of normal activities), 2= good (mild symptoms and no limitation of normal activities), 3= fair (moderate symptoms and limitation of some normal activities), 4= poor (severe symptoms and inability to carry out most normal activities), and 5= very poor (very severe symptoms and inability to carry out all normal activities). Higher scores indicated worsening of condition.
Time Frame: Baseline, Week 24
Population: The intent to treat population was defined as all randomized participants who received at least one dose of subcutaneous study medication (either tanezumab or placebo).
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg
Number analyzed (Participants) | 282 | 283 | 284
units on a scale | -0.72 (0.06) | -0.82 (0.06) | -0.90 (0.06)
Statistical Analysis 1: Comparison: Placebo vs Tanezumab 2.5 mg; Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment, randomization stratification variables (index joint and highest Kellgren-Lawrence grade) as fixed effects, baseline PGA of osteoarthritis and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p = 0.1092, ANCOVA — Threshold for significance at 0.05 level; Least Square Mean Difference = -0.11, 95% CI 2-sided [-0.24 to 0.02], Standard Error of Mean 0.07
Statistical Analysis 2: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p = 0.0051, ANCOVA — Threshold for significance at 0.05 level; Least Square Mean Difference = -0.19, 95% CI 2-sided [-0.32 to -0.06], Standard Error of Mean 0.07

4. Secondary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale at Weeks 2, 4, 8, 12 and 16
Description: WOMAC: Self-administered, disease-specific questionnaire which assesses clinically important, participant-relevant symptoms for pain, stiffness and physical function in participants with OA. The WOMAC pain subscale is a 5-item questionnaire used to assess the amount of pain experienced due to osteoarthritis of index joint (knee or hip) during past 48 hours. It was calculated as the mean of scores from 5 individual questions scored on a numerical rating scale (NRS). Scores for each question and WOMAC Pain subscale score on NRS ranged from 0 (no pain) to 10 (extreme pain), where higher scores indicated higher pain.
Time Frame: Baseline, Weeks 2, 4, 8, 12 and 16
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg
Number analyzed (Participants) | 282 | 283 | 284
units on a scale
  Change at Week 2 | -1.35 (0.14) | -2.02 (0.14) | -1.69 (0.14)
  Change at Week 4 | -1.78 (0.15) | -2.57 (0.15) | -2.56 (0.15)
  Change at Week 8 | -1.84 (0.15) | -2.47 (0.15) | -2.61 (0.15)
  Change at Week 12 | -2.19 (0.17) | -2.91 (0.16) | -2.96 (0.16)
  Change at Week 16 | -2.10 (0.17) | -2.69 (0.17) | -2.69 (0.17)
Statistical Analysis 1: Comparison: Placebo vs Tanezumab 2.5 mg; Week 2: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets includes treatment, randomization stratification variables (index joint and highest Kellgren-Lawrence grade) as fixed effects, baseline WOMAC pain subscales and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p < .0001, ANCOVA; Least Square Mean Difference = -0.67, 95% CI 2-sided [-0.94 to -0.40], Standard Error of Mean 0.14
Statistical Analysis 2: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.0149, ANCOVA; Least Square Mean Difference = -0.34, 95% CI 2-sided [-0.61 to -0.07], Standard Error of Mean 0.14
Statistical Analysis 3: Comparison: Placebo vs Tanezumab 2.5 mg; Week 4: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets includes treatment, randomization stratification variables (index joint and highest Kellgren-Lawrence grade) as fixed effects, baseline WOMAC pain subscales and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p < .0001, ANCOVA; Least Square Mean Difference = -0.79, 95% CI 2-sided [-1.08 to -0.50], Standard Error of Mean 0.15
Statistical Analysis 4: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 4, analysis 3]; Test type: Superiority; p < .0001, ANCOVA; Least Square Mean Difference = -0.78, 95% CI 2-sided [-1.07 to -0.50], Standard Error of Mean 0.15
Statistical Analysis 5: Comparison: Placebo vs Tanezumab 2.5 mg; Week 8: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets includes treatment, randomization stratification variables (index joint and highest Kellgren-Lawrence grade) as fixed effects, baseline WOMAC pain subscales and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p < .0001, ANCOVA; Least Square Mean Difference = -0.62, 95% CI 2-sided [-0.92 to -0.32], Standard Error of Mean 0.15
Statistical Analysis 6: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 4, analysis 5]; Test type: Superiority; p < .0001, ANCOVA; Least Square Mean Difference = -0.77, 95% CI 2-sided [-1.07 to -0.47], Standard Error of Mean 0.15
Statistical Analysis 7: Comparison: Placebo vs Tanezumab 2.5 mg; Week 12: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets includes treatment, randomization stratification variables (index joint and highest Kellgren-Lawrence grade) as fixed effects, baseline WOMAC pain subscales and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p < .0001, ANCOVA; Least Square Mean Difference = -0.72, 95% CI 2-sided [-1.05 to -0.39], Standard Error of Mean 0.17
Statistical Analysis 8: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 4, analysis 7]; Test type: Superiority; p < .0001, ANCOVA; Least Square Mean Difference = -0.77, 95% CI 2-sided [-1.09 to -0.44], Standard Error of Mean 0.17
Statistical Analysis 9: Comparison: Placebo vs Tanezumab 2.5 mg; Week 16: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets includes treatment, randomization stratification variables (index joint and highest Kellgren-Lawrence grade) as fixed effects, baseline WOMAC pain subscales and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p = 0.0005, ANCOVA; Least Square Mean Difference = -0.59, 95% CI 2-sided [-0.93 to -0.26], Standard Error of Mean 0.17
Statistical Analysis 10: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 4, analysis 9]; Test type: Superiority; p = 0.0004, ANCOVA; Least Square Mean Difference = -0.60, 95% CI 2-sided [-0.93 to -0.27], Standard Error of Mean 0.17

5. Secondary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale at Week 32
Description: as for outcome 4
Time Frame: Baseline, Week 32
Population: The intent to treat population included all randomized participants who received at least one dose of subcutaneous study medication (either tanezumab or placebo). Here, 'Number analyzed' = Participants evaluable for this outcome measure at specified time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg
Number analyzed (Participants) | 282 | 283 | 284
units on a scale
  Baseline: number analyzed (Participants) | 281 | 282 | 284
  Baseline | 6.59 (0.94) | 6.70 (0.94) | 6.60 (0.89)
  Change at Week 32: number analyzed (Participants) | 231 | 247 | 246
  Change at Week 32 | -2.70 (2.06) | -2.29 (1.95) | -2.26 (2.24)

6. Secondary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Physical Function Subscale at Weeks 2, 4, 8, 12 and 16
Description: as for outcome 2
Time Frame: Baseline, Weeks 2, 4, 8, 12 and 16
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg
Number analyzed (Participants) | 282 | 283 | 284
units on a scale
  Change at Week 2 | -1.26 (0.14) | -1.95 (0.14) | -1.69 (0.14)
  Change at Week 4 | -1.71 (0.15) | -2.52 (0.15) | -2.50 (0.15)
  Change at Week 8 | -1.76 (0.15) | -2.38 (0.15) | -2.52 (0.15)
  Change at Week 12 | -2.04 (2.16) | -2.83 (0.16) | -2.87 (0.16)
  Change at Week 16 | -2.02 (0.17) | -2.68 (0.16) | -2.69 (0.16)
Statistical Analysis 1: Comparison: Placebo vs Tanezumab 2.5 mg; Week 2: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets includes treatment, randomization stratification variables (index joint and highest Kellgren-Lawrence grade) as fixed effects, baseline WOMAC physical function subscale and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p < .0001, ANCOVA; Least Square Mean Difference = -0.69, 95% CI 2-sided [-0.95 to -0.42], Standard Error of Mean 0.14
Statistical Analysis 2: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = 0.0014, ANCOVA; Least Square Mean Difference = -0.43, 95% CI 2-sided [-0.70 to -0.17], Standard Error of Mean 0.14
Statistical Analysis 3: Comparison: Placebo vs Tanezumab 2.5 mg; Week 4: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets includes treatment, randomization stratification variables (index joint and highest Kellgren-Lawrence grade) as fixed effects, baseline WOMAC physical function subscale and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p < .0001, ANCOVA; Least Square Mean Difference = -0.81, 95% CI 2-sided [-1.09 to -0.53], Standard Error of Mean 0.14
Statistical Analysis 4: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 6, analysis 3]; Test type: Superiority; p < .0001, ANCOVA; Least Square Mean Difference = -0.79, 95% CI 2-sided [-1.08 to -0.51], Standard Error of Mean 0.14
Statistical Analysis 5: Comparison: Placebo vs Tanezumab 2.5 mg; Week 8: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets includes treatment, randomization stratification variables (index joint and highest Kellgren-Lawrence grade) as fixed effects, baseline WOMAC physical function subscale and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p < .0001, ANCOVA; Least Square Mean Difference = -0.63, 95% CI 2-sided [-0.93 to -0.33], Standard Error of Mean 0.15
Statistical Analysis 6: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 6, analysis 5]; Test type: Superiority; p < .0001, ANCOVA; Least Square Mean Difference = -0.76, 95% CI 2-sided [-1.06 to -0.47], Standard Error of Mean 0.15
Statistical Analysis 7: Comparison: Placebo vs Tanezumab 2.5 mg; Week 12: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets includes treatment, randomization stratification variables (index joint and highest Kellgren-Lawrence grade) as fixed effects, baseline WOMAC physical function subscale and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p < .0001, ANCOVA; Least Square Mean Difference = -0.79, 95% CI 2-sided [-1.11 to -0.46], Standard Error of Mean 0.16
Statistical Analysis 8: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 6, analysis 7]; Test type: Superiority; p < .0001, ANCOVA; Least Square Mean Difference = -0.82, 95% CI 2-sided [-1.15 to -0.50], Standard Error of Mean 0.16
Statistical Analysis 9: Comparison: Placebo vs Tanezumab 2.5 mg; Week 16: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets includes treatment, randomization stratification variables (index joint and highest Kellgren-Lawrence grade) as fixed effects, baseline WOMAC physical function subscale and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p < .0001, ANCOVA; Least Square Mean Difference = -0.67, 95% CI 2-sided [-1.00 to -0.34], Standard Error of Mean 0.17
Statistical Analysis 10: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 6, analysis 9]; Test type: Superiority; p < .0001, ANCOVA; Least Square Mean Difference = -0.68, 95% CI 2-sided [-1.00 to -0.35], Standard Error of Mean 0.17

7. Secondary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Physical Function Subscale at Week 32
Description: as for outcome 2
Time Frame: Baseline, Week 32
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg
Number analyzed (Participants) | 282 | 283 | 284
units on a scale
  Baseline: number analyzed (Participants) | 281 | 282 | 284
  Baseline | 6.59 (0.94) | 6.70 (0.94) | 6.60 (0.89)
  Change at Week 32: number analyzed (Participants) | 231 | 247 | 246
  Change at Week 32 | -2.70 (2.06) | -2.29 (1.95) | -2.26 (2.24)

8. Secondary Outcome: Change From Baseline in Patient's Global Assessment (PGA) of Osteoarthritis at Weeks 2, 4, 8, 12 and 16
Description: PGA of OA was assessed by asking a question from participants: "Considering all the ways your osteoarthritis in your knee or hip (index joint) affects you, how are you doing today?" Participants responded on a scale ranging from 1-5, where 1=very good (no symptom and no limitation of normal activities), 2= good (mild symptoms and no limitation of normal activities), 3= fair (moderate symptoms and limitation of some normal activities), 4= poor (severe symptoms and inability to carry out most normal activities), and 5 = very poor (very severe symptoms and inability to carry out all normal activities).
Time Frame: Baseline, Weeks 2, 4, 8, 12 and 16
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg
Number analyzed (Participants) | 282 | 283 | 284
units on a scale
  Change at Week 2 | -0.50 (0.05) | -0.73 (0.05) | -0.67 (0.05)
  Change at Week 4 | -0.60 (0.05) | -0.85 (0.05) | -0.93 (0.05)
  Change at Week 8 | -0.62 (0.05) | -0.79 (0.05) | -0.88 (0.05)
  Change at Week 12 | -0.71 (0.06) | -0.99 (0.06) | -1.03 (0.06)
  Change at Week 16 | -0.64 (0.06) | -0.78 (0.06) | -0.90 (0.06)
Statistical Analysis 1: Comparison: Placebo vs Tanezumab 2.5 mg; Week 2: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets includes treatment, randomization stratification variables (index joint and highest Kellgren-Lawrence grade) as fixed effects, baseline PGA of osteoarthritis and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p < .0001, ANCOVA; Least Square Mean Difference = -0.23, 95% CI 2-sided [-0.33 to -0.12], Standard Error of Mean 0.05
Statistical Analysis 2: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.0022, ANCOVA; Least Square Mean Difference = -0.17, 95% CI 2-sided [-0.27 to -0.06], Standard Error of Mean 0.05
Statistical Analysis 3: Comparison: Placebo vs Tanezumab 2.5 mg; Week 4: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets includes treatment, randomization stratification variables (index joint and highest Kellgren-Lawrence grade) as fixed effects, baseline PGA of osteoarthritis and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p < .0001, ANCOVA; Least Square Mean Difference = -0.24, 95% CI 2-sided [-0.35 to -0.14], Standard Error of Mean 0.05
Statistical Analysis 4: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 8, analysis 3]; Test type: Superiority; p < .0001, ANCOVA; Least Square Mean Difference = -0.32, 95% CI 2-sided [-0.43 to -0.22], Standard Error of Mean 0.05
Statistical Analysis 5: Comparison: Placebo vs Tanezumab 2.5 mg; Week 8: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets includes treatment, randomization stratification variables (index joint and highest Kellgren-Lawrence grade) as fixed effects, baseline PGA of osteoarthritis and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p = 0.0029, ANCOVA; Least Square Mean Difference = -0.17, 95% CI 2-sided [-0.28 to -0.06], Standard Error of Mean 0.06
Statistical Analysis 6: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 8, analysis 5]; Test type: Superiority; p < .0001, ANCOVA; Least Square Mean Difference = -0.26, 95% CI 2-sided [-0.37 to -0.15], Standard Error of Mean 0.06
Statistical Analysis 7: Comparison: Placebo vs Tanezumab 2.5 mg; Week 12: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets includes treatment, randomization stratification variables (index joint and highest Kellgren-Lawrence grade) as fixed effects, baseline PGA of osteoarthritis and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p < .0001, ANCOVA; Least Square Mean Difference = -0.29, 95% CI 2-sided [-0.40 to -0.17], Standard Error of Mean 0.06
Statistical Analysis 8: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 8, analysis 7]; Test type: Superiority; p < .0001, ANCOVA; Least Square Mean Difference = -0.32, 95% CI 2-sided [-0.43 to -0.20], Standard Error of Mean 0.06
Statistical Analysis 9: Comparison: Placebo vs Tanezumab 2.5 mg; Week 16: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets includes treatment, randomization stratification variables (index joint and highest Kellgren-Lawrence grade) as fixed effects, baseline PGA of osteoarthritis and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p = 0.0352, ANCOVA; Least Square Mean Difference = -0.13, 95% CI 2-sided [-0.26 to -0.01], Standard Error of Mean 0.06
Statistical Analysis 10: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 8, analysis 9]; Test type: Superiority; p < .0001, ANCOVA; Least Square Mean Difference = -0.25, 95% CI 2-sided [-0.37 to -0.13], Standard Error of Mean 0.06

9. Secondary Outcome: Change From Baseline in Patient's Global Assessment (PGA) of Osteoarthritis at Week 32
Description: PGA of OA was assessed by asking a question from participants: "Considering all the ways your osteoarthritis in your knee or hip (index joint) affects you, how are you doing today?" Participants responded on a scale ranging from 1-5, where 1=very good (no symptom and no limitation of normal activities), 2= good (mild symptoms and no limitation of normal activities), 3= fair (moderate symptoms and limitation of some normal activities), 4= poor (severe symptoms and inability to carry out most normal activities), and 5 = very poor (very severe symptoms and inability to carry out all normal activities). Higher scores indicated worse condition.
Time Frame: Baseline, Week 32
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg
Number analyzed (Participants) | 282 | 283 | 284
units on a scale
  Baseline: number analyzed (Participants) | 281 | 282 | 284
  Baseline | 3.55 (0.62) | 3.61 (0.62) | 3.56 (0.63)
  Change at Week 32: number analyzed (Participants) | 231 | 247 | 246
  Change at Week 32 | -0.84 (0.87) | -0.64 (0.88) | -0.63 (0.91)

10. Secondary Outcome: Percentage of Participants Meeting Outcomes Measures in Arthritis Clinical Trials-Osteoarthritis Research Society International (OMERACT-OARSI) Responder Index
Description: Participants were considered as OMERACT-OARSI responders: if the change (improvement) from baseline to week of interest was greater than or equal to (>=) 50 percent and >= 2 units in either WOMAC pain subscale or physical function subscale score; if change (improvement) from baseline to week of interest was >=20 percent and >=1 unit in at least 2 of the following: 1) WOMAC pain subscale score, 2) WOMAC physical function subscale score, 3) PGA of osteoarthritis. WOMAC pain subscale assess amount of pain experienced (score: 0 [no pain] to 10 [extreme pain], higher score = more pain), WOMAC physical function subscale assess degree of difficulty experienced (score: 0 [minimum difficulty] to 10 [extreme difficulty], higher score = worse physical function) and PGA of OA (score: 1 [very good] to 5 [very poor], higher score = worse condition). Missing data was imputed using mixed baseline/last observation carried forward (BOCF/LOCF).
Time Frame: Weeks 2, 4, 8, 12, 16, 24 and 32
Population: ITT population included all randomized participants who received at least one dose of subcutaneous study medication (either tanezumab or placebo). Here 'Overall number of participants analyzed' = participants who were evaluable for this outcome measure and 'Number analyzed' = participants evaluable for this outcome measure at specified time points.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg
Number analyzed (Participants) | 281 | 282 | 284
percentage of participants
  Week 2 | 44.1 | 63.1 | 54.9
  Week 4 | 53.0 | 74.8 | 71.8
  Week 8 | 61.9 | 75.5 | 75.4
  Week 12 | 68.7 | 80.9 | 81.0
  Week 16 | 64.4 | 78.7 | 76.1
  Week 24 | 65.1 | 76.2 | 77.1
  Week 32: number analyzed (Participants) | 231 | 247 | 246
  Week 32 | 74.0 | 66.4 | 63.0
Statistical Analysis 1: Comparison: Placebo vs Tanezumab 2.5 mg; Week 2: Odds ratio and 95 percent (%) confidence interval (CI) estimated from logistic regression model. Logistic regression model included baseline WOMAC pain subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p < .0001, Regression, Logistic; Odds Ratio (OR) = 2.23, 95% CI 2-sided [1.59 to 3.14]
Statistical Analysis 2: Comparison: Placebo vs Tanezumab 5 mg; Week 2: Odds ratio and 95% CI estimated from logistic regression model. Logistic regression model included baseline WOMAC pain subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p = 0.0085, Regression, Logistic; Odds Ratio (OR) = 1.56, 95% CI 2-sided [1.12 to 2.18]
Statistical Analysis 3: Comparison: Placebo vs Tanezumab 2.5 mg; Week 4: Odds ratio and 95% CI estimated from logistic regression model. Logistic regression model included baseline WOMAC pain subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p < .0001, Regression, Logistic; Odds Ratio (OR) = 2.71, 95% CI 2-sided [1.89 to 3.88]
Statistical Analysis 4: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 10, analysis 3]; Test type: Superiority; p < .0001, Regression, Logistic; Odds Ratio (OR) = 2.31, 95% CI 2-sided [1.62 to 3.28]
Statistical Analysis 5: Comparison: Placebo vs Tanezumab 2.5 mg; Week 8: Odds ratio and 95% CI estimated from logistic regression model. Logistic regression model included baseline WOMAC pain subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p = 0.0005, Regression, Logistic; Odds Ratio (OR) = 1.91, 95% CI 2-sided [1.33 to 2.75]
Statistical Analysis 6: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 10, analysis 5]; Test type: Superiority; p = 0.0005, Regression, Logistic; Odds Ratio (OR) = 1.90, 95% CI 2-sided [1.32 to 2.73]
Statistical Analysis 7: Comparison: Placebo vs Tanezumab 2.5 mg; Week 12: Odds ratio and 95% CI estimated from logistic regression model. Logistic regression model included baseline WOMAC pain subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p = 0.0009, Regression, Logistic; Odds Ratio (OR) = 1.94, 95% CI 2-sided [1.31 to 2.86]
Statistical Analysis 8: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 10, analysis 7]; Test type: Superiority; p = 0.0008, Regression, Logistic; Odds Ratio (OR) = 1.95, 95% CI 2-sided [1.32 to 2.89]
Statistical Analysis 9: Comparison: Placebo vs Tanezumab 2.5 mg; Week 16: Odds ratio and 95% CI estimated from logistic regression model. Logistic regression model included baseline WOMAC pain subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p = 0.0002, Regression, Logistic; Odds Ratio (OR) = 2.06, 95% CI 2-sided [1.41 to 3.01]
Statistical Analysis 10: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 10, analysis 9]; Test type: Superiority; p = 0.0022, Regression, Logistic; Odds Ratio (OR) = 1.78, 95% CI 2-sided [1.23 to 2.57]
Statistical Analysis 11: Comparison: Placebo vs Tanezumab 2.5 mg; Week 24: Odds ratio and 95% CI estimated from logistic regression model. Logistic regression model included baseline WOMAC pain subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p = 0.0032, Regression, Logistic; Odds Ratio (OR) = 1.75, 95% CI 2-sided [1.21 to 2.54]
Statistical Analysis 12: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 10, analysis 11]; Test type: Superiority; p = 0.0013, Regression, Logistic; Odds Ratio (OR) = 1.85, 95% CI 2-sided [1.27 to 2.69]

11. Secondary Outcome: Percentage of Participants With Cumulative Percent Change From Baseline in the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale at Weeks 16 and 24
Description: WOMAC: Self-administered, disease-specific questionnaire which assesses clinically important, participant-relevant symptoms for pain, stiffness and physical function in participants with OA. The WOMAC pain subscale is a 5-item questionnaire used to assess the amount of pain experienced due to OA of index joint during past 48 hours. It was calculated as the mean of scores from 5 individual questions scored on a NRS. Scores for each question and WOMAC Pain subscale score on NRS ranged from 0 (no pain) to 10 (extreme pain), where higher scores indicated higher pain. Percentage of participants with cumulative reduction (as percent) (greater than 0% ; >= 10, 20, 30, 40, 50, 60, 70, 80 and 90%; = 100 %) in WOMAC pain subscale from Baseline to Weeks 16 and 24 were reported, participants (%) are reported more than once in categories specified. Missing data was imputed using mixed BOCF/LOCF.
Time Frame: Baseline, Weeks 16 and 24
Population: The intent to treat population included all randomized participants who received at least one dose of subcutaneous study medication (either tanezumab or placebo). Here, 'Overall number of participants analyzed' = Participants evaluable for this outcome measure.
Measure: Number; unit: percentage of Participants
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg
Number analyzed (Participants) | 281 | 282 | 284
percentage of Participants
  Week 16: >0% | 81.9 | 91.8 | 89.4
  Week 16: >=10% | 77.6 | 87.6 | 82.0
  Week 16: >=20% | 66.9 | 79.4 | 76.1
  Week 16: >=30% | 56.2 | 68.1 | 68.7
  Week 16: >=40% | 45.2 | 57.8 | 59.9
  Week 16: >=50% | 35.9 | 49.6 | 47.5
  Week 16: >=60% | 27.0 | 34.4 | 36.6
  Week 16: >=70% | 17.1 | 22.3 | 24.3
  Week 16: >=80% | 10.0 | 14.5 | 14.4
  Week 16: >=90% | 3.2 | 7.4 | 4.9
  Week 16: =100% | 1.1 | 1.8 | 3.2
  Week 24: >0% | 80.1 | 89.7 | 88.4
  Week 24: >=10% | 70.8 | 83.0 | 83.5
  Week 24: >=20% | 65.8 | 76.2 | 76.8
  Week 24: >=30% | 56.6 | 65.6 | 68.7
  Week 24: >=40% | 44.8 | 55.0 | 59.2
  Week 24: >=50% | 33.8 | 45.4 | 47.9
  Week 24: >=60% | 24.9 | 33.3 | 36.6
  Week 24: >=70% | 17.8 | 21.3 | 23.2
  Week 24: >=80% | 11.4 | 12.1 | 14.1
  Week 24: >=90% | 3.2 | 5.3 | 6.0
  Week 24: =100% | 1.1 | 0.7 | 2.8

12. Secondary Outcome: Percentage of Participants Achieving Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale Reduction >=30 Percent (%), >=50%, >=70% and >=90% Response
Description: Percentage of participants with reduction in WOMAC pain intensity of at least (>=) 30%, 50%, 70% and 90% at Weeks 2, 4, 8, 12, 16, 24 and 32 compared to baseline were classified as responders to WOMAC pain subscale and are reported here. WOMAC: Self-administered, disease-specific questionnaire which assesses clinically important, participant-relevant symptoms for pain, stiffness and physical function in participants with OA. The WOMAC pain subscale is a 5-item questionnaire used to assess the amount of pain experienced due to OA of index joint (knee or hip) during past 48 hours. It was calculated as the mean of scores from 5 individual questions scored on a NRS. Scores for each question and WOMAC Pain subscale score on NRS ranged from 0 (no pain) to 10 (extreme pain), where higher scores indicated higher pain. Missing data was imputed using mixed BOCF/LOCF.
Time Frame: Week 2, 4, 8, 12, 16, 24 and 32
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg
Number analyzed (Participants) | 281 | 282 | 284
percentage of participants
  Week 2: At least 30% reduction | 33.5 | 46.8 | 42.6
  Week 2: At least 50% reduction | 16.7 | 27.7 | 18.3
  Week 2: At least 70% reduction | 5.0 | 10.3 | 6.7
  Week 2: At least 90% reduction | 1.1 | 2.5 | 1.4
  Week 4: At least 30% reduction | 45.2 | 61.3 | 58.8
  Week 4: At least 50% reduction | 22.8 | 33.0 | 37.7
  Week 4: At least 70% reduction | 8.5 | 13.1 | 15.8
  Week 4: At least 90% reduction | 1.4 | 3.9 | 4.9
  Week 8: At least 30% reduction | 50.5 | 64.2 | 61.6
  Week 8: At least 50% reduction | 26.0 | 37.2 | 44.4
  Week 8: At least 70% reduction | 10.7 | 15.2 | 22.2
  Week 8: At least 90% reduction | 2.1 | 4.3 | 5.6
  Week 12: At least 30% reduction | 58.4 | 71.6 | 71.1
  Week 12: At least 50% reduction | 33.8 | 46.8 | 50.7
  Week 12: At least 70% reduction | 15.7 | 24.1 | 23.2
  Week 12: At least 90% reduction | 1.8 | 8.5 | 7.0
  Week 16: At least 30% reduction | 56.2 | 68.1 | 68.7
  Week 16: At least 50% reduction | 35.9 | 49.6 | 47.5
  Week 16: At least 70% reduction | 17.1 | 22.3 | 24.3
  Week 16: At least 90% reduction | 3.2 | 7.4 | 4.9
  Week 24: At least 30% reduction | 56.6 | 65.6 | 68.7
  Week 24: At least 50% reduction | 33.8 | 45.4 | 47.9
  Week 24: At least 70% reduction | 17.8 | 21.3 | 23.2
  Week 24: At least 90% reduction | 3.2 | 5.3 | 6.0
  Week 32: At least 30% reduction: number analyzed (Participants) | 231 | 247 | 246
  Week 32: At least 30% reduction | 65.4 | 54.7 | 57.3
  Week 32: At least 50% reduction: number analyzed (Participants) | 231 | 247 | 246
  Week 32: At least 50% reduction | 43.7 | 32.8 | 32.9
  Week 32: At least 70% reduction: number analyzed (Participants) | 231 | 247 | 246
  Week 32: At least 70% reduction | 21.2 | 12.1 | 15.4
  Week 32: At least 90% reduction: number analyzed (Participants) | 231 | 247 | 246
  Week 32: At least 90% reduction | 4.8 | 1.6 | 4.9
Statistical Analysis 1: Comparison: Placebo vs Tanezumab 2.5 mg; Week 2, >=30%: Odds ratio and 95% CI estimated from logistic regression model. Logistic regression model included baseline WOMAC pain subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p = 0.0006, Regression, Logistic; Odds Ratio (OR) = 1.83, 95% CI 2-sided [1.30 to 2.59]
Statistical Analysis 2: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 12, analysis 1]; Test type: Superiority; p = 0.0160, Regression, Logistic; Odds Ratio (OR) = 1.53, 95% CI 2-sided [1.08 to 2.16]
Statistical Analysis 3: Comparison: Placebo vs Tanezumab 2.5 mg; Week 2, >=50%: Odds ratio and 95% CI estimated from logistic regression model. Logistic regression model included baseline WOMAC pain subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p = 0.0008, Regression, Logistic; Odds Ratio (OR) = 2.03, 95% CI 2-sided [1.34 to 3.07]
Statistical Analysis 4: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 12, analysis 3]; Test type: Superiority; p = 0.5118, Regression, Logistic; Odds Ratio (OR) = 1.16, 95% CI 2-sided [0.75 to 1.80]
Statistical Analysis 5: Comparison: Placebo vs Tanezumab 2.5 mg; Week 2, >=70%: Odds ratio and 95% CI estimated from logistic regression model. Logistic regression model included baseline WOMAC pain subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p = 0.0093, Regression, Logistic; Odds Ratio (OR) = 2.45, 95% CI 2-sided [1.25 to 4.81]
Statistical Analysis 6: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 12, analysis 5]; Test type: Superiority; p = 0.3017, Regression, Logistic; Odds Ratio (OR) = 1.46, 95% CI 2-sided [0.71 to 3.01]
Statistical Analysis 7: Comparison: Placebo vs Tanezumab 2.5 mg; Week 2, >=90%: Odds ratio and 95% CI estimated from logistic regression model. Logistic regression model included baseline WOMAC pain subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p = 0.2160, Regression, Logistic; Odds Ratio (OR) = 2.40, 95% CI 2-sided [0.60 to 9.58]
Statistical Analysis 8: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 12, analysis 7]; Test type: Superiority; p = 0.7174, Regression, Logistic; Odds Ratio (OR) = 1.33, 95% CI 2-sided [0.29 to 6.08]
Statistical Analysis 9: Comparison: Placebo vs Tanezumab 2.5 mg; Week 4, >=30%: Odds ratio and 95% CI estimated from logistic regression model. Logistic regression model included baseline WOMAC pain subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p < .0001, Regression, Logistic; Odds Ratio (OR) = 2.04, 95% CI 2-sided [1.45 to 2.87]
Statistical Analysis 10: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 12, analysis 9]; Test type: Superiority; p = 0.0006, Regression, Logistic; Odds Ratio (OR) = 1.81, 95% CI 2-sided [1.29 to 2.54]
Statistical Analysis 11: Comparison: Placebo vs Tanezumab 2.5 mg; Week 4, >=50%: Odds ratio and 95% CI estimated from logistic regression model. Logistic regression model included baseline WOMAC pain subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p = 0.0024, Regression, Logistic; Odds Ratio (OR) = 1.81, 95% CI 2-sided [1.23 to 2.65]
Statistical Analysis 12: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 12, analysis 11]; Test type: Superiority; p < .0001, Regression, Logistic; Odds Ratio (OR) = 2.17, 95% CI 2-sided [1.49 to 3.16]
Statistical Analysis 13: Comparison: Placebo vs Tanezumab 2.5 mg; Week 4, >=70%: Odds ratio and 95% CI estimated from logistic regression model. Logistic regression model included baseline WOMAC pain subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p = 0.0373, Regression, Logistic; Odds Ratio (OR) = 1.80, 95% CI 2-sided [1.04 to 3.14]
Statistical Analysis 14: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 12, analysis 13]; Test type: Superiority; p = 0.0046, Regression, Logistic; Odds Ratio (OR) = 2.17, 95% CI 2-sided [1.27 to 3.72]
Statistical Analysis 15: Comparison: Placebo vs Tanezumab 2.5 mg; Week 4, >=90%: Odds ratio and 95% CI estimated from logistic regression model. Logistic regression model included baseline WOMAC pain subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p = 0.0683, Regression, Logistic; Odds Ratio (OR) = 2.95, 95% CI 2-sided [0.92 to 9.47]
Statistical Analysis 16: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 12, analysis 15]; Test type: Superiority; p = 0.0214, Regression, Logistic; Odds Ratio (OR) = 3.77, 95% CI 2-sided [1.22 to 11.66]
Statistical Analysis 17: Comparison: Placebo vs Tanezumab 2.5 mg; Week 8, >=30%: Odds ratio and 95% CI estimated from logistic regression model. Logistic regression model included baseline WOMAC pain subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p = 0.0006, Regression, Logistic; Odds Ratio (OR) = 1.83, 95% CI 2-sided [1.30 to 2.58]
Statistical Analysis 18: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 12, analysis 17]; Test type: Superiority; p = 0.0048, Regression, Logistic; Odds Ratio (OR) = 1.63, 95% CI 2-sided [1.16 to 2.28]
Statistical Analysis 19: Comparison: Placebo vs Tanezumab 2.5 mg; Week 8, >=50%: Odds ratio and 95% CI estimated from logistic regression model. Logistic regression model included baseline WOMAC pain subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p = 0.0012, Regression, Logistic; Odds Ratio (OR) = 1.84, 95% CI 2-sided [1.27 to 2.65]
Statistical Analysis 20: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 12, analysis 19]; Test type: Superiority; p < .0001, Regression, Logistic; Odds Ratio (OR) = 2.41, 95% CI 2-sided [1.68 to 3.47]
Statistical Analysis 21: Comparison: Placebo vs Tanezumab 2.5 mg; Week 8, >=70%: Odds ratio and 95% CI estimated from logistic regression model. Logistic regression model included baseline WOMAC pain subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p = 0.0537, Regression, Logistic; Odds Ratio (OR) = 1.65, 95% CI 2-sided [0.99 to 2.74]
Statistical Analysis 22: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 12, analysis 21]; Test type: Superiority; p = 0.0001, Regression, Logistic; Odds Ratio (OR) = 2.55, 95% CI 2-sided [1.58 to 4.13]
Statistical Analysis 23: Comparison: Placebo vs Tanezumab 2.5 mg; Week 8, >=90%: Odds ratio and 95% CI estimated from logistic regression model. Logistic regression model included baseline WOMAC pain subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p = 0.1155, Regression, Logistic; Odds Ratio (OR) = 2.26, 95% CI 2-sided [0.82 to 6.27]
Statistical Analysis 24: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 12, analysis 23]; Test type: Superiority; p = 0.0271, Regression, Logistic; Odds Ratio (OR) = 3.00, 95% CI 2-sided [1.13 to 7.96]
Statistical Analysis 25: Comparison: Placebo vs Tanezumab 2.5 mg; Week 12, >=30%: Odds ratio and 95% CI estimated from logistic regression model. Logistic regression model included baseline WOMAC pain subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p = 0.0007, Regression, Logistic; Odds Ratio (OR) = 1.85, 95% CI 2-sided [1.30 to 2.63]
Statistical Analysis 26: Comparison: Placebo; [analysis description as in outcome 12, analysis 25]; Test type: Superiority; p = 0.0011, Regression, Logistic; Odds Ratio (OR) = 1.80, 95% CI 2-sided [1.26 to 2.56]
Statistical Analysis 27: Comparison: Placebo vs Tanezumab 2.5 mg; Week 12, >=50%: Odds ratio and 95% CI estimated from logistic regression model. Logistic regression model included baseline WOMAC pain subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p = 0.0009, Regression, Logistic; Odds Ratio (OR) = 1.79, 95% CI 2-sided [1.27 to 2.52]
Statistical Analysis 28: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 12, analysis 27]; Test type: Superiority; p < .0001, Regression, Logistic; Odds Ratio (OR) = 2.07, 95% CI 2-sided [1.47 to 2.91]
Statistical Analysis 29: Comparison: Placebo vs Tanezumab 2.5 mg; Week 12, >=70%: Odds ratio and 95% CI estimated from logistic regression model. Logistic regression model included baseline WOMAC pain subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p = 0.0064, Regression, Logistic; Odds Ratio (OR) = 1.81, 95% CI 2-sided [1.18 to 2.78]
Statistical Analysis 30: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 12, analysis 29]; Test type: Superiority; p = 0.0180, Regression, Logistic; Odds Ratio (OR) = 1.68, 95% CI 2-sided [1.09 to 2.58]
Statistical Analysis 31: Comparison: Placebo vs Tanezumab 2.5 mg; Week 12, >=90%: Odds ratio and 95% CI estimated from logistic regression model. Logistic regression model included baseline WOMAC pain subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p = 0.0006, Regression, Logistic; Odds Ratio (OR) = 5.61, 95% CI 2-sided [2.09 to 15.08]
Statistical Analysis 32: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 12, analysis 31]; Test type: Superiority; p = 0.0034, Regression, Logistic; Odds Ratio (OR) = 4.46, 95% CI 2-sided [1.64 to 12.13]
Statistical Analysis 33: Comparison: Placebo vs Tanezumab 2.5 mg; Week 16, >=30%: Odds ratio and 95% CI estimated from logistic regression model. Logistic regression model included baseline WOMAC pain subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p = 0.0022, Regression, Logistic; Odds Ratio (OR) = 1.72, 95% CI 2-sided [1.22 to 2.44]
Statistical Analysis 34: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 12, analysis 33]; Test type: Superiority; p = 0.0014, Regression, Logistic; Odds Ratio (OR) = 1.77, 95% CI 2-sided [1.25 to 2.50]
Statistical Analysis 35: Comparison: Placebo vs Tanezumab 2.5 mg; Week 16, >=50%: Odds ratio and 95% CI estimated from logistic regression model. Logistic regression model included baseline WOMAC pain subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p = 0.0003, Regression, Logistic; Odds Ratio (OR) = 1.87, 95% CI 2-sided [1.33 to 2.64]
Statistical Analysis 36: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 12, analysis 35]; Test type: Superiority; p = 0.0030, Regression, Logistic; Odds Ratio (OR) = 1.68, 95% CI 2-sided [1.19 to 2.36]
Statistical Analysis 37: Comparison: Placebo vs Tanezumab 2.5 mg; Week 16, >=70%: Odds ratio and 95% CI estimated from logistic regression model. Logistic regression model included baseline WOMAC pain subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p = 0.0754, Regression, Logistic; Odds Ratio (OR) = 1.47, 95% CI 2-sided [0.96 to 2.24]
Statistical Analysis 38: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 12, analysis 37]; Test type: Superiority; p = 0.0253, Regression, Logistic; Odds Ratio (OR) = 1.61, 95% CI 2-sided [1.06 to 2.44]
Statistical Analysis 39: Comparison: Placebo vs Tanezumab 2.5 mg; Week 16, >=90%: Odds ratio and 95% CI estimated from logistic regression model. Logistic regression model included baseline WOMAC pain subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p = 0.0098, Regression, Logistic; Odds Ratio (OR) = 2.98, 95% CI 2-sided [1.30 to 6.83]
Statistical Analysis 40: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 12, analysis 39]; Test type: Superiority; p = 0.2230, Regression, Logistic; Odds Ratio (OR) = 1.72, 95% CI 2-sided [0.72 to 4.13]
Statistical Analysis 41: Comparison: Placebo vs Tanezumab 2.5 mg; Week 24, >=30%: Odds ratio and 95% CI estimated from logistic regression model. Logistic regression model included baseline WOMAC pain subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p = 0.0201, Regression, Logistic; Odds Ratio (OR) = 1.50, 95% CI 2-sided [1.07 to 2.12]
Statistical Analysis 42: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 12, analysis 41]; Test type: Superiority; p = 0.0021, Regression, Logistic; Odds Ratio (OR) = 1.73, 95% CI 2-sided [1.22 to 2.44]
Statistical Analysis 43: Comparison: Placebo vs Tanezumab 2.5 mg; Week 24, >=50%: Odds ratio and 95% CI estimated from logistic regression model. Logistic regression model included baseline WOMAC pain subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p = 0.0022, Regression, Logistic; Odds Ratio (OR) = 1.72, 95% CI 2-sided [1.22 to 2.43]
Statistical Analysis 44: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 12, analysis 43]; Test type: Superiority; p = 0.0004, Regression, Logistic; Odds Ratio (OR) = 1.87, 95% CI 2-sided [1.32 to 2.64]
Statistical Analysis 45: Comparison: Placebo vs Tanezumab 2.5 mg; Week 24, >=70%: Odds ratio and 95% CI estimated from logistic regression model. Logistic regression model included baseline WOMAC pain subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p = 0.2031, Regression, Logistic; Odds Ratio (OR) = 1.32, 95% CI 2-sided [0.86 to 2.01]
Statistical Analysis 46: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 12, analysis 45]; Test type: Superiority; p = 0.0867, Regression, Logistic; Odds Ratio (OR) = 1.44, 95% CI 2-sided [0.95 to 2.18]
Statistical Analysis 47: Comparison: Placebo vs Tanezumab 2.5 mg; Week 24, >=90%: Odds ratio and 95% CI estimated from logistic regression model. Logistic regression model included baseline WOMAC pain subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p = 0.1746, Regression, Logistic; Odds Ratio (OR) = 1.80, 95% CI 2-sided [0.77 to 4.22]
Statistical Analysis 48: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 12, analysis 47]; Test type: Superiority; p = 0.1039, Regression, Logistic; Odds Ratio (OR) = 1.99, 95% CI 2-sided [0.87 to 4.57]

13. Secondary Outcome: Percentage of Participants Achieving Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Physical Function Subscale Reduction >=30%, >=50%, >=70% and >=90% Response
Description: Percentage of participants with reduction in WOMAC physical function of at least (>=)30%,50%,70% and 90% at weeks 2,4,8,12,16,24 and 32 compared to baseline were classified as responders to WOMAC physical function subscale. WOMAC: Self-administered, disease-specific questionnaire which assesses clinically important, participant-relevant symptoms for pain, stiffness and physical function in participants with OA. Physical function:Participant's ability to move around and perform usual activities of daily living. WOMAC physical function subscale17-item questionnaire used to assess the degree of difficulty experienced due to OA in index joint (knee/hip) during past 48 hours, calculated as mean of the scores from 17 individual questions scored on a NRS. Scores for each question and WOMAC physical subscale on NRS ranged from 0 (no difficulty) to 10 (extreme difficulty), where higher scores indicated extreme difficulty/worse physical function. Missing data was imputed using mixed BOCF/LOCF.
Time Frame: Weeks 2, 4, 8, 12, 16, 24 and 32
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg
Number analyzed (Participants) | 281 | 282 | 284
percentage of participants
  Week 2: At least 30% reduction | 30.2 | 44.3 | 38.7
  Week 2: At least 50% reduction | 14.6 | 19.1 | 18.3
  Week 2: At least 70% reduction | 3.9 | 9.2 | 5.3
  Week 2: At least 90% reduction | 1.1 | 2.5 | 1.8
  Week 4: At least 30% reduction | 36.3 | 55.0 | 53.9
  Week 4: At least 50% reduction | 18.1 | 28.0 | 32.4
  Week 4: At least 70% reduction | 6.4 | 11.7 | 12.0
  Week 4: At least 90% reduction | 1.1 | 2.8 | 4.6
  Week 8: At least 30% reduction | 45.6 | 57.4 | 59.2
  Week 8: At least 50% reduction | 22.8 | 33.7 | 37.3
  Week 8: At least 70% reduction | 7.5 | 16.0 | 15.5
  Week 8: At least 90% reduction | 1.4 | 5.0 | 4.9
  Week 12: At least 30% reduction | 51.2 | 67.4 | 69.4
  Week 12: At least 50% reduction | 27.8 | 43.6 | 43.7
  Week 12: At least 70% reduction | 12.8 | 19.9 | 21.1
  Week 12: At least 90% reduction | 0.7 | 6.7 | 5.6
  Week 16: At least 30% reduction | 53.0 | 65.2 | 66.2
  Week 16: At least 50% reduction | 32.0 | 42.9 | 44.0
  Week 16: At least 70% reduction | 14.2 | 21.3 | 18.3
  Week 16: At least 90% reduction | 2.5 | 6.0 | 6.0
  Week 24: At least 30% reduction | 51.2 | 64.9 | 68.7
  Week 24: At least 50% reduction | 32.4 | 41.5 | 44.7
  Week 24: At least 70% reduction | 14.6 | 19.1 | 17.3
  Week 24: At least 90% reduction | 1.8 | 5.3 | 5.3
  Week 32: At least 30% reduction: number analyzed (Participants) | 231 | 247 | 246
  Week 32: At least 30% reduction | 60.2 | 51.4 | 53.7
  Week 32: At least 50% reduction: number analyzed (Participants) | 231 | 247 | 246
  Week 32: At least 50% reduction | 40.3 | 31.2 | 30.5
  Week 32: At least 70% reduction: number analyzed (Participants) | 231 | 247 | 246
  Week 32: At least 70% reduction | 16.9 | 11.7 | 11.4
  Week 32: At least 90% reduction: number analyzed (Participants) | 231 | 247 | 246
  Week 32: At least 90% reduction | 3.5 | 2.0 | 3.3
Statistical Analysis 1: Comparison: Placebo vs Tanezumab 2.5 mg; Week 2, >=30%: Odds ratio and 95%CI estimated from logistic regression model. Logistic regression model included baseline WOMAC physical function subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p = 0.0003, Regression, Logistic; Odds Ratio (OR) = 1.89, 95% CI 2-sided [1.33 to 2.68]
Statistical Analysis 2: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 13, analysis 1]; Test type: Superiority; p = 0.0286, Regression, Logistic; Odds Ratio (OR) = 1.48, 95% CI 2-sided [1.04 to 2.10]
Statistical Analysis 3: Comparison: Placebo vs Tanezumab 2.5 mg; Week 2, >=50%: Odds ratio and 95%CI estimated from logistic regression model. Logistic regression model included baseline WOMAC physical function subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p = 0.1031, Regression, Logistic; Odds Ratio (OR) = 1.45, 95% CI 2-sided [0.93 to 2.27]
Statistical Analysis 4: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 13, analysis 3]; Test type: Superiority; p = 0.2033, Regression, Logistic; Odds Ratio (OR) = 1.34, 95% CI 2-sided [0.85 to 2.10]
Statistical Analysis 5: Comparison: Placebo vs Tanezumab 2.5 mg; Week 2, >=70%: Odds ratio and 95%CI estimated from logistic regression model. Logistic regression model included baseline WOMAC physical function subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p = 0.0064, Regression, Logistic; Odds Ratio (OR) = 2.80, 95% CI 2-sided [1.34 to 5.86]
Statistical Analysis 6: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 13, analysis 5]; Test type: Superiority; p = 0.3706, Regression, Logistic; Odds Ratio (OR) = 1.44, 95% CI 2-sided [0.65 to 3.23]
Statistical Analysis 7: Comparison: Placebo vs Tanezumab 2.5 mg; Week 2, >=90%: Odds ratio and 95%CI estimated from logistic regression model. Logistic regression model included baseline WOMAC physical function subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p = 0.2121, Regression, Logistic; Odds Ratio (OR) = 2.39, 95% CI 2-sided [0.61 to 9.41]
Statistical Analysis 8: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 13, analysis 7]; Test type: Superiority; p = 0.4859, Regression, Logistic; Odds Ratio (OR) = 1.67, 95% CI 2-sided [0.39 to 7.11]
Statistical Analysis 9: Comparison: Placebo vs Tanezumab 2.5 mg; Week 4, >=30%: Odds ratio and 95%CI estimated from logistic regression model. Logistic regression model included baseline WOMAC physical function subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p < .0001, Regression, Logistic; Odds Ratio (OR) = 2.25, 95% CI 2-sided [1.60 to 3.17]
Statistical Analysis 10: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 13, analysis 9]; Test type: Superiority; p < .0001, Regression, Logistic; Odds Ratio (OR) = 2.10, 95% CI 2-sided [1.50 to 2.96]
Statistical Analysis 11: Comparison: Placebo vs Tanezumab 2.5 mg; Week 4, >=50%: Odds ratio and 95%CI estimated from logistic regression model. Logistic regression model included baseline WOMAC physical function subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p = 0.0020, Regression, Logistic; Odds Ratio (OR) = 1.91, 95% CI 2-sided [1.27 to 2.87]
Statistical Analysis 12: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 13, analysis 11]; Test type: Superiority; p < .0001, Regression, Logistic; Odds Ratio (OR) = 2.28, 95% CI 2-sided [1.53 to 3.40]
Statistical Analysis 13: Comparison: Placebo vs Tanezumab 2.5 mg; Week 4, >=70%: Odds ratio and 95%CI estimated from logistic regression model. Logistic regression model included baseline WOMAC physical function subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p = 0.0107, Regression, Logistic; Odds Ratio (OR) = 2.23, 95% CI 2-sided [1.21 to 4.14]
Statistical Analysis 14: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 13, analysis 13]; Test type: Superiority; p = 0.0126, Regression, Logistic; Odds Ratio (OR) = 2.18, 95% CI 2-sided [1.18 to 4.02]
Statistical Analysis 15: Comparison: Placebo vs Tanezumab 2.5 mg; Week 4, >=90%: Odds ratio and 95%CI estimated from logistic regression model. Logistic regression model included baseline WOMAC physical function subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p = 0.1516, Regression, Logistic; Odds Ratio (OR) = 2.67, 95% CI 2-sided [0.70 to 10.26]
Statistical Analysis 16: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 13, analysis 15]; Test type: Superiority; p = 0.0210, Regression, Logistic; Odds Ratio (OR) = 4.49, 95% CI 2-sided [1.25 to 16.05]
Statistical Analysis 17: Comparison: Placebo vs Tanezumab 2.5 mg; Week 8, >=30%: Odds ratio and 95%CI estimated from logistic regression model. Logistic regression model included baseline WOMAC physical function subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p = 0.0034, Regression, Logistic; Odds Ratio (OR) = 1.65, 95% CI 2-sided [1.18 to 2.31]
Statistical Analysis 18: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 13, analysis 17]; Test type: Superiority; p = 0.0010, Regression, Logistic; Odds Ratio (OR) = 1.75, 95% CI 2-sided [1.26 to 2.45]
Statistical Analysis 19: Comparison: Placebo vs Tanezumab 2.5 mg; Week 8, >=50%: Odds ratio and 95%CI estimated from logistic regression model. Logistic regression model included baseline WOMAC physical function subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p = 0.0014, Regression, Logistic; Odds Ratio (OR) = 1.86, 95% CI 2-sided [1.27 to 2.71]
Statistical Analysis 20: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 13, analysis 19]; Test type: Superiority; p < .0001, Regression, Logistic; Odds Ratio (OR) = 2.13, 95% CI 2-sided [1.46 to 3.10]
Statistical Analysis 21: Comparison: Placebo vs Tanezumab 2.5 mg; Week 8, >=70%: Odds ratio and 95%CI estimated from logistic regression model. Logistic regression model included baseline WOMAC physical function subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p = 0.0007, Regression, Logistic; Odds Ratio (OR) = 2.61, 95% CI 2-sided [1.49 to 4.55]
Statistical Analysis 22: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 13, analysis 21]; Test type: Superiority; p = 0.0018, Regression, Logistic; Odds Ratio (OR) = 2.43, 95% CI 2-sided [1.39 to 4.24]
Statistical Analysis 23: Comparison: Placebo vs Tanezumab 2.5 mg; Week 8, >=90%: Odds ratio and 95%CI estimated from logistic regression model. Logistic regression model included baseline WOMAC physical function subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p = 0.0150, Regression, Logistic; Odds Ratio (OR) = 4.10, 95% CI 2-sided [1.31 to 12.79]
Statistical Analysis 24: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 13, analysis 23]; Test type: Superiority; p = 0.0211, Regression, Logistic; Odds Ratio (OR) = 3.79, 95% CI 2-sided [1.22 to 11.78]
Statistical Analysis 25: Comparison: Placebo vs Tanezumab 2.5 mg; Week 12, >=30%: Odds ratio and 95%CI estimated from logistic regression model. Logistic regression model included baseline WOMAC physical function subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p < .0001, Regression, Logistic; Odds Ratio (OR) = 2.01, 95% CI 2-sided [1.43 to 2.84]
Statistical Analysis 26: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 13, analysis 25]; Test type: Superiority; p < .0001, Regression, Logistic; Odds Ratio (OR) = 2.19, 95% CI 2-sided [1.55 to 3.10]
Statistical Analysis 27: Comparison: Placebo vs Tanezumab 2.5 mg; Week 12, >=50%: Odds ratio and 95%CI estimated from logistic regression model. Logistic regression model included baseline WOMAC physical function subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p < .0001, Regression, Logistic; Odds Ratio (OR) = 2.10, 95% CI 2-sided [1.47 to 3.00]
Statistical Analysis 28: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 13, analysis 27]; Test type: Superiority; p < .0001, Regression, Logistic; Odds Ratio (OR) = 2.08, 95% CI 2-sided [1.46 to 2.96]
Statistical Analysis 29: Comparison: Placebo vs Tanezumab 2.5 mg; Week 12, >=70%: Odds ratio and 95%CI estimated from logistic regression model. Logistic regression model included baseline WOMAC physical function subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p = 0.0180, Regression, Logistic; Odds Ratio (OR) = 1.74, 95% CI 2-sided [1.10 to 2.76]
Statistical Analysis 30: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 13, analysis 29]; Test type: Superiority; p = 0.0072, Regression, Logistic; Odds Ratio (OR) = 1.86, 95% CI 2-sided [1.18 to 2.94]
Statistical Analysis 31: Comparison: Placebo vs Tanezumab 2.5 mg; Week 12, >=90%: Odds ratio and 95%CI estimated from logistic regression model. Logistic regression model included baseline WOMAC physical function subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p = 0.0015, Regression, Logistic; Odds Ratio (OR) = 10.84, 95% CI 2-sided [2.49 to 47.22]
Statistical Analysis 32: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 13, analysis 31]; Test type: Superiority; p = 0.0044, Regression, Logistic; Odds Ratio (OR) = 8.62, 95% CI 2-sided [1.96 to 37.96]
Statistical Analysis 33: Comparison: Placebo vs Tanezumab 2.5 mg; Week 16, >=30%: Odds ratio and 95%CI estimated from logistic regression model. Logistic regression model included baseline WOMAC physical function subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p = 0.0018, Regression, Logistic; Odds Ratio (OR) = 1.72, 95% CI 2-sided [1.22 to 2.43]
Statistical Analysis 34: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 13, analysis 33]; Test type: Superiority; p = 0.0011, Regression, Logistic; Odds Ratio (OR) = 1.77, 95% CI 2-sided [1.26 to 2.50]
Statistical Analysis 35: Comparison: Placebo vs Tanezumab 2.5 mg; Week 16, >=50%: Odds ratio and 95%CI estimated from logistic regression model. Logistic regression model included baseline WOMAC physical function subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p = 0.0035, Regression, Logistic; Odds Ratio (OR) = 1.68, 95% CI 2-sided [1.19 to 2.38]
Statistical Analysis 36: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 13, analysis 35]; Test type: Superiority; p = 0.0022, Regression, Logistic; Odds Ratio (OR) = 1.72, 95% CI 2-sided [1.22 to 2.43]
Statistical Analysis 37: Comparison: Placebo vs Tanezumab 2.5 mg; Week 16, >=70%: Odds ratio and 95%CI estimated from logistic regression model. Logistic regression model included baseline WOMAC physical function subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p = 0.0155, Regression, Logistic; Odds Ratio (OR) = 1.74, 95% CI 2-sided [1.11 to 2.72]
Statistical Analysis 38: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 13, analysis 37]; Test type: Superiority; p = 0.1549, Regression, Logistic; Odds Ratio (OR) = 1.39, 95% CI 2-sided [0.88 to 2.20]
Statistical Analysis 39: Comparison: Placebo vs Tanezumab 2.5 mg; Week 16, >=90%: Odds ratio and 95%CI estimated from logistic regression model. Logistic regression model included baseline WOMAC physical function subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p = 0.0212, Regression, Logistic; Odds Ratio (OR) = 2.94, 95% CI 2-sided [1.18 to 7.37]
Statistical Analysis 40: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 13, analysis 39]; Test type: Superiority; p = 0.0373, Regression, Logistic; Odds Ratio (OR) = 2.64, 95% CI 2-sided [1.06 to 6.57]
Statistical Analysis 41: Comparison: Placebo vs Tanezumab 2.5 mg; Week 24, >=30%: Odds ratio and 95%CI estimated from logistic regression model. Logistic regression model included baseline WOMAC physical function subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p = 0.0006, Regression, Logistic; Odds Ratio (OR) = 1.83, 95% CI 2-sided [1.29 to 2.57]
Statistical Analysis 42: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 13, analysis 41]; Test type: Superiority; p < .0001, Regression, Logistic; Odds Ratio (OR) = 2.13, 95% CI 2-sided [1.51 to 3.02]
Statistical Analysis 43: Comparison: Placebo vs Tanezumab 2.5 mg; Week 24, >=50%: Odds ratio and 95%CI estimated from logistic regression model. Logistic regression model included baseline WOMAC physical function subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p = 0.0152, Regression, Logistic; Odds Ratio (OR) = 1.54, 95% CI 2-sided [1.09 to 2.18]
Statistical Analysis 44: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 13, analysis 43]; Test type: Superiority; p = 0.0018, Regression, Logistic; Odds Ratio (OR) = 1.73, 95% CI 2-sided [1.23 to 2.45]
Statistical Analysis 45: Comparison: Placebo vs Tanezumab 2.5 mg; Week 24, >=70%: Odds ratio and 95%CI estimated from logistic regression model. Logistic regression model included baseline WOMAC physical function subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p = 0.0970, Regression, Logistic; Odds Ratio (OR) = 1.47, 95% CI 2-sided [0.93 to 2.31]
Statistical Analysis 46: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 13, analysis 45]; Test type: Superiority; p = 0.3435, Regression, Logistic; Odds Ratio (OR) = 1.25, 95% CI 2-sided [0.79 to 1.98]
Statistical Analysis 47: Comparison: Placebo vs Tanezumab 2.5 mg; Week 24, >=90%: Odds ratio and 95%CI estimated from logistic regression model. Logistic regression model included baseline WOMAC physical function subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p = 0.0236, Regression, Logistic; Odds Ratio (OR) = 3.30, 95% CI 2-sided [1.17 to 9.27]
Statistical Analysis 48: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 13, analysis 47]; Test type: Superiority; p = 0.0296, Regression, Logistic; Odds Ratio (OR) = 3.14, 95% CI 2-sided [1.12 to 8.81]

14. Secondary Outcome: Percentage of Participants With Cumulative Percent Change From Baseline Reduction in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Physical Function Subscale at Weeks 16 and 24
Description: Percentage of participants with cumulative reduction (as percent) (greater than 0 %; >= 10 %, 20 %, 30 %, 40 %, 50 %, 60 %, 70 %, 80 % and 90%; =100 %) in WOMAC physical function subscale from Baseline to Weeks 16 and 24 were reported. WOMAC:Self-administered, disease-specific questionnaire which assesses clinically important, participant-relevant symptoms for pain, stiffness and physical function in participants with OA. Physical function: participant's ability to move around and perform usual activities of daily living. WOMAC physical function subscale:17-item questionnaire to assess the degree of difficulty experienced due to OA in index joint (knee or hip) during past 48 hours, calculated as mean of the scores from 17 individual questions scored on a NRS. Scores for each question and WOMAC Pain subscale on NRS ranged from 0 (no difficulty) to 10 (extreme difficulty), higher scores indicate extreme difficulty/worse physical function. Missing data was imputed using mixed BOCF/LOCF.
Time Frame: Baseline, Weeks 16 and 24
Population: as for outcome 11
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg
Number analyzed (Participants) | 281 | 282 | 284
percentage of participants
  Week 16: >=0% | 84.7 | 93.6 | 93.0
  Week 16: >=10% | 75.1 | 87.2 | 83.8
  Week 16: >=20% | 61.6 | 73.8 | 73.9
  Week 16: >=30% | 53.0 | 65.2 | 66.2
  Week 16: >=40% | 44.1 | 55.3 | 56.0
  Week 16: >=50% | 32.0 | 42.9 | 44.0
  Week 16: >=60% | 20.3 | 30.1 | 30.3
  Week 16: >=70% | 14.2 | 21.3 | 18.3
  Week 16: >=80% | 7.1 | 12.4 | 11.3
  Week 16: >=90% | 2.5 | 6.0 | 6.0
  Week 16: =100% | 0.7 | 0.7 | 1.8
  Week 24: >=0% | 79.7 | 89.0 | 90.1
  Week 24: >=10% | 70.1 | 85.8 | 84.2
  Week 24: >=20% | 61.6 | 74.8 | 78.2
  Week 24: >=30% | 51.2 | 64.9 | 68.7
  Week 24: >=40% | 41.3 | 51.1 | 57.0
  Week 24: >=50% | 32.4 | 41.5 | 44.7
  Week 24: >=60% | 21.0 | 30.9 | 30.6
  Week 24: >=70% | 14.6 | 19.1 | 17.3
  Week 24: >=80% | 6.4 | 10.6 | 10.2
  Week 24: >=90% | 1.8 | 5.3 | 5.3
  Week 24: =100% | 0 | 0.4 | 1.8

15. Secondary Outcome: Percentage of Participants Achieving Improvement of >=2 Points in Patient's Global Assessment (PGA) of Osteoarthritis
Description: PGA of OA was assessed by asking a question from participants: "Considering all the ways your osteoarthritis in your knee or hip affects you, how are you doing today?" Participants responded on a scale ranging from 1-5, where, 1=very good (no symptom and no limitation of normal activities), 2= good (mild symptoms and no limitation of normal activities), 3= fair (moderate symptoms and limitation of some normal activities), 4= poor (severe symptoms and inability to carry out most normal activities), and 5 = very poor (very severe symptoms and inability to carry out all normal activities). Higher scores indicated worse condition. Percentage of participants with improvement of at least 2 points from Baseline in PGA of OA were reported. Missing data was imputed using mixed BOCF/LOCF.
Time Frame: Weeks 2, 4, 8, 12, 16, 24 and 32
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg
Number analyzed (Participants) | 281 | 282 | 284
percentage of participants
  Week 2 | 8.5 | 15.6 | 12.0
  Week 4 | 8.5 | 17.7 | 19.0
  Week 8 | 12.8 | 21.3 | 21.8
  Week 12 | 14.6 | 26.2 | 28.5
  Week 16 | 14.6 | 22.7 | 27.1
  Week 24 | 17.4 | 24.1 | 25.7
  Week 32: number analyzed (Participants) | 231 | 247 | 246
  Week 32 | 19.9 | 14.2 | 15.4
Statistical Analysis 1: Comparison: Placebo vs Tanezumab 2.5 mg; Week 2: Odds ratio and 95% CI estimated from logistic regression model. Logistic regression model included baseline patient global assessment of osteoarthritis scale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p = 0.0132, Regression, Logistic; Odds Ratio (OR) = 2.14, 95% CI 2-sided [1.17 to 3.90]
Statistical Analysis 2: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 15, analysis 1]; Test type: Superiority; p = 0.1274, Regression, Logistic; Odds Ratio (OR) = 1.62, 95% CI 2-sided [0.87 to 3.02]
Statistical Analysis 3: Comparison: Placebo vs Tanezumab 2.5 mg; Week 4: Odds ratio and 95% CI estimated from logistic regression model. Logistic regression model included baseline patient global assessment of osteoarthritis scale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p = 0.0016, Regression, Logistic; Odds Ratio (OR) = 2.62, 95% CI 2-sided [1.44 to 4.76]
Statistical Analysis 4: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 15, analysis 3]; Test type: Superiority; p < .0001, Regression, Logistic; Odds Ratio (OR) = 3.34, 95% CI 2-sided [1.84 to 6.03]
Statistical Analysis 5: Comparison: Placebo vs Tanezumab 2.5 mg; Week 8: Odds ratio and 95% CI estimated from logistic regression model. Logistic regression model included baseline patient global assessment of osteoarthritis scale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p = 0.0089, Regression, Logistic; Odds Ratio (OR) = 2.04, 95% CI 2-sided [1.20 to 3.49]
Statistical Analysis 6: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 15, analysis 5]; Test type: Superiority; p = 0.0012, Regression, Logistic; Odds Ratio (OR) = 2.41, 95% CI 2-sided [1.42 to 4.10]
Statistical Analysis 7: Comparison: Placebo vs Tanezumab 2.5 mg; Week 12: Odds ratio and 95% CI estimated from logistic regression model. Logistic regression model included baseline patient global assessment of osteoarthritis scale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p = 0.0006, Regression, Logistic; Odds Ratio (OR) = 2.40, 95% CI 2-sided [1.45 to 3.98]
Statistical Analysis 8: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 15, analysis 7]; Test type: Superiority; p < .0001, Regression, Logistic; Odds Ratio (OR) = 3.16, 95% CI 2-sided [1.92 to 5.21]
Statistical Analysis 9: Comparison: Placebo vs Tanezumab 2.5 mg; Week 16: Odds ratio and 95% CI estimated from logistic regression model. Logistic regression model included baseline patient global assessment of osteoarthritis scale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p = 0.0203, Regression, Logistic; Odds Ratio (OR) = 1.83, 95% CI 2-sided [1.10 to 3.06]
Statistical Analysis 10: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 15, analysis 9]; Test type: Superiority; p < .0001, Regression, Logistic; Odds Ratio (OR) = 2.94, 95% CI 2-sided [1.77 to 4.86]
Statistical Analysis 11: Comparison: Placebo vs Tanezumab 2.5 mg; Week 24: Odds ratio and 95% CI estimated from logistic regression model. Logistic regression model included baseline patient global assessment of osteoarthritis scale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p = 0.0775, Regression, Logistic; Odds Ratio (OR) = 1.56, 95% CI 2-sided [0.95 to 2.55]
Statistical Analysis 12: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 15, analysis 11]; Test type: Superiority; p = 0.0064, Regression, Logistic; Odds Ratio (OR) = 1.97, 95% CI 2-sided [1.21 to 3.21]

16. Secondary Outcome: Change From Baseline for Average Pain Score in the Index Joint at Weeks 1, 2, 3, 4, 6, 8, 10, 12, 16, 20 and 24
Description: Participants assessed their average pain in the index hip/knee in the past 24 hours using a scale ranging from 0 (no pain) to 10 (worst possible pain). Higher scores indicated higher pain. Data represents averages of the values reported during the 8-week interval up to and including the given week. Change from baseline was calculated using the difference between each post-baseline weekly mean and the baseline mean score.
Time Frame: Baseline, Weeks 1, 2, 3, 4, 6, 8, 10, 12, 16, 20 and 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg
Number analyzed (Participants) | 282 | 283 | 284
units on a scale
  Change at Week 1 | -0.57 (0.11) | -1.06 (0.11) | -0.93 (0.11)
  Change at Week 2 | -0.98 (0.14) | -1.72 (0.14) | -1.49 (0.14)
  Change at Week 3 | -1.19 (0.15) | -1.97 (0.15) | -1.67 (0.15)
  Change at Week 4 | -1.37 (0.15) | -2.28 (0.15) | -2.13 (0.15)
  Change at Week 6 | -1.48 (0.16) | -2.38 (0.16) | -2.43 (0.16)
  Change at Week 8 | -1.57 (0.16) | -2.19 (0.16) | -2.39 (0.16)
  Change at Week 10 | -1.79 (0.17) | -2.51 (0.17) | -2.56 (0.17)
  Change at Week 12 | -1.84 (0.17) | -2.57 (0.17) | -2.64 (0.17)
  Change at Week 16 | -1.98 (0.18) | -2.50 (0.17) | -2.61 (0.17)
  Change at Week 20 | -2.17 (0.18) | -2.87 (0.18) | -2.86 (0.18)
  Change at Week 24 | -2.21 (0.19) | -2.60 (0.18) | -2.73 (0.18)
Statistical Analysis 1: Comparison: Placebo vs Tanezumab 2.5 mg; Week 1: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets includes treatment, randomization stratification variables (index joint and highest Kellgren-Lawrence grade) as fixed effects, baseline pain in the index joint as covariate, and study site as a random effect; Test type: Superiority; p < .0001, ANCOVA; Least Square Mean Difference = -0.49, 95% CI 2-sided [-0.70 to -0.27], Standard Error of Mean 0.11
Statistical Analysis 2: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 16, analysis 1]; Test type: Superiority; p = 0.0009, ANCOVA; Least Square Mean Difference = -0.36, 95% CI 2-sided [-0.58 to -0.15], Standard Error of Mean 0.11
Statistical Analysis 3: Comparison: Placebo vs Tanezumab 2.5 mg; Week 2: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets includes treatment, randomization stratification variables (index joint and highest Kellgren-Lawrence grade) as fixed effects, baseline pain in the index joint as covariate, and study site as a random effect; Test type: Superiority; p < .0001, ANCOVA; Least Square Mean Difference = -0.74, 95% CI 2-sided [-1.00 to -0.48], Standard Error of Mean 0.13
Statistical Analysis 4: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 16, analysis 3]; Test type: Superiority; p = 0.0001, ANCOVA; Least Square Mean Difference = -0.51, 95% CI 2-sided [-0.77 to -0.25], Standard Error of Mean 0.13
Statistical Analysis 5: Comparison: Placebo vs Tanezumab 2.5 mg; Week 3: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets includes treatment, randomization stratification variables (index joint and highest Kellgren-Lawrence grade) as fixed effects, baseline pain in the index joint as covariate, and study site as a random effect; Test type: Superiority; p < .0001, ANCOVA; Least Square Mean Difference = -0.78, 95% CI 2-sided [-1.06 to -0.50], Standard Error of Mean 0.14
Statistical Analysis 6: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 16, analysis 5]; Test type: Superiority; p = 0.0006, ANCOVA; Least Square Mean Difference = -0.49, 95% CI 2-sided [-0.77 to -0.21], Standard Error of Mean 0.14
Statistical Analysis 7: Comparison: Placebo vs Tanezumab 2.5 mg; Week 4: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets includes treatment, randomization stratification variables (index joint and highest Kellgren-Lawrence grade) as fixed effects, baseline pain in the index joint as covariate, and study site as a random effect; Test type: Superiority; p < .0001, ANCOVA; Least Square Mean Difference = -0.91, 95% CI 2-sided [-1.20 to -0.62], Standard Error of Mean 0.15
Statistical Analysis 8: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 16, analysis 7]; Test type: Superiority; p < .0001, ANCOVA; Least Square Mean Difference = -0.77, 95% CI 2-sided [-1.06 to -0.47], Standard Error of Mean 0.15
Statistical Analysis 9: Comparison: Placebo vs Tanezumab 2.5 mg; Week 6: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets includes treatment, randomization stratification variables (index joint and highest Kellgren-Lawrence grade) as fixed effects, baseline pain in the index joint as covariate, and study site as a random effect; Test type: Superiority; p < .0001, ANCOVA; Least Square Mean Difference = -0.90, 95% CI 2-sided [-1.20 to -0.59], Standard Error of Mean 0.16
Statistical Analysis 10: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 16, analysis 9]; Test type: Superiority; p < .0001, ANCOVA; Least Square Mean Difference = -0.95, 95% CI 2-sided [-1.25 to -0.64], Standard Error of Mean 0.16
Statistical Analysis 11: Comparison: Placebo vs Tanezumab 2.5 mg; Week 8: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets includes treatment, randomization stratification variables (index joint and highest Kellgren-Lawrence grade) as fixed effects, baseline pain in the index joint as covariate, and study site as a random effect; Test type: Superiority; p = 0.0001, ANCOVA; Least Square Mean Difference = -0.61, 95% CI 2-sided [-0.93 to -0.30], Standard Error of Mean 0.16
Statistical Analysis 12: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 16, analysis 11]; Test type: Superiority; p < .0001, ANCOVA; Least Square Mean Difference = -0.81, 95% CI 2-sided [-1.13 to -0.50], Standard Error of Mean 0.16
Statistical Analysis 13: Comparison: Placebo vs Tanezumab 2.5 mg; Week 10: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets includes treatment, randomization stratification variables (index joint and highest Kellgren-Lawrence grade) as fixed effects, baseline pain in the index joint as covariate, and study site as a random effect; Test type: Superiority; p < .0001, ANCOVA; Least Square Mean Difference = -0.72, 95% CI 2-sided [-1.05 to -0.39], Standard Error of Mean 0.17
Statistical Analysis 14: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 16, analysis 13]; Test type: Superiority; p < .0001, ANCOVA; Least Square Mean Difference = -0.77, 95% CI 2-sided [-1.10 to -0.44], Standard Error of Mean 0.17
Statistical Analysis 15: Comparison: Placebo vs Tanezumab 2.5 mg; Week 12: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets includes treatment, randomization stratification variables (index joint and highest Kellgren-Lawrence grade) as fixed effects, baseline pain in the index joint as covariate, and study site as a random effect; Test type: Superiority; p < .0001, ANCOVA; Least Square Mean Difference = -0.73, 95% CI 2-sided [-1.06 to -0.39], Standard Error of Mean 0.17
Statistical Analysis 16: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 16, analysis 15]; Test type: Superiority; p < .0001, ANCOVA; Least Square Mean Difference = -0.80, 95% CI 2-sided [-1.13 to -0.46], Standard Error of Mean 0.17
Statistical Analysis 17: Comparison: Placebo vs Tanezumab 2.5 mg; Week 16: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets includes treatment, randomization stratification variables (index joint and highest Kellgren-Lawrence grade) as fixed effects, baseline pain in the index joint as covariate, and study site as a random effect; Test type: Superiority; p = 0.0040, ANCOVA; Least Square Mean Difference = -0.52, 95% CI 2-sided [-0.87 to -0.16], Standard Error of Mean 0.18
Statistical Analysis 18: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 16, analysis 17]; Test type: Superiority; p = 0.0005, ANCOVA; Least Square Mean Difference = -0.63, 95% CI 2-sided [-0.98 to -0.27], Standard Error of Mean 0.18
Statistical Analysis 19: Comparison: Placebo vs Tanezumab 2.5 mg; Week 20: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets includes treatment, randomization stratification variables (index joint and highest Kellgren-Lawrence grade) as fixed effects, baseline pain in the index joint as covariate, and study site as a random effect; Test type: Superiority; p = 0.0002, ANCOVA; Least Square Mean Difference = -0.70, 95% CI 2-sided [-1.06 to -0.33], Standard Error of Mean 0.19
Statistical Analysis 20: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 16, analysis 19]; Test type: Superiority; p = 0.0002, ANCOVA; Least Square Mean Difference = -0.68, 95% CI 2-sided [-1.05 to -0.32], Standard Error of Mean 0.19
Statistical Analysis 21: Comparison: Placebo vs Tanezumab 2.5 mg; Week 24: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets includes treatment, randomization stratification variables (index joint and highest Kellgren-Lawrence grade) as fixed effects, baseline pain in the index joint as covariate, and study site as a random effect; Test type: Superiority; p = 0.0506, ANCOVA; Least Square Mean Difference = -0.39, 95% CI 2-sided [-0.78 to 0.00], Standard Error of Mean 0.20
Statistical Analysis 22: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 16, analysis 21]; Test type: Superiority; p = 0.0086, ANCOVA; Least Square Mean Difference = -0.52, 95% CI 2-sided [-0.91 to -0.13], Standard Error of Mean 0.20

17. Secondary Outcome: Change From Baseline for Average Pain Score in the Index Joint at Weeks 28 and 32
Description: as for outcome 16
Time Frame: Baseline, Weeks 28 and 32
Population: The intent to treat population included all randomized participants who received at least one dose of subcutaneous study medication (either tanezumab or placebo). Here, 'Number analyzed' = Participants evaluable for this outcome measure at specified time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg
Number analyzed (Participants) | 282 | 283 | 284
units on a scale
  Baseline: number analyzed (Participants) | 278 | 280 | 280
  Baseline | 6.79 (1.56) | 7.03 (1.38) | 6.90 (1.43)
  Change at Week 28: number analyzed (Participants) | 239 | 260 | 254
  Change at Week 28 | -2.26 (2.27) | -2.63 (2.32) | -2.58 (2.33)
  Change at Week 32: number analyzed (Participants) | 226 | 250 | 245
  Change at Week 32 | -2.19 (2.40) | -2.07 (2.33) | -2.13 (2.40)

18. Secondary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Stiffness Subscale at Weeks 2, 4, 8, 12, 16 and 24
Description: WOMAC: self-administered, disease-specific questionnaire which assesses clinically important, participant-relevant symptoms for pain, stiffness and physical function in participants with OA. Stiffness was defined as a sensation of decreased ease of movement in the index joint (knee or hip). The WOMAC stiffness subscale is a 2-item questionnaire used to assess the amount of stiffness experienced due to OA in the index joint (knee or hip) during the past 48 hours. It was calculated as the mean of scores from 2 individual questions scored on NRS. Scores for each question and WOMAC stiffness subscale score on NRS ranged from 0 (no stiffness) to 10 (extreme stiffness), where higher scores indicated higher stiffness.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16 and 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg
Number analyzed (Participants) | 282 | 283 | 284
units on a scale
  Change at Week 2 | -1.25 (0.15) | -2.03 (0.15) | -1.90 (0.15)
  Change at Week 4 | -1.90 (0.16) | -2.62 (0.16) | -2.74 (0.16)
  Change at Week 8 | -1.82 (0.17) | -2.41 (0.17) | -2.81 (0.17)
  Change at Week 12 | -2.10 (0.18) | -2.90 (0.17) | -2.95 (0.17)
  Change at Week 16 | -2.00 (0.18) | -2.65 (0.18) | -2.77 (0.18)
  Change at Week 24 | -1.97 (0.19) | -2.59 (0.19) | -2.84 (0.19)
Statistical Analysis 1: Comparison: Placebo vs Tanezumab 2.5 mg; Week 2: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets includes treatment, randomization stratification variables (index joint and highest Kellgren-Lawrence grade) as fixed effects, baseline WOMAC stiffness subscales and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p < .0001, ANCOVA; Least Square Mean Difference = -0.77, 95% CI 2-sided [-1.07 to -0.48], Standard Error of Mean 0.15
Statistical Analysis 2: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 18, analysis 1]; Test type: Superiority; p < .0001, ANCOVA; Least Square Mean Difference = -0.64, 95% CI 2-sided [-0.94 to -0.35], Standard Error of Mean 0.15
Statistical Analysis 3: Comparison: Placebo vs Tanezumab 2.5 mg; Week 4: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets includes treatment, randomization stratification variables (index joint and highest Kellgren-Lawrence grade) as fixed effects, baseline WOMAC stiffness subscales and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p < .0001, ANCOVA; Least Square Mean Difference = -0.72, 95% CI 2-sided [-1.03 to -0.41], Standard Error of Mean 0.16
Statistical Analysis 4: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 18, analysis 3]; Test type: Superiority; p < .0001, ANCOVA; Least Square Mean Difference = -0.84, 95% CI 2-sided [-1.15 to -0.53], Standard Error of Mean 0.16
Statistical Analysis 5: Comparison: Placebo vs Tanezumab 2.5 mg; Week 8: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets includes treatment, randomization stratification variables (index joint and highest Kellgren-Lawrence grade) as fixed effects, baseline WOMAC stiffness subscales and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p = 0.0004, ANCOVA; Least Square Mean Difference = -0.58, 95% CI 2-sided [-0.91 to -0.26], Standard Error of Mean 0.17
Statistical Analysis 6: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 18, analysis 5]; Test type: Superiority; p < .0001, ANCOVA; Least Square Mean Difference = -0.99, 95% CI 2-sided [-1.31 to -0.67], Standard Error of Mean 0.16
Statistical Analysis 7: Comparison: Placebo vs Tanezumab 2.5 mg; Week 12: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets includes treatment, randomization stratification variables (index joint and highest Kellgren-Lawrence grade) as fixed effects, baseline WOMAC stiffness subscales and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p < .0001, ANCOVA; Least Square Mean Difference = -0.80, 95% CI 2-sided [-1.14 to -0.46], Standard Error of Mean 0.17
Statistical Analysis 8: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 18, analysis 7]; Test type: Superiority; p < .0001, ANCOVA; Least Square Mean Difference = -0.84, 95% CI 2-sided [-1.18 to -0.50], Standard Error of Mean 0.17
Statistical Analysis 9: Comparison: Placebo vs Tanezumab 2.5 mg; Week 16: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets includes treatment, randomization stratification variables (index joint and highest Kellgren-Lawrence grade) as fixed effects, baseline WOMAC stiffness subscales and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p = 0.0002, ANCOVA; Least Square Mean Difference = -0.65, 95% CI 2-sided [-1.00 to -0.30], Standard Error of Mean 0.18
Statistical Analysis 10: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 18, analysis 9]; Test type: Superiority; p < .0001, ANCOVA; Least Square Mean Difference = -0.77, 95% CI 2-sided [-1.12 to -0.43], Standard Error of Mean 0.18
Statistical Analysis 11: Comparison: Placebo vs Tanezumab 2.5 mg; [analysis description as in outcome 16, analysis 21]; Test type: Superiority; p = 0.0013, ANCOVA; Least Square Mean Difference = -0.62, 95% CI 2-sided [-0.99 to -0.24], Standard Error of Mean 0.19
Statistical Analysis 12: Comparison: Placebo vs Tanezumab 5 mg; Week 24: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets includes treatment, randomization stratification variables (index joint and highest Kellgren-Lawrence grade) as fixed effects, baseline WOMAC stiffness subscales and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p < .0001, ANCOVA; Least Square Mean Difference = -0.87, 95% CI 2-sided [-1.25 to -0.50], Standard Error of Mean 0.19

19. Secondary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Stiffness Subscale at Week 32
Description: WOMAC: self-administered, disease-specific questionnaire which assesses clinically important, participant-relevant symptoms for pain, stiffness and physical function in participants with OA. Stiffness was defined as a sensation of decreased ease of movement in the index joint (knee or hip). The WOMAC stiffness subscale is a 2-item questionnaire used to assess the amount of stiffness experienced due to OA in the index joint (knee or hip) during the past 48 hours. It was calculated as the mean of scores from 2 individual questions scored on a NRS. Scores for each question and WOMAC stiffness subscale score on NRS ranged from 0 (no stiffness) to 10 (extreme stiffness), where higher scores indicated higher stiffness.
Time Frame: Baseline, Week 32
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg
Number analyzed (Participants) | 282 | 283 | 284
units on a scale
  Baseline: number analyzed (Participants) | 281 | 282 | 284
  Baseline | 6.46 (1.43) | 6.44 (1.59) | 6.44 (1.53)
  Change at Week 32: number analyzed (Participants) | 231 | 247 | 246
  Change at Week 32 | -2.57 (2.22) | -2.34 (2.18) | -2.31 (2.51)

20. Secondary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Average Score at Weeks 2, 4, 8, 12, 16 and 24
Description: WOMAC: self-administered, disease-specific questionnaire which assesses clinically important, participant-relevant symptoms for pain, stiffness and physical function in participants with OA of index joint (knee or hip). WOMAC pain subscale assess amount of pain experienced (score: 0 [no pain] to 10 [extreme pain], higher score = more pain), WOMAC physical function subscale assess degree of difficulty experienced (score: 0 [no difficulty] to 10 [extreme difficulty], higher score = worse physical function) and WOMAC stiffness subscale assess the amount of stiffness experienced (score: 0 [no stiffness] to 10 [extreme stiffness], higher score = higher stiffness). WOMAC average score was the mean of WOMAC pain, physical function and stiffness subscale scores and ranges from 0 to 10, where higher scores indicated worse response.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16 and 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg
Number analyzed (Participants) | 282 | 283 | 284
units on a scale
  Change at Week 2 | -1.28 (0.13) | -1.99 (0.13) | -1.75 (0.13)
  Change at Week 4 | -1.80 (0.14) | -2.57 (0.14) | -2.60 (0.14)
  Change at Week 8 | -1.81 (0.15) | -2.42 (0.15) | -2.65 (0.15)
  Change at Week 12 | -2.11 (0.16) | -2.89 (0.16) | -2.92 (0.16)
  Change at Week 16 | -2.04 (0.17) | -2.67 (0.17) | -2.71 (0.16)
  Change at Week 24 | -2.11 (0.17) | -2.66 (0.17) | -2.83 (0.17)
Statistical Analysis 1: Comparison: Placebo vs Tanezumab 2.5 mg; Week 2: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets includes treatment, randomization stratification variables (index joint and highest Kellgren-Lawrence grade) as fixed effects, baseline WOMAC average scores and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p < .0001, ANCOVA; Least Square Mean Difference = -0.71, 95% CI 2-sided [-0.96 to -0.45], Standard Error of Mean 0.13
Statistical Analysis 2: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 20, analysis 1]; Test type: Superiority; p = 0.0004, ANCOVA; Least Square Mean Difference = -0.47, 95% CI 2-sided [-0.73 to -0.21], Standard Error of Mean 0.13
Statistical Analysis 3: Comparison: Placebo vs Tanezumab 2.5 mg; Week 4: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets includes treatment, randomization stratification variables (index joint and highest Kellgren-Lawrence grade) as fixed effects, baseline WOMAC average scores and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p < .0001, ANCOVA; Least Square Mean Difference = -0.77, 95% CI 2-sided [-1.04 to -0.49], Standard Error of Mean 0.14
Statistical Analysis 4: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 20, analysis 3]; Test type: Superiority; p < .0001, ANCOVA; Least Square Mean Difference = -0.80, 95% CI 2-sided [-1.08 to -0.53], Standard Error of Mean 0.14
Statistical Analysis 5: Comparison: Placebo vs Tanezumab 2.5 mg; Week 8: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets includes treatment, randomization stratification variables (index joint and highest Kellgren-Lawrence grade) as fixed effects, baseline WOMAC average scores and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p < .0001, ANCOVA; Least Square Mean Difference = -0.61, 95% CI 2-sided [-0.90 to -0.32], Standard Error of Mean 0.15
Statistical Analysis 6: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 20, analysis 5]; Test type: Superiority; p < .0001, ANCOVA; Least Square Mean Difference = -0.84, 95% CI 2-sided [-1.13 to -0.56], Standard Error of Mean 0.15
Statistical Analysis 7: Comparison: Placebo vs Tanezumab 2.5 mg; Week 12: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets includes treatment, randomization stratification variables (index joint and highest Kellgren-Lawrence grade) as fixed effects, baseline WOMAC average scores and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p < .0001, ANCOVA; Least Square Mean Difference = -0.78, 95% CI 2-sided [-1.09 to -0.47], Standard Error of Mean 0.16
Statistical Analysis 8: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 20, analysis 7]; Test type: Superiority; p < .0001, ANCOVA; Least Square Mean Difference = -0.81, 95% CI 2-sided [-1.12 to -0.50], Standard Error of Mean 0.16
Statistical Analysis 9: Comparison: Placebo vs Tanezumab 2.5 mg; Week 16: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets includes treatment, randomization stratification variables (index joint and highest Kellgren-Lawrence grade) as fixed effects, baseline WOMAC average scores and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p = 0.0001, ANCOVA; Least Square Mean Difference = -0.63, 95% CI 2-sided [-0.95 to -0.35], Standard Error of Mean 0.16
Statistical Analysis 10: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 20, analysis 9]; Test type: Superiority; p < .0001, ANCOVA; Least Square Mean Difference = -0.67, 95% CI 2-sided [-0.99 to -0.35], Standard Error of Mean 0.16
Statistical Analysis 11: Comparison: Placebo vs Tanezumab 2.5 mg; Week 24: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets includes treatment, randomization stratification variables (index joint and highest Kellgren-Lawrence grade) as fixed effects, baseline WOMAC average scores and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p = 0.0015, ANCOVA; Least Square Mean Difference = -0.55, 95% CI 2-sided [-0.89 to -0.21], Standard Error of Mean 0.17
Statistical Analysis 12: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 20, analysis 11]; Test type: Superiority; p < .0001, ANCOVA; Least Square Mean Difference = -0.73, 95% CI 2-sided [-1.07 to -0.39], Standard Error of Mean 0.17

21. Secondary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Average Score at Week 32
Description: as for outcome 20
Time Frame: Baseline, Week 32
Population: The intent to treat population included all randomized participants who received at least one dose of subcutaneous study medication (either tanezumab or placebo).Here, 'Number analyzed' = Participants evaluable for this outcome measure at specified time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg
Number analyzed (Participants) | 282 | 283 | 284
units on a scale
  Baseline: number analyzed (Participants) | 281 | 282 | 284
  Baseline | 6.57 (0.90) | 6.63 (0.96) | 6.60 (0.91)
  Change at Week 32: number analyzed (Participants) | 231 | 247 | 246
  Change at Week 32 | -2.61 (1.96) | -2.28 (1.87) | -2.27 (2.12)

22. Secondary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale Item (Pain When Walking on a Flat Surface) at Weeks 2, 4, 8, 12, 16 and 24
Description: WOMAC: self-administered, disease-specific questionnaire which assesses clinically important, participant-relevant symptoms for pain, stiffness and physical function in participants with OA in index joint (knee or hip). Participants answered a question: "How much pain have you had when walking on a flat surface?". Participants responded about the amount of pain they experienced when walking on a flat surface by using a NRS of 0 (no pain) to 10 (extreme pain), where higher scores indicated higher pain.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16 and 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg
Number analyzed (Participants) | 282 | 283 | 284
units on a scale
  Change at Week 2 | -1.27 (0.14) | -1.94 (0.14) | -1.64 (0.14)
  Change at Week 4 | -1.69 (0.15) | -2.51 (0.15) | -2.54 (0.15)
  Change at Week 8 | -1.77 (0.16) | -2.36 (0.15) | -2.49 (0.15)
  Change at Week 12 | -2.17 (0.17) | -2.91 (0.16) | -2.97 (0.16)
  Change at Week 16 | -2.06 (0.18) | -2.68 (0.17) | -2.66 (0.17)
  Change at Week 24 | -2.21 (0.18) | -2.61 (0.17) | -2.80 (0.17)
Statistical Analysis 1: Comparison: Placebo vs Tanezumab 2.5 mg; Week 2: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets includes treatment, randomization stratification variables (index joint and highest Kellgren-Lawrence grade) as fixed effects, baseline WOMAC pain when walking on a flat surface and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p < .0001, ANCOVA; Least Square Mean Difference = -0.67, 95% CI 2-sided [-0.96 to -0.38], Standard Error of Mean 0.15
Statistical Analysis 2: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 22, analysis 1]; Test type: Superiority; p = 0.0139, ANCOVA; Least Square Mean Difference = -0.37, 95% CI 2-sided [-0.67 to -0.08], Standard Error of Mean 0.15
Statistical Analysis 3: Comparison: Placebo vs Tanezumab 2.5 mg; Week 4: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets includes treatment, randomization stratification variables (index joint and highest Kellgren-Lawrence grade) as fixed effects, baseline WOMAC pain when walking on a flat surface and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p < .0001, ANCOVA; Least Square Mean Difference = -0.82, 95% CI 2-sided [-1.13 to -0.51], Standard Error of Mean 0.16
Statistical Analysis 4: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 22, analysis 3]; Test type: Superiority; p < .0001, ANCOVA; Least Square Mean Difference = -0.86, 95% CI 2-sided [-1.16 to -0.55], Standard Error of Mean 0.16
Statistical Analysis 5: Comparison: Placebo vs Tanezumab 2.5 mg; Week 8: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets includes treatment, randomization stratification variables (index joint and highest Kellgren-Lawrence grade) as fixed effects, baseline WOMAC pain when walking on a flat surface and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p = 0.0003, ANCOVA; Least Square Mean Difference = -0.59, 95% CI 2-sided [-0.91 to -0.27], Standard Error of Mean 0.16
Statistical Analysis 6: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 22, analysis 5]; Test type: Superiority; p < .0001, ANCOVA; Least Square Mean Difference = -0.72, 95% CI 2-sided [-1.04 to -0.40], Standard Error of Mean 0.16
Statistical Analysis 7: Comparison: Placebo vs Tanezumab 2.5 mg; Week 12: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets includes treatment, randomization stratification variables (index joint and highest Kellgren-Lawrence grade) as fixed effects, baseline WOMAC pain when walking on a flat surface and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p < .0001, ANCOVA; Least Square Mean Difference = -0.74, 95% CI 2-sided [-1.08 to -0.39], Standard Error of Mean 0.18
Statistical Analysis 8: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 22, analysis 7]; Test type: Superiority; p < .0001, ANCOVA; Least Square Mean Difference = -0.79, 95% CI 2-sided [-1.14 to -0.44], Standard Error of Mean 0.18
Statistical Analysis 9: Comparison: Placebo vs Tanezumab 2.5 mg; Week 16: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets includes treatment, randomization stratification variables (index joint and highest Kellgren-Lawrence grade) as fixed effects, baseline WOMAC pain when walking on a flat surface and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p = 0.0006, ANCOVA; Least Square Mean Difference = -0.62, 95% CI 2-sided [-0.98 to -0.27], Standard Error of Mean 0.18
Statistical Analysis 10: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 22, analysis 9]; Test type: Superiority; p = 0.0009, ANCOVA; Least Square Mean Difference = -0.60, 95% CI 2-sided [-0.96 to -0.25], Standard Error of Mean 0.18
Statistical Analysis 11: Comparison: Placebo vs Tanezumab 2.5 mg; Week 24: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets includes treatment, randomization stratification variables (index joint and highest Kellgren-Lawrence grade) as fixed effects, baseline WOMAC pain when walking on a flat surface and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p = 0.0377, ANCOVA; Least Square Mean Difference = -0.40, 95% CI 2-sided [-0.78 to -0.02], Standard Error of Mean 0.19
Statistical Analysis 12: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 22, analysis 11]; Test type: Superiority; p = 0.0019, ANCOVA; Least Square Mean Difference = -0.59, 95% CI 2-sided [-0.96 to -0.22], Standard Error of Mean 0.19

23. Secondary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale Item (Pain When Walking on a Flat Surface) at Week 32
Description: as for outcome 22
Time Frame: Baseline, Week 32
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg
Number analyzed (Participants) | 282 | 283 | 284
units on a scale
  Baseline: number analyzed (Participants) | 281 | 282 | 284
  Baseline | 6.73 (1.25) | 6.77 (1.27) | 6.79 (1.19)
  Change at Week 32: number analyzed (Participants) | 231 | 247 | 246
  Change at Week 32 | -2.46 (2.24) | -2.01 (2.10) | -1.99 (2.49)

24. Secondary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale Item (Pain When Going Up or Downstairs) at Weeks 2, 4, 8, 12, 16 and 24
Description: WOMAC: self-administered, disease-specific questionnaire which assesses clinically important, participant-relevant symptoms for pain, stiffness and physical function in participants with OA in index joint (knee or hip). Participants answered a question: "How much pain have you had when going up or down the stairs?" Participants responded about the amount of pain they experienced when going up or down stairs by using a NRS of 0 (no pain) to 10 (extreme pain), where higher scores indicated higher pain.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16 and 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg
Number analyzed (Participants) | 282 | 283 | 284
units on a scale
  Change at Week 2 | -1.39 (0.15) | -2.08 (0.15) | -1.96 (0.15)
  Change at Week 4 | -1.76 (0.16) | -2.73 (0.15) | -2.72 (0.15)
  Change at Week 8 | -1.72 (0.17) | -2.49 (0.17) | -2.74 (0.17)
  Change at Week 12 | -2.17 (0.18) | -2.92 (0.18) | -3.05 (0.18)
  Change at Week 16 | -2.06 (0.18) | -2.72 (0.18) | -2.83 (0.18)
  Change at Week 24 | -2.32 (0.19) | -2.76 (0.18) | -3.04 (0.18)
Statistical Analysis 1: Comparison: Placebo vs Tanezumab 2.5 mg; Week 2: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets includes treatment, randomization stratification variables (index joint and highest Kellgren-Lawrence grade) as fixed effects, baseline WOMAC pain when going up or down stairs and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p < .0001, ANCOVA; Least Square Mean Difference = -0.69, 95% CI 2-sided [-0.99 to -0.39], Standard Error of Mean 0.15
Statistical Analysis 2: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 24, analysis 1]; Test type: Superiority; p = 0.0002, ANCOVA; Least Square Mean Difference = -0.57, 95% CI 2-sided [-0.87 to -0.27], Standard Error of Mean 0.15
Statistical Analysis 3: Comparison: Placebo vs Tanezumab 2.5 mg; Week 4: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets includes treatment, randomization stratification variables (index joint and highest Kellgren-Lawrence grade) as fixed effects, baseline WOMAC pain when going up or down stairs and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p < .0001, ANCOVA; Least Square Mean Difference = -0.97, 95% CI 2-sided [-1.29 to -0.65], Standard Error of Mean 0.16
Statistical Analysis 4: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 24, analysis 3]; Test type: Superiority; p < .0001, ANCOVA; Least Square Mean Difference = -0.96, 95% CI 2-sided [-1.28 to -0.65], Standard Error of Mean 0.16
Statistical Analysis 5: Comparison: Placebo vs Tanezumab 2.5 mg; Week 8: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets includes treatment, randomization stratification variables (index joint and highest Kellgren-Lawrence grade) as fixed effects, baseline WOMAC pain when going up or down stairs and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p < .0001, ANCOVA; Least Square Mean Difference = -0.76, 95% CI 2-sided [-1.11 to -0.42], Standard Error of Mean 0.18
Statistical Analysis 6: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 24, analysis 5]; Test type: Superiority; p < .0001, ANCOVA; Least Square Mean Difference = -1.01, 95% CI 2-sided [-1.35 to -0.67], Standard Error of Mean 0.17
Statistical Analysis 7: Comparison: Placebo vs Tanezumab 2.5 mg; Week 12: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets includes treatment, randomization stratification variables (index joint and highest Kellgren-Lawrence grade) as fixed effects, baseline WOMAC pain when going up or down stairs and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p < .0001, ANCOVA; Least Square Mean Difference = -0.75, 95% CI 2-sided [-1.11 to -0.39], Standard Error of Mean 0.18
Statistical Analysis 8: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 24, analysis 7]; Test type: Superiority; p < .0001, ANCOVA; Least Square Mean Difference = -0.87, 95% CI 2-sided [-1.23 to -0.51], Standard Error of Mean 0.18
Statistical Analysis 9: Comparison: Placebo vs Tanezumab 2.5 mg; Week 16: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets includes treatment, randomization stratification variables (index joint and highest Kellgren-Lawrence grade) as fixed effects, baseline WOMAC pain when going up or down stairs and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p = 0.0005, ANCOVA; Least Square Mean Difference = -0.66, 95% CI 2-sided [-1.03 to -0.29], Standard Error of Mean 0.19
Statistical Analysis 10: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 24, analysis 9]; Test type: Superiority; p < .0001, ANCOVA; Least Square Mean Difference = -0.77, 95% CI 2-sided [-1.13 to -0.40], Standard Error of Mean 0.19
Statistical Analysis 11: Comparison: Placebo vs Tanezumab 2.5 mg; Week 24: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets includes treatment, randomization stratification variables (index joint and highest Kellgren-Lawrence grade) as fixed effects, baseline WOMAC pain when going up or down stairs and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p = 0.0246, ANCOVA; Least Square Mean Difference = -0.44, 95% CI 2-sided [-0.82 to -0.06], Standard Error of Mean 0.20
Statistical Analysis 12: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 24, analysis 11]; Test type: Superiority; p = 0.0003, ANCOVA; Least Square Mean Difference = -0.71, 95% CI 2-sided [-1.10 to -0.33], Standard Error of Mean 0.20

25. Secondary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale Item (Pain When Going Up or Downstairs) at Week 32
Description: as for outcome 24
Time Frame: Baseline, Week 32
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg
Number analyzed (Participants) | 282 | 283 | 284
units on a scale
  Baseline: number analyzed (Participants) | 281 | 282 | 284
  Baseline | 7.65 (1.13) | 7.79 (1.06) | 7.66 (1.18)
  Change at Week 32: number analyzed (Participants) | 231 | 247 | 246
  Change at Week 32 | -2.72 (2.32) | -2.23 (2.09) | -2.15 (2.41)

26. Secondary Outcome: Work Productivity and Activity Impairment Questionnaire for Osteoarthritis (WPAI:OA) Scores at Baseline
Description: WPAI is 6-question participant rated questionnaire to determine the impact of OA on absenteeism, presenteeism, work productivity, and daily activity impairment for a period of 7 days prior to a visit. It yields 4 sub-scores: work time missed (absenteeism), impairment while working (presenteeism), overall work impairment (work productivity) and activity impairment (daily activity impairment). These sub-scores are expressed as an impairment percentage (range from 0 to 100), with higher numbers indicating greater impairment and less productivity.
Time Frame: Baseline
Population: The intent to treat population included all randomized participants who received at least one dose of subcutaneous study medication (either tanezumab or placebo). Here, 'Number analyzed' = Participants evaluable for this outcome measure for specified categories.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg
Number analyzed (Participants) | 282 | 283 | 284
units on a scale
  Percent Work Time Missed: number analyzed (Participants) | 81 | 76 | 72
  Percent Work Time Missed | 9.7 (23.46) | 5.6 (18.33) | 6.9 (21.33)
  Percent Impairment While Working: number analyzed (Participants) | 78 | 74 | 69
  Percent Impairment While Working | 56.5 (22.26) | 58.9 (21.81) | 57.4 (18.44)
  Percent Overall Work Impairment: number analyzed (Participants) | 78 | 74 | 69
  Percent Overall Work Impairment | 59.3 (21.32) | 60.2 (21.20) | 58.3 (18.89)
  Percent Activity Impairment: number analyzed (Participants) | 277 | 278 | 283
  Percent Activity Impairment | 66.6 (13.35) | 67.7 (15.53) | 67.5 (13.26)

27. Secondary Outcome: Change From Baseline in Work Productivity and Activity Impairment Questionnaire for Osteoarthritis (WPAI:OA) Impairment Scores at Weeks 8, 16 and 24
Description: as for outcome 26
Time Frame: Baseline, Weeks 8, 16 and 24
Population: as for outcome 26
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg
Number analyzed (Participants) | 282 | 283 | 284
units on a scale
  Change at Week 8: Percent Work Time Missed: number analyzed (Participants) | 65 | 62 | 60
  Change at Week 8: Percent Work Time Missed | 0.04 (2.12) | 1.24 (2.12) | -2.05 (2.11)
  Change at Week 8:Percent Impairment While Working: number analyzed (Participants) | 64 | 60 | 57
  Change at Week 8:Percent Impairment While Working | -13.57 (3.11) | -20.26 (3.10) | -26.26 (3.12)
  Change at Week 8: Percent Overall Work Impairment: number analyzed (Participants) | 64 | 60 | 57
  Change at Week 8: Percent Overall Work Impairment | -13.78 (3.20) | -20.53 (3.18) | -26.26 (3.22)
  Change at Week 8: Percent Activity Impairment: number analyzed (Participants) | 268 | 272 | 281
  Change at Week 8: Percent Activity Impairment | -15.66 (1.55) | -21.84 (1.54) | -24.79 (1.53)
  Change at Week 16: Percent Work Time Missed: number analyzed (Participants) | 64 | 59 | 51
  Change at Week 16: Percent Work Time Missed | 2.36 (2.24) | 1.74 (2.29) | -2.16 (2.36)
  Change at Week 16:Percent Impairment While Working: number analyzed (Participants) | 61 | 58 | 50
  Change at Week 16:Percent Impairment While Working | -15.92 (3.28) | -26.23 (3.33) | -26.48 (3.42)
  Change at Week 16: Percent Overall Work Impairment: number analyzed (Participants) | 61 | 58 | 50
  Change at Week 16: Percent Overall Work Impairment | -16.38 (3.33) | -25.79 (3.37) | -26.42 (3.47)
  Change at Week 16: Percent Activity Impairment: number analyzed (Participants) | 254 | 261 | 270
  Change at Week 16: Percent Activity Impairment | -19.15 (1.77) | -25.16 (1.77) | -26.13 (1.74)
  Change at Week 24: Percent Work Time Missed: number analyzed (Participants) | 50 | 57 | 51
  Change at Week 24: Percent Work Time Missed | 4.09 (3.27) | 2.77 (3.18) | 1.16 (3.27)
  Change at Week 24:Percent Impairment While Working: number analyzed (Participants) | 47 | 55 | 48
  Change at Week 24:Percent Impairment While Working | -15.03 (3.86) | -19.31 (3.50) | -17.77 (3.74)
  Change at Week 24: Percent Overall Work Impairment: number analyzed (Participants) | 47 | 55 | 48
  Change at Week 24: Percent Overall Work Impairment | -15.17 (3.92) | -19.03 (3.56) | -17.29 (3.82)
  Change at Week 24: Percent Activity Impairment: number analyzed (Participants) | 231 | 252 | 254
  Change at Week 24: Percent Activity Impairment | -21.49 (1.84) | -24.57 (1.79) | -26.44 (1.79)
Statistical Analysis 1: Comparison: Placebo vs Tanezumab 2.5 mg; Week 8: Percent Work Time Missed: WPAI parameters were analyzed using ANCOVA model which included covariates of the corresponding baseline score, baseline diary average pain, index joint, highest Kellgren-Lawrence grade (2, 3 or 4), and treatment, with study site as a random effect; Test type: Superiority; p = 0.6427, ANCOVA; Least Square Mean Difference = 1.20, 95% CI 2-sided [-3.90 to 6.29], Standard Error of Mean 2.57
Statistical Analysis 2: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 27, analysis 1]; Test type: Superiority; p = 0.4208, ANCOVA; Least Square Mean Difference = -2.09, 95% CI 2-sided [-7.22 to 3.04], Standard Error of Mean 2.59
Statistical Analysis 3: Comparison: Placebo vs Tanezumab 2.5 mg; Week 16: Percent Work Time Missed: WPAI parameters were analyzed using ANCOVA model which included covariates of the corresponding baseline score, baseline diary average pain, index joint, highest Kellgren-Lawrence grade (2, 3 or 4), and treatment, with study site as a random effect; Test type: Superiority; p = 0.8204, ANCOVA; Least Square Mean Difference = -0.62, 95% CI 2-sided [-6.03 to 4.79], Standard Error of Mean 2.73
Statistical Analysis 4: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 27, analysis 3]; Test type: Superiority; p = 0.1157, ANCOVA; Least Square Mean Difference = -4.52, 95% CI 2-sided [-10.16 to 1.13], Standard Error of Mean 2.85
Statistical Analysis 5: Comparison: Placebo vs Tanezumab 2.5 mg; Week 24: Percent Work Time Missed: WPAI parameters were analyzed using ANCOVA model which included covariates of the corresponding baseline score, baseline diary average pain, index joint, highest Kellgren-Lawrence grade (2, 3 or 4), and treatment, with study site as a random effect; Test type: Superiority; p = 0.5845, ANCOVA; Least Square Mean Difference = -1.32, 95% CI 2-sided [-6.12 to 3.47], Standard Error of Mean 2.41
Statistical Analysis 6: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 27, analysis 5]; Test type: Superiority; p = 0.2514, ANCOVA; Least Square Mean Difference = -2.93, 95% CI 2-sided [-7.97 to 2.11], Standard Error of Mean 2.54
Statistical Analysis 7: Comparison: Placebo vs Tanezumab 2.5 mg; Week 8: Percent Impairment While Working: WPAI parameters were analyzed using ANCOVA model which included covariates of the corresponding baseline score, baseline diary average pain, index joint, highest Kellgren-Lawrence grade (2, 3 or 4), and treatment, with study site as a random effect; Test type: Superiority; p = 0.0717, ANCOVA; Least Square Mean Difference = -6.68, 95% CI 2-sided [-13.97 to 0.60], Standard Error of Mean 3.67
Statistical Analysis 8: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 27, analysis 7]; Test type: Superiority; p = 0.0010, ANCOVA; Least Square Mean Difference = -12.69, 95% CI 2-sided [-20.11 to -5.26], Standard Error of Mean 3.74
Statistical Analysis 9: Comparison: Placebo vs Tanezumab 2.5 mg; Week 16: Percent Impairment While Working: WPAI parameters were analyzed using ANCOVA model which included covariates of the corresponding baseline score, baseline diary average pain, index joint, highest Kellgren-Lawrence grade (2, 3 or 4), and treatment, with study site as a random effect; Test type: Superiority; p = 0.0079, ANCOVA; Least Square Mean Difference = -10.31, 95% CI 2-sided [-17.85 to -2.77], Standard Error of Mean 3.80
Statistical Analysis 10: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 27, analysis 9]; Test type: Superiority; p = 0.0096, ANCOVA; Least Square Mean Difference = -10.56, 95% CI 2-sided [-18.49 to -2.63], Standard Error of Mean 4.00
Statistical Analysis 11: Comparison: Placebo vs Tanezumab 2.5 mg; Week 24: Percent Impairment While Working: WPAI parameters were analyzed using ANCOVA model which included covariates of the corresponding baseline score, baseline diary average pain, index joint, highest Kellgren-Lawrence grade (2, 3 or 4), and treatment, with study site as a random effect; Test type: Superiority; p = 0.3302, ANCOVA; Least Square Mean Difference = -4.28, 95% CI 2-sided [-12.97 to 4.41], Standard Error of Mean 4.37
Statistical Analysis 12: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 27, analysis 11]; Test type: Superiority; p = 0.5483, ANCOVA; Least Square Mean Difference = -2.74, 95% CI 2-sided [-11.78 to 6.30], Standard Error of Mean 4.54
Statistical Analysis 13: Comparison: Placebo vs Tanezumab 2.5 mg; Week 8: Percent Overall Work Impairment: WPAI parameters were analyzed using ANCOVA model which included covariates of the corresponding baseline score, baseline diary average pain, index joint, highest Kellgren-Lawrence grade (2, 3 or 4), and treatment, with study site as a random effect; Test type: Superiority; p = 0.0774, ANCOVA; Least Square Mean Difference = -6.75, 95% CI 2-sided [-14.26 to 0.76], Standard Error of Mean 3.79
Statistical Analysis 14: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 27, analysis 13]; Test type: Superiority; p = 0.0017, ANCOVA; Least Square Mean Difference = -12.48, 95% CI 2-sided [-20.15 to -4.81], Standard Error of Mean 3.87
Statistical Analysis 15: Comparison: Placebo vs Tanezumab 2.5 mg; Week 16: Percent Overall Work Impairment: WPAI parameters were analyzed using ANCOVA model which included covariates of the corresponding baseline score, baseline diary average pain, index joint, highest Kellgren-Lawrence grade (2, 3 or 4), and treatment, with study site as a random effect; Test type: Superiority; p = 0.0135, ANCOVA; Least Square Mean Difference = -9.41, 95% CI 2-sided [-16.83 to -1.99], Standard Error of Mean 3.74
Statistical Analysis 16: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 27, analysis 15]; Test type: Superiority; p = 0.0129, ANCOVA; Least Square Mean Difference = -10.04, 95% CI 2-sided [-17.91 to -2.17], Standard Error of Mean 3.97
Statistical Analysis 17: Comparison: Placebo vs Tanezumab 2.5 mg; Week 24: Percent Overall Work Impairment: WPAI parameters were analyzed using ANCOVA model which included covariates of the corresponding baseline score, baseline diary average pain, index joint, highest Kellgren-Lawrence grade (2, 3 or 4), and treatment, with study site as a random effect; Test type: Superiority; p = 0.3869, ANCOVA; Least Square Mean Difference = -3.85, 95% CI 2-sided [-12.66 to 4.96], Standard Error of Mean 4.43
Statistical Analysis 18: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 27, analysis 17]; Test type: Superiority; p = 0.6485, ANCOVA; Least Square Mean Difference = -2.11, 95% CI 2-sided [-11.31 to 7.08], Standard Error of Mean 4.62
Statistical Analysis 19: Comparison: Placebo vs Tanezumab 2.5 mg; Week 8: Percent Activity Impairment: WPAI parameters were analyzed using ANCOVA model which included covariates of the corresponding baseline score, baseline diary average pain, index joint, highest Kellgren-Lawrence grade (2, 3 or 4), and treatment, with study site as a random effect; Test type: Superiority; p = 0.0001, ANCOVA; Least Square Mean Difference = -6.18, 95% CI 2-sided [-9.34 to -3.03], Standard Error of Mean 1.61
Statistical Analysis 20: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 27, analysis 19]; Test type: Superiority; p < .0001, ANCOVA; Least Square Mean Difference = -9.13, 95% CI 2-sided [-12.26 to -6.00], Standard Error of Mean 1.60
Statistical Analysis 21: Comparison: Placebo vs Tanezumab 2.5 mg; Week 16: Percent Activity Impairment: WPAI parameters were analyzed using ANCOVA model which included covariates of the corresponding baseline score, baseline diary average pain, index joint, highest Kellgren-Lawrence grade (2, 3 or 4), and treatment, with study site as a random effect; Test type: Superiority; p = 0.0008, ANCOVA; Least Square Mean Difference = -6.00, 95% CI 2-sided [-9.51 to -2.50], Standard Error of Mean 1.79
Statistical Analysis 22: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 27, analysis 21]; Test type: Superiority; p < .0001, ANCOVA; Least Square Mean Difference = -6.97, 95% CI 2-sided [-10.44 to -3.51], Standard Error of Mean 1.77
Statistical Analysis 23: Comparison: Placebo vs Tanezumab 2.5 mg; Week 24: Percent Activity Impairment: WPAI parameters were analyzed using ANCOVA model which included covariates of the corresponding baseline score, baseline diary average pain, index joint, highest Kellgren-Lawrence grade (2, 3 or 4), and treatment, with study site as a random effect; Test type: Superiority; p = 0.1004, ANCOVA; Least Square Mean Difference = -3.08, 95% CI 2-sided [-6.76 to 0.60], Standard Error of Mean 1.87
Statistical Analysis 24: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 27, analysis 23]; Test type: Superiority; p = 0.0079, ANCOVA; Least Square Mean Difference = -4.94, 95% CI 2-sided [-8.59 to -1.30], Standard Error of Mean 1.86

28. Secondary Outcome: European Quality of Life- 5 Dimension-5 Levels (EQ-5D-5L) Dimensions Score
Description: EQ-5D-5L is a standardized participant completed questionnaire that measures health-related quality of life and translates that score into an index value or utility score. EQ-5D-5L consists of two components: a health state profile and an optional visual analogue scale (VAS). EQ-5D health state profile is comprised of 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: 1=no problems, 2=slight problems, 3=moderate problems, 4=severe problems, and 5=extreme problems. The health utility score for a participant with no problems in all 5 items is 1 for all countries (except for Zimbabwe where it is 0.9), and is reduced where a participant reports greater levels of problems across the five dimensions.
Time Frame: Baseline, Weeks 8, 16 and 24
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg
Number analyzed (Participants) | 282 | 283 | 284
units on a scale
  Baseline: Mobility: number analyzed (Participants) | 277 | 278 | 283
  Baseline: Mobility | 3.1 (0.63) | 3.1 (0.62) | 3.2 (0.65)
  Baseline: Self-care: number analyzed (Participants) | 277 | 278 | 283
  Baseline: Self-care | 2.4 (0.92) | 2.3 (0.92) | 2.3 (0.90)
  Baseline: Usual activities: number analyzed (Participants) | 277 | 278 | 283
  Baseline: Usual activities | 3.0 (0.65) | 3.0 (0.68) | 3.0 (0.68)
  Baseline: Pain/Discomfort: number analyzed (Participants) | 277 | 278 | 283
  Baseline: Pain/Discomfort | 3.3 (0.72) | 3.2 (0.73) | 3.3 (0.69)
  Baseline: Anxiety/Depression: number analyzed (Participants) | 277 | 278 | 283
  Baseline: Anxiety/Depression | 1.7 (0.87) | 1.7 (0.88) | 1.7 (0.87)
  Week 8: Mobility: number analyzed (Participants) | 273 | 276 | 282
  Week 8: Mobility | 2.6 (0.82) | 2.3 (0.83) | 2.3 (0.80)
  Week 8: Self-care: number analyzed (Participants) | 273 | 276 | 282
  Week 8: Self-care | 2.0 (0.90) | 1.8 (0.80) | 1.6 (0.78)
  Week 8: Usual activities: number analyzed (Participants) | 273 | 276 | 282
  Week 8: Usual activities | 2.5 (0.78) | 2.3 (0.82) | 2.2 (0.78)
  Week 8: Pain/Discomfort: number analyzed (Participants) | 273 | 276 | 282
  Week 8: Pain/Discomfort | 2.7 (0.85) | 2.5 (0.80) | 2.4 (0.79)
  Week 8: Anxiety/Depression: number analyzed (Participants) | 273 | 276 | 282
  Week 8: Anxiety/Depression | 1.5 (0.80) | 1.4 (0.64) | 1.4 (0.71)
  Week 16: Mobility: number analyzed (Participants) | 259 | 266 | 271
  Week 16: Mobility | 2.4 (0.88) | 2.2 (0.84) | 2.2 (0.84)
  Week 16: Self-care: number analyzed (Participants) | 259 | 266 | 271
  Week 16: Self-care | 1.8 (0.88) | 1.7 (0.78) | 1.6 (0.80)
  Week 16: Usual activities: number analyzed (Participants) | 259 | 266 | 272
  Week 16: Usual activities | 2.3 (0.81) | 2.2 (0.78) | 2.1 (0.84)
  Week 16: Pain/Discomfort: number analyzed (Participants) | 259 | 266 | 271
  Week 16: Pain/Discomfort | 2.5 (0.82) | 2.3 (0.80) | 2.3 (0.80)
  Week 16: Anxiety/Depression: number analyzed (Participants) | 259 | 266 | 271
  Week 16: Anxiety/Depression | 1.4 (0.78) | 1.3 (0.61) | 1.4 (0.68)
  Week 24: Mobility: number analyzed (Participants) | 236 | 257 | 255
  Week 24: Mobility | 2.4 (0.78) | 2.3 (0.84) | 2.3 (0.84)
  Week 24: Self-care: number analyzed (Participants) | 236 | 257 | 255
  Week 24: Self-care | 1.7 (0.83) | 1.7 (0.77) | 1.6 (0.76)
  Week 24: Usual activities: number analyzed (Participants) | 236 | 257 | 255
  Week 24: Usual activities | 2.3 (0.78) | 2.2 (0.82) | 2.2 (0.82)
  Week 24: Pain/Discomfort: number analyzed (Participants) | 236 | 257 | 255
  Week 24: Pain/Discomfort | 2.5 (0.81) | 2.4 (0.78) | 2.4 (0.77)
  Week 24: Anxiety/Depression: number analyzed (Participants) | 236 | 257 | 255
  Week 24: Anxiety/Depression | 1.4 (0.67) | 1.4 (0.71) | 1.4 (0.68)

29. Secondary Outcome: European Quality of Life- 5 Dimension-5 Levels (EQ-5D-5L) Overall Health Utility Score/ Index Value
Description: EQ-5D-5L: standardized participant completed questionnaire that measures health-related quality of life and translates that score into an index value or utility score. EQ-5D-5L consists of two components: a health state profile and an optional VAS. EQ-5D health state profile comprises of 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: 1=no problems, 2=slight problems, 3=moderate problems, 4=severe problems, and 5=extreme problems. Responses from the five domains were used to calculate a single utility index (the Overall health utility score) where values are less than equal to (<=) 1. The Overall health utility score for a participant with no problems in all 5 items is 1 for all countries (except for Zimbabwe where it is 0.9), and is reduced where a participant reports greater levels of problems across the five dimensions.
Time Frame: Baseline, Weeks 8, 16 and 24
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg
Number analyzed (Participants) | 282 | 283 | 284
units on a scale
  Baseline: number analyzed (Participants) | 277 | 278 | 283
  Baseline | 0.57 (0.18) | 0.56 (0.18) | 0.56 (0.18)
  Week 8: number analyzed (Participants) | 273 | 276 | 282
  Week 8 | 0.67 (0.17) | 0.71 (0.16) | 0.73 (0.17)
  Week 16: number analyzed (Participants) | 259 | 266 | 271
  Week 16 | 0.70 (0.19) | 0.73 (0.15) | 0.73 (0.17)
  Week 24: number analyzed (Participants) | 236 | 257 | 255
  Week 24 | 0.70 (0.16) | 0.72 (0.16) | 0.73 (0.15)

30. Secondary Outcome: Patient Reported Treatment Impact Assessment-Modified (mPRTI) Score at Weeks 16 and 24: Participant Reported Treatment Impact Assessment-Overall, How Satisfied Are You With The Drug That You Received in This Study?
Description: The mPRTI is a self-administered questionnaire containing participant reported treatment impact assessment (to assess participant satisfaction), participant global preference assessment (to assess previous treatment and preference to continue using the investigational product) and participant willingness to use drug again assessment. For participant satisfaction, participants responded using interactive response technology (IRT) on a 5 point likert scale from 1-5, where 1=extremely dissatisfied, 2=dissatisfied, 3=neither satisfied nor dissatisfied, 4=satisfied and 5=extremely satisfied. Higher scores indicated greater satisfaction.
Time Frame: Weeks 16 and 24
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg
Number analyzed (Participants) | 282 | 283 | 284
Participants
  Week 16: number analyzed (Participants) | 268 | 270 | 278
  Week 16: Extremely Satisfied | 41 | 65 | 65
  Week 16: Satisfied | 109 | 141 | 137
  Week 16: Neither satisfied nor dissatisfied | 78 | 50 | 63
  Week 16: Dissatisfied | 31 | 13 | 11
  Week 16: Extremely dissatisfied | 9 | 1 | 2
  Week 24: number analyzed (Participants) | 238 | 257 | 255
  Week 24: Extremely Satisfied | 46 | 72 | 66
  Week 24: Satisfied | 97 | 119 | 128
  Week 24: Neither satisfied nor dissatisfied | 64 | 54 | 48
  Week 24: Dissatisfied | 28 | 10 | 9
  Week 24: Extremely dissatisfied | 3 | 2 | 4

31. Secondary Outcome: Patient Reported Treatment Impact Assessment-Modified (mPRTI) Score at Weeks 16 and 24: Participant Global Preference Assessment- What is The Current or Most Recent Treatment You Were Receiving For Osteoarthritis Pain Before Enrolling?
Description: The mPRTI is a self-administered questionnaire containing participant reported treatment impact assessment (to assess participant satisfaction), participant global preference assessment (to assess previous treatment and preference to continue using the investigational product) and participant willingness to use drug again assessment. To assess previous treatment, participants responded for, 1=injectable prescription medicines, 2=prescription medicines taken by mouth, 3=surgery, 4=prescription medicines and surgery and 5=no treatment.
Time Frame: Weeks 16 and 24
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg
Number analyzed (Participants) | 282 | 283 | 284
Participants
  Week 16: number analyzed (Participants) | 268 | 270 | 278
  Week 16: Injectable prescription medicines | 23 | 34 | 28
  Week 16: Prescription medicines taken by mouth | 214 | 212 | 224
  Week 16: Surgery | 5 | 0 | 1
  Week 16: Prescription medicines and surgery | 8 | 5 | 5
  Week 16: No treatment | 18 | 19 | 20
  Week 24: number analyzed (Participants) | 238 | 257 | 255
  Week 24: Injectable prescription medicines | 16 | 21 | 35
  Week 24: Prescription medicines taken by mouth | 196 | 211 | 196
  Week 24: Surgery | 3 | 0 | 3
  Week 24: Prescription medicines and surgery | 4 | 3 | 4
  Week 24: No treatment | 19 | 22 | 17

32. Secondary Outcome: Patient Reported Treatment Impact Assessment-Modified (mPRTI) Score at Weeks 16 and 24: Participant Global Preference Assessment- Overall, do You Prefer The Drug That You Received in This Study to Previous Treatment?
Description: The mPRTI is a self-administered questionnaire containing participant reported treatment impact assessment (to assess participant satisfaction), participant global preference assessment (to assess previous treatment and preference to continue using the investigational product) and participant willingness to use drug again assessment. To assess preference to continue using the investigational product, participants responded using interactive response technology (IRT) on a 5 point likert scale from 1-5, where, 1= yes, I definitely prefer the drug that I am receiving now, 2= I have a slight preference for the drug that I am receiving now, 3= I have no preference either way, 4= I have a slight preference for my previous treatment, 5= No, I definitely prefer my previous treatment. Higher scores indicate lesser preference to use the investigational product.
Time Frame: Weeks 16 and 24
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg
Number analyzed (Participants) | 282 | 283 | 284
Participants
  Week 16: number analyzed (Participants) | 268 | 270 | 278
  Week 16: Yes, definitely prefer the study drug | 106 | 129 | 138
  Week 16: Slight preference for the study drug | 66 | 86 | 83
  Week 16: No preference either way | 65 | 41 | 48
  Week 16: Slight preference for my previous treatment | 14 | 11 | 4
  Week 16: No, definitely prefer my previous treatment | 17 | 3 | 5
  Week 24: number analyzed (Participants) | 238 | 257 | 255
  Week 24: Yes, definitely prefer the study drug | 87 | 129 | 127
  Week 24: Slight preference for the study drug | 73 | 79 | 78
  Week 24: No preference either way | 58 | 43 | 36
  Week 24: Slight preference for my previous treatment | 14 | 4 | 8
  Week 24: No, definitely prefer my previous treatment | 6 | 2 | 6

33. Secondary Outcome: Patient Reported Treatment Impact Assessment-Modified (mPRTI) Score at Weeks 16 and 24: Participant Willingness to Use Drug Again Assessment- Willing to Use The Same Drug That You Have Received in This Study For Your Osteoarthritis Pain?
Description: The mPRTI is a self-administered questionnaire containing participant reported treatment impact assessment (to assess participant satisfaction), participant global preference assessment (to assess previous treatment and preference to continue using the investigational product) and participant willingness to use drug again assessment. To assess Patient willingness to use drug again, participants responded using interactive response technology (IRT) on a 5 point likert scale from 1-5, where, 1= yes, I would definitely want to use the same drug again, 2= I might want to use the same drug again, 3= I am not sure, 4= I might not want to use the same drug again, 5= no, I definitely would not want to use the same drug again. Higher scores indicate lesser willingness to use the investigational product.
Time Frame: Weeks 16 and 24
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg
Number analyzed (Participants) | 282 | 283 | 284
Participants
  Week 16: number analyzed (Participants) | 268 | 270 | 278
  Week 16: Yes, definitely want to use the same drug again | 111 | 144 | 155
  Week 16: Might want to use the same drug again | 67 | 83 | 74
  Week 16: I am not sure | 59 | 29 | 41
  Week 16: Might not want to use the same drug again | 10 | 9 | 5
  Week 16: No:definitely wouldn't want to use same drug again | 21 | 5 | 3
  Week 24: number analyzed (Participants) | 238 | 257 | 255
  Week 24: Yes, definitely want to use the same drug again | 101 | 131 | 139
  Week 24: Might want to use the same drug again | 62 | 73 | 63
  Week 24: I am not sure | 53 | 43 | 38
  Week 24: Might not want to use the same drug again | 13 | 5 | 9
  Week 24: No:definitely wouldn't want to use same drug again | 9 | 5 | 6

34. Secondary Outcome: Health Care Resource Utilization (HCRU): Number of Visits of Services Directly Related to Osteoarthritis
Description: Osteoarthritis HCRU assessed healthcare usage during last 3 months (for Baseline and Week 48) and past 8 weeks (for Week 32). Visits of services directly related to osteoarthritis evaluated were: visits to primary care physician, neurologist, rheumatologist, physician assistant or nurse practitioner, pain specialist, orthopedist, physical therapist, chiropractor, alternative medicine or therapy, podiatrist, nutritionist/dietitian, radiologist, home healthcare services and other practitioner.
Time Frame: Baseline, Weeks 32 and 48
Population: as for outcome 26
Measure: Median (Full Range); unit: visits
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg
Number analyzed (Participants) | 282 | 283 | 284
visits
  Baseline: Primary Care Physician: number analyzed (Participants) | 116 | 115 | 112
  Baseline: Primary Care Physician | 2.0 [1.0 to 14.0] | 2.0 [1.0 to 10.0] | 2.0 [1.0 to 7.0]
  Baseline: Neurologist: number analyzed (Participants) | 4 | 7 | 5
  Baseline: Neurologist | 1.0 [1.0 to 3.0] | 1.0 [1.0 to 100.0] | 1.0 [1.0 to 2.0]
  Baseline: Rheumatologist: number analyzed (Participants) | 82 | 99 | 89
  Baseline: Rheumatologist | 2.0 [1.0 to 102.0] | 2.0 [1.0 to 11.0] | 2.0 [1.0 to 5.0]
  Baseline:Physician assistant or nurse Practitioner: number analyzed (Participants) | 7 | 6 | 5
  Baseline:Physician assistant or nurse Practitioner | 3.0 [1.0 to 7.0] | 2.5 [1.0 to 5.0] | 3.0 [3.0 to 8.0]
  Baseline: Pain specialist: number analyzed (Participants) | 12 | 21 | 24
  Baseline: Pain specialist | 1.0 [1.0 to 3.0] | 2.0 [1.0 to 5.0] | 1.0 [1.0 to 6.0]
  Baseline: Orthopedist: number analyzed (Participants) | 84 | 83 | 85
  Baseline: Orthopedist | 2.0 [1.0 to 12.0] | 2.0 [1.0 to 12.0] | 2.0 [1.0 to 7.0]
  Baseline: Physical therapist: number analyzed (Participants) | 25 | 20 | 30
  Baseline: Physical therapist | 10.0 [1.0 to 24.0] | 3.5 [1.0 to 100.0] | 2.5 [1.0 to 60.0]
  Baseline: Chiropractor: number analyzed (Participants) | 3 | 1 | 1
  Baseline: Chiropractor | 2.0 [1.0 to 3.0] | 1.0 [1.0 to 1.0] | 2.0 [2.0 to 2.0]
  Baseline: Alternative medicine or therapy: number analyzed (Participants) | 4 | 2 | 4
  Baseline: Alternative medicine or therapy | 1.0 [1.0 to 3.0] | 2.0 [2.0 to 2.0] | 2.5 [1.0 to 4.0]
  Baseline: Podiatrist: number analyzed (Participants) | 7 | 4 | 3
  Baseline: Podiatrist | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 1.0] | 3.0 [2.0 to 3.0]
  Baseline: Nutritionist/dietitian: number analyzed (Participants) | 3 | 2 | 7
  Baseline: Nutritionist/dietitian | 3.0 [2.0 to 5.0] | 2.0 [1.0 to 3.0] | 3.0 [1.0 to 8.0]
  Baseline: Radiologist: number analyzed (Participants) | 44 | 34 | 46
  Baseline: Radiologist | 1.0 [1.0 to 4.0] | 1.0 [1.0 to 3.0] | 1.0 [1.0 to 4.0]
  Baseline: Home healthcare services: number analyzed (Participants) | 1 | 1 | 1
  Baseline: Home healthcare services | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 24.0 [24.0 to 24.0]
  Baseline: Other practitioner: number analyzed (Participants) | 13 | 15 | 21
  Baseline: Other practitioner | 1.0 [1.0 to 6.0] | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 12.0]
  Week 32: Primary Care Physician: number analyzed (Participants) | 62 | 61 | 57
  Week 32: Primary Care Physician | 1.0 [1.0 to 101.0] | 1.0 [1.0 to 100.0] | 1.0 [1.0 to 190.0]
  Week 32: Neurologist: number analyzed (Participants) | 1 | 4 | 2
  Week 32: Neurologist | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 51.0 [1.0 to 101.0]
  Week 32: Rheumatologist: number analyzed (Participants) | 23 | 34 | 33
  Week 32: Rheumatologist | 1.0 [1.0 to 10.0] | 1.0 [1.0 to 3.0] | 1.0 [1.0 to 20.0]
  Week 32: Physician assistant or nurse Practitioner: number analyzed (Participants) | 9 | 4 | 3
  Week 32: Physician assistant or nurse Practitioner | 1.0 [1.0 to 111.0] | 2.0 [1.0 to 3.0] | 4.0 [1.0 to 101.0]
  Week 32: Pain specialist: number analyzed (Participants) | 6 | 7 | 9
  Week 32: Pain specialist | 1.0 [1.0 to 3.0] | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 16.0]
  Week 32: Orthopedist: number analyzed (Participants) | 34 | 36 | 35
  Week 32: Orthopedist | 1.0 [1.0 to 111.0] | 1.0 [1.0 to 6.0] | 1.0 [1.0 to 2.0]
  Week 32: Physical therapist: number analyzed (Participants) | 11 | 12 | 12
  Week 32: Physical therapist | 8.0 [1.0 to 111.0] | 2.0 [1.0 to 12.0] | 5.5 [1.0 to 16.0]
  Week 32: Chiropractor: number analyzed (Participants) | 0 | 1 | 1
  Week 32: Chiropractor |  | 8.0 [8.0 to 8.0] | 2.0 [2.0 to 2.0]
  Week 32: Alternative medicine or therapy: number analyzed (Participants) | 5 | 2 | 6
  Week 32: Alternative medicine or therapy | 3.0 [1.0 to 10.0] | 2.5 [1.0 to 4.0] | 1.5 [1.0 to 10.0]
  Week 32: Podiatrist: number analyzed (Participants) | 4 | 4 | 1
  Week 32: Podiatrist | 1.0 [1.0 to 1.0] | 1.5 [1.0 to 2.0] | 1.0 [1.0 to 1.0]
  Week 32: Nutritionist/dietitian: number analyzed (Participants) | 2 | 1 | 1
  Week 32: Nutritionist/dietitian | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 2.0 [2.0 to 2.0]
  Week 32: Radiologist: number analyzed (Participants) | 10 | 10 | 14
  Week 32: Radiologist | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 3.0] | 1.0 [1.0 to 2.0]
  Week 32: Home healthcare services: number analyzed (Participants) | 1 | 1 | 1
  Week 32: Home healthcare services | 10.0 [10.0 to 10.0] | 1.0 [1.0 to 1.0] | 10.0 [10.0 to 10.0]
  Week 32: Other practitioner: number analyzed (Participants) | 13 | 12 | 14
  Week 32: Other practitioner | 1.0 [1.0 to 8.0] | 1.0 [1.0 to 8.0] | 1.0 [1.0 to 16.0]
  Week 48: Primary Care Physician: number analyzed (Participants) | 53 | 63 | 64
  Week 48: Primary Care Physician | 1.0 [1.0 to 7.0] | 1.0 [1.0 to 90.0] | 2.0 [1.0 to 100.0]
  Week 48: Neurologist: number analyzed (Participants) | 3 | 5 | 1
  Week 48: Neurologist | 1.0 [1.0 to 4.0] | 1.0 [1.0 to 2.0] | 2.0 [2.0 to 2.0]
  Week 48: Rheumatologist: number analyzed (Participants) | 16 | 34 | 27
  Week 48: Rheumatologist | 1.0 [1.0 to 3.0] | 1.0 [1.0 to 90.0] | 1.0 [1.0 to 3.0]
  Week 48: Physician assistant or nurse Practitioner: number analyzed (Participants) | 4 | 8 | 4
  Week 48: Physician assistant or nurse Practitioner | 5.5 [2.0 to 55.0] | 2.5 [1.0 to 90.0] | 2.0 [1.0 to 4.0]
  Week 48: Pain specialist: number analyzed (Participants) | 4 | 3 | 2
  Week 48: Pain specialist | 1.0 [1.0 to 1.0] | 3.0 [1.0 to 90.0] | 1.0 [1.0 to 1.0]
  Week 48: Orthopedist: number analyzed (Participants) | 31 | 44 | 55
  Week 48: Orthopedist | 2.0 [1.0 to 6.0] | 2.0 [1.0 to 90.0] | 2.0 [1.0 to 8.0]
  Week 48: Physical therapist: number analyzed (Participants) | 13 | 19 | 20
  Week 48: Physical therapist | 6.0 [1.0 to 16.0] | 6.0 [1.0 to 90.0] | 10.0 [1.0 to 36.0]
  Week 48: Chiropractor: number analyzed (Participants) | 2 | 2 | 1
  Week 48: Chiropractor | 1.0 [1.0 to 1.0] | 46.5 [3.0 to 90.0] | 3.0 [3.0 to 3.0]
  Week 48: Alternative medicine or therapy: number analyzed (Participants) | 0 | 6 | 3
  Week 48: Alternative medicine or therapy |  | 11.0 [3.0 to 90.0] | 3.0 [2.0 to 5.0]
  Week 48: Podiatrist: number analyzed (Participants) | 5 | 3 | 3
  Week 48: Podiatrist | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 190.0] | 3.0 [1.0 to 110.0]
  Week 48: Nutritionist/dietitian: number analyzed (Participants) | 3 | 1 | 3
  Week 48: Nutritionist/dietitian | 1.0 [1.0 to 2.0] | 130.0 [130.0 to 130.0] | 1.0 [1.0 to 2.0]
  Week 48: Radiologist: number analyzed (Participants) | 5 | 8 | 11
  Week 48: Radiologist | 1.0 [1.0 to 1.0] | 1.5 [1.0 to 190.0] | 1.0 [1.0 to 91.0]
  Week 48: Home healthcare services: number analyzed (Participants) | 0 | 3 | 0
  Week 48: Home healthcare services |  | 5.0 [1.0 to 90.0] |
  Week 48: Other practitioner: number analyzed (Participants) | 6 | 13 | 9
  Week 48: Other practitioner | 1.0 [1.0 to 3.0] | 1.0 [1.0 to 90.0] | 2.0 [1.0 to 4.0]

35. Secondary Outcome: Health Care Resource Utilization (HCRU): Number of Participants Who Visited the Emergency Room Due to Osteoarthritis
Description: Osteoarthritis HCRU assessed healthcare usage during last 3 months (for Baseline and Week 48) and past 8 weeks (for Week 32). Domain evaluated was number of participants who visited the emergency room due to osteoarthritis.
Time Frame: Baseline, Weeks 32 and 48
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg
Number analyzed (Participants) | 282 | 283 | 284
Participants
  Baseline: number analyzed (Participants) | 281 | 282 | 284
  Baseline | 1 | 3 | 2
  Week 32: number analyzed (Participants) | 250 | 260 | 251
  Week 32 | 2 | 2 | 0
  Week 48: number analyzed (Participants) | 218 | 240 | 231
  Week 48 | 2 | 1 | 2

36. Secondary Outcome: Health Care Resource Utilization (HCRU): Number of Visits to the Emergency Room Due to Osteoarthritis
Description: Osteoarthritis HCRU assessed healthcare usage during last 3 months (for Baseline and Week 48) and past 8 weeks (for Week 32). Domain evaluated was number of visits to the emergency room due to OA.
Time Frame: Baseline, Weeks 32 and 48
Population: as for outcome 17
Measure: Median (Full Range); unit: visits
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg
Number analyzed (Participants) | 282 | 283 | 284
visits
  Baseline: number analyzed (Participants) | 1 | 3 | 2
  Baseline | 1.0 [1.0 to 1.0] | 2.0 [1.0 to 2.0] | 1.5 [1.0 to 2.0]
  Week 32: number analyzed (Participants) | 2 | 2 | 0
  Week 32 | 1.5 [1.0 to 2.0] | 1.0 [1.0 to 1.0] |
  Week 48: number analyzed (Participants) | 2 | 1 | 2
  Week 48 | 2.0 [1.0 to 3.0] | 2.0 [2.0 to 2.0] | 1.0 [1.0 to 1.0]

37. Secondary Outcome: Health Care Resource Utilization (HCRU): Number of Participants Hospitalized Due to Osteoarthritis
Description: Osteoarthritis HCRU assessed healthcare usage during last 3 months (for Baseline and Week 48) and past 8 weeks (for Week 32). Domain evaluated was number of participants who were hospitalized due to OA.
Time Frame: Baseline, Weeks 32 and 48
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg
Number analyzed (Participants) | 282 | 283 | 284
Participants
  Baseline: number analyzed (Participants) | 281 | 282 | 284
  Baseline | 1 | 2 | 1
  Week 32: number analyzed (Participants) | 250 | 260 | 251
  Week 32 | 1 | 1 | 1
  Week 48: number analyzed (Participants) | 218 | 240 | 231
  Week 48 | 0 | 1 | 5

38. Secondary Outcome: Health Care Resource Utilization (HCRU): Number of Nights Stayed in the Hospital Due to Osteoarthritis
Description: Osteoarthritis HCRU assessed healthcare usage during last 3 months (for Baseline and Week 48) and past 8 weeks (for Week 32). Domain evaluated was number of nights stayed in the hospital due to OA.
Time Frame: Baseline, Weeks 32 and 48
Population: as for outcome 17
Measure: Median (Full Range); unit: nights
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg
Number analyzed (Participants) | 282 | 283 | 284
nights
  Baseline: number analyzed (Participants) | 1 | 2 | 1
  Baseline | 1.0 [1.0 to 1.0] | 11.0 [1.0 to 21.0] | 1.0 [1.0 to 1.0]
  Week 32: number analyzed (Participants) | 1 | 1 | 1
  Week 32 | 5.0 [5.0 to 5.0] | 21.0 [21.0 to 21.0] | 2.0 [2.0 to 2.0]
  Week 48: number analyzed (Participants) | 0 | 1 | 5
  Week 48 |  | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 9.0]

39. Secondary Outcome: Health Care Resource Utilization (HCRU): Number of Participants Who Used Any Aids/Devices for Doing Things
Description: Osteoarthritis HCRU assessed healthcare usage during last 3 months (for Baseline and Week 48) and past 8 weeks (for Week 32). Domain evaluated was number of participants who used any aids/devices for doing things. Aids such as walking aid, wheelchair, device or utensil for dress/bathe/eat and any other aids/devices.
Time Frame: Baseline, Weeks 32 and 48
Population: The intent to treat (ITT) population included all randomized participants who received at least one dose of subcutaneous (SC) study medication (either tanezumab or placebo). Here, 'Number analyzed' = Participants evaluable for this outcome measure for specified categories.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg
Number analyzed (Participants) | 282 | 283 | 284
Participants
  Baseline:Walking aid use: number analyzed (Participants) | 281 | 282 | 284
  Baseline:Walking aid use: Never | 250 | 240 | 242
  Baseline:Walking aid use: Rarely | 4 | 8 | 5
  Baseline:Walking aid use: Sometimes | 11 | 13 | 15
  Baseline:Walking aid use: Often | 7 | 12 | 7
  Baseline:Walking aid use: Always | 9 | 9 | 15
  Baseline: Wheelchair use: number analyzed (Participants) | 281 | 282 | 284
  Baseline: Wheelchair use: Never | 281 | 282 | 283
  Baseline: Wheelchair use: Rarely | 0 | 0 | 0
  Baseline: Wheelchair use: Sometimes | 0 | 0 | 0
  Baseline: Wheelchair use: Often | 0 | 0 | 1
  Baseline: Wheelchair use: Always | 0 | 0 | 0
  Baseline:Device/Utensil to dress bathe eat: number analyzed (Participants) | 281 | 282 | 284
  Baseline:Device/Utensil to dress bathe eat: Never | 271 | 274 | 279
  Baseline:Device/Utensil to dress bathe eat: Rarely | 1 | 2 | 0
  Baseline:Device/Utensil to dress bathe eat: Sometimes | 4 | 2 | 2
  Baseline:Device/Utensil to dress bathe eat: Often | 2 | 0 | 3
  Baseline:Device/Utensil to dress bathe eat: Always | 3 | 4 | 0
  Baseline:Other aids or devices: number analyzed (Participants) | 281 | 282 | 284
  Baseline:Other aids or devices: Never | 275 | 265 | 270
  Baseline:Other aids or devices: Rarely | 2 | 2 | 5
  Baseline:Other aids or devices: Sometimes | 0 | 8 | 4
  Baseline:Other aids or devices: Often | 3 | 5 | 3
  Baseline:Other aids or devices: Always | 1 | 2 | 2
  Week 32: Walking aid use: number analyzed (Participants) | 250 | 260 | 251
  Week 32: Walking aid use: Never | 225 | 232 | 214
  Week 32: Walking aid use: Rarely | 4 | 1 | 6
  Week 32: Walking aid use: Sometimes | 8 | 8 | 10
  Week 32: Walking aid use: Often | 4 | 7 | 12
  Week 32: Walking aid use: Always | 9 | 12 | 9
  Week 32: Wheelchair use: number analyzed (Participants) | 250 | 260 | 251
  Week 32: Wheelchair use: Never | 248 | 260 | 250
  Week 32: Wheelchair use: Rarely | 1 | 0 | 0
  Week 32: Wheelchair use: Sometimes | 0 | 0 | 0
  Week 32: Wheelchair use: Often | 0 | 0 | 1
  Week 32: Wheelchair use: Always | 1 | 0 | 0
  Week 32: Device/Utensil to dress bathe eat: number analyzed (Participants) | 250 | 260 | 251
  Week 32: Device/Utensil to dress bathe eat: Never | 248 | 257 | 246
  Week 32: Device/Utensil to dress bathe eat: Rarely | 0 | 0 | 1
  Week 32: Device/Utensil to dress bathe eat: Sometimes | 1 | 2 | 2
  Week 32: Device/Utensil to dress bathe eat: Often | 0 | 0 | 1
  Week 32: Device/Utensil to dress bathe eat: Always | 1 | 1 | 1
  Week 32: Other aids or devices: number analyzed (Participants) | 250 | 260 | 251
  Week 32: Other aids or devices: Never | 246 | 252 | 245
  Week 32: Other aids or devices: Rarely | 0 | 0 | 1
  Week 32: Other aids or devices: Sometimes | 2 | 4 | 3
  Week 32: Other aids or devices: Often | 1 | 4 | 1
  Week 32: Other aids or devices: Always | 1 | 0 | 1
  Week 48: Walking aid use: number analyzed (Participants) | 218 | 240 | 231
  Week 48: Walking aid use: Never | 200 | 211 | 191
  Week 48: Walking aid use: Rarely | 1 | 2 | 3
  Week 48: Walking aid use: Sometimes | 6 | 12 | 13
  Week 48: Walking aid use: Often | 4 | 8 | 10
  Week 48: Walking aid use: Always | 7 | 7 | 14
  Week 48: Wheelchair use: number analyzed (Participants) | 218 | 240 | 231
  Week 48: Wheelchair use: Never | 217 | 240 | 230
  Week 48: Wheelchair use: Rarely | 0 | 0 | 0
  Week 48: Wheelchair use: Sometimes | 0 | 0 | 0
  Week 48: Wheelchair use: Often | 0 | 0 | 1
  Week 48: Wheelchair use: Always | 1 | 0 | 0
  Week 48: Device/Utensil to dress bathe eat: number analyzed (Participants) | 218 | 240 | 231
  Week 48: Device/Utensil to dress bathe eat: Never | 217 | 238 | 228
  Week 48: Device/Utensil to dress bathe eat: Rarely | 1 | 0 | 0
  Week 48: Device/Utensil to dress bathe eat: Sometimes | 0 | 0 | 2
  Week 48: Device/Utensil to dress bathe eat: Often | 0 | 0 | 0
  Week 48: Device/Utensil to dress bathe eat: Always | 0 | 2 | 1
  Week 48: Other aids or devices: number analyzed (Participants) | 218 | 240 | 231
  Week 48: Other aids or devices: Never | 215 | 234 | 225
  Week 48: Other aids or devices: Rarely | 1 | 0 | 1
  Week 48: Other aids or devices: Sometimes | 2 | 2 | 1
  Week 48: Other aids or devices: Often | 0 | 3 | 3
  Week 48: Other aids or devices: Always | 0 | 1 | 1

40. Secondary Outcome: Health Care Resource Utilization (HCRU): Number of Participants Who Quit Job Due to Osteoarthritis
Description: Osteoarthritis HCRU assessed healthcare usage (during 3 months prior to baseline) at baseline, Week 32 and Week 48. Domain evaluated was number of participants who quit job due to OA.
Time Frame: Baseline, Weeks 32 and 48
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg
Number analyzed (Participants) | 282 | 283 | 284
Participants
  Baseline: number analyzed (Participants) | 281 | 282 | 284
  Baseline | 13 | 12 | 9
  Week 32: number analyzed (Participants) | 250 | 260 | 251
  Week 32 | 7 | 9 | 4
  Week 48: number analyzed (Participants) | 218 | 240 | 231
  Week 48 | 7 | 7 | 4

41. Secondary Outcome: Health Care Resource Utilization (HCRU): Duration Since Quitting Job Due to Osteoarthritis
Description: Osteoarthritis HCRU assessed healthcare usage (during 3 months prior to baseline) at baseline, Week 32 and Week 48. Domain evaluated was duration since quitting job due to OA.
Time Frame: Baseline, Weeks 32 and 48
Population: ITT population: all randomized participants who received at least one dose of SC study medication (either Tanezumab or placebo). One additional participant apart from the ones who had responded for quitting job responded to duration since quitting job. 'Number analyzed' = Participants evaluable for this outcome measure at specified time points.
Measure: Median (Full Range); unit: years
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg
Number analyzed (Participants) | 282 | 283 | 284
years
  Baseline: number analyzed (Participants) | 13 | 12 | 9
  Baseline | 2.0 [0.1 to 20.9] | 1.0 [0.2 to 7.0] | 5.3 [0.1 to 30.0]
  Week 32: number analyzed (Participants) | 7 | 10 | 4
  Week 32 | 0.5 [0.3 to 2.9] | 2.4 [0.2 to 17.8] | 1.1 [0.1 to 10.2]
  Week 48: number analyzed (Participants) | 7 | 7 | 4
  Week 48 | 0.8 [0.3 to 2.8] | 2.5 [0.6 to 10.0] | 0.7 [0.1 to 1.5]

42. Secondary Outcome: Number of Participants Who Withdrew Due to Lack of Efficacy
Description: Number of participants who withdrew from treatment due to lack of efficacy have been reported here.
Time Frame: Baseline up to Week 24
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg
Number analyzed (Participants) | 282 | 283 | 284
Participants | 18 | 2 | 3
Statistical Analysis 1: Comparison: Placebo vs Tanezumab 2.5 mg; Logistic regression model included baseline diary average pain, baseline WOMAC pain score, classification variables index joint, highest Kellgren-Lawrence grade and treatment. Odds ratio and 95% CI estimated from logistic regression model; Test type: Superiority; p = 0.0027, Regression, Logistic; Odds Ratio (OR) = 0.10, 95% CI 2-sided [0.02 to 0.46]
Statistical Analysis 2: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 42, analysis 1]; Test type: Superiority; p = 0.0033, Regression, Logistic; Odds Ratio (OR) = 0.16, 95% CI 2-sided [0.05 to 0.54]

43. Secondary Outcome: Time to Discontinuation Due to Lack of Efficacy
Description: Time to discontinuation due to lack of efficacy was defined as the time interval from the date of first study drug administration up to the date of discontinuation of participant from treatment due to lack of efficacy.
Time Frame: Baseline up to Week 24
Population: The intent to treat population included all randomized participants who received at least one dose of subcutaneous study medication (either tanezumab or placebo). Here, 'Overall number of participants analyzed' signifies participants who discontinued from the study due to lack of efficacy.
Measure: Median (Full Range); unit: days
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg
Number analyzed (Participants) | 18 | 2 | 3
days | NA [10 to NA] — Due to the Kaplan-Meier estimate not reaching the level for discontinuation due to lack of efficacy, median and upper limit could not be calculated. | NA [27 to NA] — Due to the Kaplan-Meier estimate not reaching the level for discontinuation due to lack of efficacy, median and upper limit could not be calculated. | NA [12 to NA] — Due to the Kaplan-Meier estimate not reaching the level for discontinuation due to lack of efficacy, median and upper limit could not be calculated.
Statistical Analysis 1: Comparison: Placebo vs Tanezumab 2.5 mg; Missing data for the selected percentile(s) was due to the Kaplan-Meier estimate not reaching the level for discontinuation due to lack of efficacy; Test type: Superiority; p = 0.0002, Log Rank — P-value based on the log-rank test
Statistical Analysis 2: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 43, analysis 1]; Test type: Superiority; p = 0.0007, Log Rank — P-value based on the log-rank test

44. Secondary Outcome: Number of Participants Who Took Rescue Medication During Weeks 2, 4, 8, 12, 16 and 24
Description: In case of inadequate pain relief, acetaminophen/paracetamol up to 4000 mg per day up to 5 days in a week could be taken as rescue medication between day 1 and week 24. Number of participants with any use of rescue medication during the particular study week were summarized.
Time Frame: Weeks 2, 4, 8, 12, 16 and 24
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg
Number analyzed (Participants) | 282 | 283 | 284
Participants
  Week 2 | 205 | 150 | 169
  Week 4 | 181 | 134 | 150
  Week 8 | 166 | 135 | 146
  Week 12 | 151 | 122 | 122
  Week 16 | 154 | 130 | 122
  Week 24 | 126 | 127 | 115
Statistical Analysis 1: Comparison: Placebo vs Tanezumab 2.5 mg; Week 2: Odds ratio and 95%CI estimated from logistic regression model. Logistic regression model included baseline WOMAC pain subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p < .0001, Regression, Logistic; Odds Ratio (OR) = 0.42, 95% CI 2-sided [0.29 to 0.59]
Statistical Analysis 2: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 44, analysis 1]; Test type: Superiority; p = 0.0010, Regression, Logistic; Odds Ratio (OR) = 0.55, 95% CI 2-sided [0.38 to 0.78]
Statistical Analysis 3: Comparison: Placebo vs Tanezumab 2.5 mg; Week 4: Odds ratio and 95%CI estimated from logistic regression model. Logistic regression model included baseline WOMAC pain subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p < .0001, Regression, Logistic; Odds Ratio (OR) = 0.50, 95% CI 2-sided [0.36 to 0.70]
Statistical Analysis 4: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 44, analysis 3]; Test type: Superiority; p = 0.0067, Regression, Logistic; Odds Ratio (OR) = 0.62, 95% CI 2-sided [0.44 to 0.88]
Statistical Analysis 5: Comparison: Placebo vs Tanezumab 2.5 mg; Week 8: Odds ratio and 95%CI estimated from logistic regression model. Logistic regression model included baseline WOMAC pain subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p = 0.0087, Regression, Logistic; Odds Ratio (OR) = 0.64, 95% CI 2-sided [0.45 to 0.89]
Statistical Analysis 6: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 44, analysis 5]; Test type: Superiority; p = 0.0787, Regression, Logistic; Odds Ratio (OR) = 0.74, 95% CI 2-sided [0.53 to 1.04]
Statistical Analysis 7: Comparison: Placebo vs Tanezumab 2.5 mg; Week 12: Odds ratio and 95%CI estimated from logistic regression model. Logistic regression model included baseline WOMAC pain subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p = 0.0129, Regression, Logistic; Odds Ratio (OR) = 0.65, 95% CI 2-sided [0.47 to 0.91]
Statistical Analysis 8: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 44, analysis 7]; Test type: Superiority; p = 0.0124, Regression, Logistic; Odds Ratio (OR) = 0.65, 95% CI 2-sided [0.47 to 0.91]
Statistical Analysis 9: Comparison: Placebo vs Tanezumab 2.5 mg; Week 16: Odds ratio and 95%CI estimated from logistic regression model. Logistic regression model included baseline WOMAC pain subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p = 0.0399, Regression, Logistic; Odds Ratio (OR) = 0.70, 95% CI 2-sided [0.50 to 0.98]
Statistical Analysis 10: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 44, analysis 9]; Test type: Superiority; p = 0.0060, Regression, Logistic; Odds Ratio (OR) = 0.62, 95% CI 2-sided [0.45 to 0.87]
Statistical Analysis 11: Comparison: Placebo vs Tanezumab 2.5 mg; Week 24: Odds ratio and 95%CI estimated from logistic regression model. Logistic regression model included baseline WOMAC pain subscale, baseline diary average pain, and classification variables index joint, highest Kellgren-Lawrence grade and treatment; Test type: Superiority; p = 0.9449, Regression, Logistic; Odds Ratio (OR) = 1.01, 95% CI 2-sided [0.72 to 1.42]
Statistical Analysis 12: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 44, analysis 11]; Test type: Superiority; p = 0.3238, Regression, Logistic; Odds Ratio (OR) = 0.84, 95% CI 2-sided [0.60 to 1.18]

45. Secondary Outcome: Number of Participants Who Took Rescue Medication During Week 32
Description: In case of inadequate pain relief, after Week 24, acetaminophen/paracetamol up to 4000 mg per day up to 5 days in a week could be taken as rescue medication and use was reported weekly via diary. Number of participants with any use of rescue medication during the 4 weeks up to and including the particular study week were summarized.
Time Frame: Week 32
Population: The intent to treat population included all randomized participants who received at least one dose of subcutaneous study medication (either tanezumab or placebo). Here, 'Overall number of participants analyzed' signifies participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg
Number analyzed (Participants) | 231 | 251 | 249
Participants | 130 | 158 | 149

46. Secondary Outcome: Number of Days of Rescue Medication Used at Weeks 2, 4, 8, 12, 16 and 24
Description: In case of inadequate pain relief during the treatment period, acetaminophen/paracetamol up to 4000 mg per day up to 5 days in a week a could be taken as rescue medication. Number of days the participants used the rescue medication during the particular study weeks were summarized.
Time Frame: Weeks 2, 4, 8, 12, 16 and 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: days
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg
Number analyzed (Participants) | 282 | 283 | 284
days
  Week 2 | 3.17 (0.27) | 2.12 (0.19) | 2.39 (0.21)
  Week 4 | 2.82 (0.28) | 1.81 (0.18) | 2.07 (0.21)
  Week 8 | 2.54 (0.26) | 1.83 (0.19) | 1.92 (0.20)
  Week 12 | 2.29 (0.27) | 1.70 (0.20) | 1.72 (0.20)
  Week 16 | 2.11 (0.24) | 1.64 (0.19) | 1.70 (0.19)
  Week 24 | 1.74 (0.22) | 1.49 (0.18) | 1.43 (0.18)
Statistical Analysis 1: Comparison: Placebo vs Tanezumab 2.5 mg; Week 2: Least square (LS) Mean was ratio of treatments. Analysis was performed using negative binomial model with model terms of baseline WOMAC Pain subscale score, baseline diary average pain score, index joint, Kellgren Lawrence grade, and treatment group; Test type: Superiority; p = 0.0001, Negative binomial model; LS Mean Ratio = 0.67, 95% CI 2-sided [0.54 to 0.82], Standard Error of Mean 0.07
Statistical Analysis 2: Comparison: Placebo vs Tanezumab 5 mg; Week 2: LS Mean was ratio of treatments. Analysis was performed using negative binomial model with model terms of baseline WOMAC Pain subscale score, baseline diary average pain score, index joint, Kellgren Lawrence grade, and treatment group; Test type: Superiority; p = 0.0067, Negative binomial model; LS Mean Ratio = 0.75, 95% CI 2-sided [0.61 to 0.92], Standard Error of Mean 0.08
Statistical Analysis 3: Comparison: Placebo vs Tanezumab 2.5 mg; Week 4: LS Mean was ratio of treatments. Analysis was performed using negative binomial model with model terms of baseline WOMAC Pain subscale score, baseline diary average pain score, index joint, Kellgren Lawrence grade, and treatment group; Test type: Superiority; p = 0.0003, Negative binomial model; LS Mean Ratio = 0.64, 95% CI 2-sided [0.51 to 0.82], Standard Error of Mean 0.08
Statistical Analysis 4: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 46, analysis 3]; Test type: Superiority; p = 0.0112, Negative binomial model; LS Mean Ratio = 0.74, 95% CI 2-sided [0.58 to 0.93], Standard Error of Mean 0.09
Statistical Analysis 5: Comparison: Placebo vs Tanezumab 2.5 mg; Week 8: LS Mean was ratio of treatments. Analysis was performed using negative binomial model with model terms of baseline WOMAC Pain subscale score, baseline diary average pain score, index joint, Kellgren Lawrence grade, and treatment group; Test type: Superiority; p = 0.0093, Negative binomial model; LS Mean Ratio = 0.72, 95% CI 2-sided [0.56 to 0.92], Standard Error of Mean 0.09
Statistical Analysis 6: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 46, analysis 5]; Test type: Superiority; p = 0.0237, Negative binomial model; LS Mean Ratio = 0.75, 95% CI 2-sided [0.59 to 0.96], Standard Error of Mean 0.09
Statistical Analysis 7: Comparison: Placebo vs Tanezumab 2.5 mg; Week 12: LS Mean was ratio of treatments. Analysis was performed using negative binomial model with model terms of baseline WOMAC Pain subscale score, baseline diary average pain score, index joint, Kellgren Lawrence grade, and treatment group; Test type: Superiority; p = 0.0374, Negative binomial model; LS Mean Ratio = 0.74, 95% CI 2-sided [0.56 to 0.98], Standard Error of Mean 0.11
Statistical Analysis 8: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 46, analysis 7]; Test type: Superiority; p = 0.0468, Negative binomial model; LS Mean Ratio = 0.75, 95% CI 2-sided [0.57 to 1.00], Standard Error of Mean 0.11
Statistical Analysis 9: Comparison: Placebo vs Tanezumab 2.5 mg; Week 16: LS Mean was ratio of treatments. Analysis was performed using negative binomial model with model terms of baseline WOMAC Pain subscale score, baseline diary average pain score, index joint, Kellgren Lawrence grade, and treatment group; Test type: Superiority; p = 0.0751, Negative binomial model; LS Mean Ratio = 0.78, 95% CI 2-sided [0.59 to 1.03], Standard Error of Mean 0.11
Statistical Analysis 10: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 46, analysis 9]; Test type: Superiority; p = 0.1305, Negative binomial model; LS Mean Ratio = 0.81, 95% CI 2-sided [0.61 to 1.06], Standard Error of Mean 0.11
Statistical Analysis 11: Comparison: Placebo vs Tanezumab 2.5 mg; Week 24: LS Mean was ratio of treatments. Analysis was performed using negative binomial model with model terms of baseline WOMAC Pain subscale score, baseline diary average pain score, index joint, Kellgren Lawrence grade, and treatment group; Test type: Superiority; p = 0.3057, Negative binomial model; LS Mean Ratio = 0.85, 95% CI 2-sided [0.63 to 1.16], Standard Error of Mean 0.13
Statistical Analysis 12: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 46, analysis 11]; Test type: Superiority; p = 0.2056, Negative binomial model; LS Mean Ratio = 0.82, 95% CI 2-sided [0.61 to 1.11], Standard Error of Mean 0.13

47. Secondary Outcome: Number of Days of Rescue Medication Used at Week 32
Description: In case of inadequate pain relief, after Week 24, acetaminophen/paracetamol up to 4000 mg per day up to 7 days in a week could be taken as rescue medication and use was reported weekly via diary. Number of days per week the participants used the rescue medication during the 4 weeks up to and including the particular study week were summarized.
Time Frame: Week 32
Population: The intent to treat population included all randomized participants who received at least one dose of subcutaneous study medication (either tanezumab or placebo). Here, 'Overall number of participants analyzed' signifies participants who took rescue medication.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg
Number analyzed (Participants) | 231 | 251 | 249
days | 1.8 (2.24) | 2.2 (2.34) | 2.0 (2.28)

48. Secondary Outcome: Amount of Rescue Medication Used at Weeks 2, 4, 8, 12, 16 and 24
Description: In case of inadequate pain relief, acetaminophen/paracetamol up to 4000 mg per day up to 5 days in a week could be taken as rescue medication. The total dosage of acetaminophen in milligrams used during the specified week were summarized.
Time Frame: Weeks 2, 4, 8, 12, 16 and 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: milligrams
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg
Number analyzed (Participants) | 282 | 283 | 284
milligrams
  Week 2 | 3690.6 (714.30) | 2283.4 (444.56) | 2703.4 (516.83)
  Week 4 | 3139.0 (707.35) | 1868.9 (396.26) | 2366.6 (529.63)
  Week 8 | 2940.9 (678.61) | 1902.4 (425.30) | 2269.4 (523.10)
  Week 12 | 2893.1 (749.38) | 1950.1 (495.07) | 1992.3 (509.28)
  Week 16 | 2627.1 (658.47) | 1864.2 (458.32) | 1897.6 (466.14)
  Week 24 | 2273.8 (625.84) | 1868.1 (482.13) | 1828.8 (491.51)
Statistical Analysis 1: Comparison: Placebo vs Tanezumab 2.5 mg; [analysis description as in outcome 46, analysis 2]; Test type: Superiority; p = 0.0441, Negative binomial model; LS Mean Ratio = 0.62, 95% CI 2-sided [0.39 to 0.99], Standard Error of Mean 0.15
Statistical Analysis 2: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 46, analysis 2]; Test type: Superiority; p = 0.1895, Negative binomial model; LS Mean Ratio = 0.73, 95% CI 2-sided [0.46 to 1.17], Standard Error of Mean 0.17
Statistical Analysis 3: Comparison: Placebo vs Tanezumab 2.5 mg; [analysis description as in outcome 46, analysis 3]; Test type: Superiority; p = 0.0567, Negative binomial model; LS Mean Ratio = 0.60, 95% CI 2-sided [0.35 to 1.01], Standard Error of Mean 0.16
Statistical Analysis 4: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 46, analysis 3]; Test type: Superiority; p = 0.2960, Negative binomial model; LS Mean Ratio = 0.75, 95% CI 2-sided [0.44 to 1.28], Standard Error of Mean 0.20
Statistical Analysis 5: Comparison: Placebo vs Tanezumab 2.5 mg; [analysis description as in outcome 46, analysis 5]; Test type: Superiority; p = 0.1215, Negative binomial model; LS Mean Ratio = 0.65, 95% CI 2-sided [0.37 to 1.12], Standard Error of Mean 0.18
Statistical Analysis 6: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 46, analysis 5]; Test type: Superiority; p = 0.3569, Negative binomial model; LS Mean Ratio = 0.77, 95% CI 2-sided [0.44 to 1.34], Standard Error of Mean 0.22
Statistical Analysis 7: Comparison: Placebo vs Tanezumab 2.5 mg; [analysis description as in outcome 46, analysis 7]; Test type: Superiority; p = 0.2096, Negative binomial model; LS Mean Ratio = 0.67, 95% CI 2-sided [0.36 to 1.25], Standard Error of Mean 0.21
Statistical Analysis 8: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 46, analysis 7]; Test type: Superiority; p = 0.2387, Negative binomial model; LS Mean Ratio = 0.69, 95% CI 2-sided [0.37 to 1.28], Standard Error of Mean 0.22
Statistical Analysis 9: Comparison: Placebo vs Tanezumab 2.5 mg; [analysis description as in outcome 46, analysis 9]; Test type: Superiority; p = 0.2627, Negative binomial model; LS Mean Ratio = 0.71, 95% CI 2-sided [0.39 to 1.29], Standard Error of Mean 0.22
Statistical Analysis 10: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 46, analysis 9]; Test type: Superiority; p = 0.2863, Negative binomial model; LS Mean Ratio = 0.72, 95% CI 2-sided [0.40 to 1.31], Standard Error of Mean 0.22
Statistical Analysis 11: Comparison: Placebo vs Tanezumab 2.5 mg; [analysis description as in outcome 46, analysis 11]; Test type: Superiority; p = 0.5560, Negative binomial model; LS Mean Ratio = 0.82, 95% CI 2-sided [0.43 to 1.58], Standard Error of Mean 0.27
Statistical Analysis 12: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 46, analysis 11]; Test type: Superiority; p = 0.5076, Negative binomial model; LS Mean Ratio = 0.80, 95% CI 2-sided [0.42 to 1.53], Standard Error of Mean 0.26

49. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs) up to End of Study
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent were events between first dose of study drug and up to week 48 that were absent before treatment or that worsened relative to pretreatment state. AEs included both serious and non-serious AEs.
Time Frame: Baseline up to Week 48
Population: The safety population was defined as all participants treated with tanezumab or placebo subcutaneously.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg
Number analyzed (Participants) | 282 | 283 | 284
Participants
  AEs | 178 | 184 | 198
  SAEs | 11 | 24 | 27

50. Secondary Outcome: Number of Participants With Treatment-Emergent Treatment-Related Adverse Events (AEs) and Serious Adverse Events (SAEs) up to End of Study
Description: Treatment-related AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent were events between first dose of study drug and up to week 48 that were absent before treatment or that worsened relative to pre-treatment state. Relatedness to study drug was assessed by the investigator.
Time Frame: Baseline up to Week 48
Population: The safety population was defined as all participants treated with tanezumab or placebo subcutaneously.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg
Number analyzed (Participants) | 282 | 283 | 284
Participants
  AEs | 46 | 52 | 59
  SAEs | 1 | 0 | 3

51. Secondary Outcome: Number of Participants With Laboratory Test Abnormalities With Regard to Normal Baseline
Description: Primary Abnormality criteria: HGB, hematocrit, RBC count <0.8* lower limit of normal(LLN); Ery. mean corpuscular volume/hemoglobin/ HGB concentration, RBCs distribution width <0.9*LLN, >1.1*upper limit of normal(ULN); platelets <0.5*LLN,>1.75*ULN; WBC count<0.6*LLN, >1.5*ULN; Lymphocytes,Leukocytes,Neutrophils <0.8*LLN, >1.2*ULN; Basophils,Eosinophils,Monocytes>1.2*ULN; Prothrombin time/Intl. normalized ratio>1.1*ULN; total bilirubin>1.5*ULN; aspartate aminotransferase,alanine aminotransferase,gamma GT,LDH,alkaline phosphatase >3.0*ULN; total protein; albumin<0.8*LLN, >1.2*ULN; blood urea nitrogen,creatinine,Cholesterol,triglycerides >1.3*ULN; Urate>1.2*ULN; sodium<0.95*LLN,>1.05*ULN; potassium,chloride,calcium,magnesium,bicarbonate <0.9*LLN, >1.1*ULN; phosphate<0.8*LLN, >1.2*ULN; glucose<0.6*LLN, >1.5*ULN; HGB A1C >1.3*ULN; creatine kinase>2.0*ULN, specific gravity<1.003, >1.030; pH<4.5, >8; Urine Glucose, protein,HGB,bilirubin >=1; Ketones>=1;Urine erythrocytes,Leukocytes>=20.
Time Frame: Baseline up to Week 48
Population: The safety population was defined as all participants treated with tanezumab or placebo subcutaneously. Here 'Overall number of participants analyzed' signifies participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg
Number analyzed (Participants) | 265 | 271 | 274
Participants | 32 | 34 | 34

52. Secondary Outcome: Number of Participants With Laboratory Test Abnormalities With Regard to Abnormal Baseline
Description: Primary Abnormality criteria: hemoglobin; hematocrit; RBC count < 0.8*LLN; Ery. mean corpuscular volume/ hemoglobin/ HGB concentration, erythrocytes distribution width <0.9*LLN, >1.1*ULN; platelets <0.5*LLN,>1.75*upper limit of normal (ULN); white blood cell count<0.6*LLN, >1.5*ULN; Lymphocytes, Leukocytes, Neutrophils <0.8*LLN, >1.2*ULN; Basophils, Eosinophils, Monocytes >1.2*ULN; total bilirubin>1.5*ULN; aspartate aminotransferase, alanine aminotransferase, gamma GT,LDH, alkaline phosphatase >3.0*ULN; total protein; albumin<0.8*LLN, >1.2*ULN; blood urea nitrogen, creatinine, Cholesterol, triglycerides >1.3*ULN; Urate >1.2*ULN; sodium <0.95*LLN,>1.05*ULN; potassium, chloride, calcium, magnesium, bicarbonate <0.9*LLN, >1.1*ULN; phosphate <0.8*LLN, >1.2*ULN; glucose <0.6*LLN, >1.5*ULN; Hemoglobin A1C >1.3*ULN; creatine kinase >2.0*ULN; Nitrite >=1.
Time Frame: Baseline up to Week 48
Population: The safety population was defined as all participants treated with tanezumab or placebo subcutaneously. Here "Overall number of participants analysed" signifies participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg
Number analyzed (Participants) | 205 | 215 | 207
Participants | 19 | 26 | 22

53. Secondary Outcome: Change From Baseline in Blood Pressure (BP) at Weeks 2, 4, 8, 12, 16, 24, 32 and 48
Description: Measurement of BP included sitting systolic blood pressure (SBP) and diastolic blood pressure (DBP).
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, 24, 32 and 48
Population: The safety population was defined as all participants treated with tanezumab or placebo subcutaneously. Here, 'Number analyzed' = Participants evaluable for this outcome measure for specified categories.
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg
Number analyzed (Participants) | 282 | 283 | 284
millimeters of mercury (mmHg)
  SBP: Baseline | 132.0 (13.54) | 132.7 (12.59) | 132.0 (12.12)
  SBP:Change at Week 2: number analyzed (Participants) | 276 | 278 | 278
  SBP:Change at Week 2 | -1.0 (10.26) | -2.0 (11.24) | -2.4 (11.24)
  SBP:Change at Week 4: number analyzed (Participants) | 272 | 280 | 278
  SBP:Change at Week 4 | -0.3 (11.09) | -2.0 (10.94) | -2.4 (11.52)
  SBP:Change at Week 8: number analyzed (Participants) | 265 | 275 | 275
  SBP:Change at Week 8 | -0.8 (10.89) | -2.1 (10.63) | -2.5 (12.07)
  SBP:Change at Week 12: number analyzed (Participants) | 255 | 274 | 271
  SBP:Change at Week 12 | -1.2 (11.38) | -1.8 (11.53) | -2.8 (11.64)
  SBP:Change at Week 16: number analyzed (Participants) | 242 | 265 | 265
  SBP:Change at Week 16 | -0.4 (12.18) | -1.6 (12.92) | -2.3 (11.63)
  SBP:Change at Week 24: number analyzed (Participants) | 236 | 255 | 254
  SBP:Change at Week 24 | -1.5 (11.47) | -2.0 (12.55) | -2.5 (12.11)
  SBP:Change at Week 32: number analyzed (Participants) | 228 | 251 | 139
  SBP:Change at Week 32 | -2.1 (12.61) | -1.8 (12.40) | -1.0 (12.55)
  SBP:Change at Week 48: number analyzed (Participants) | 220 | 242 | 229
  SBP:Change at Week 48 | -0.7 (10.38) | -1.7 (11.60) | -1.8 (11.34)
  DBP: Baseline | 79.7 (8.28) | 79.3 (8.45) | 79.5 (8.10)
  DBP:Change at Week 2: number analyzed (Participants) | 276 | 278 | 278
  DBP:Change at Week 2 | -0.4 (6.81) | -1.7 (7.18) | -1.7 (7.33)
  DBP:Change at Week 4: number analyzed (Participants) | 272 | 280 | 278
  DBP:Change at Week 4 | -0.6 (7.06) | -1.7 (7.35) | -1.8 (7.85)
  DBP:Change at Week 8: number analyzed (Participants) | 265 | 275 | 275
  DBP:Change at Week 8 | -0.1 (7.59) | -1.0 (7.11) | -1.7 (7.65)
  DBP:Change at Week 12: number analyzed (Participants) | 255 | 274 | 271
  DBP:Change at Week 12 | -1.0 (7.44) | -1.3 (7.79) | -2.8 (7.94)
  DBP:Change at Week 16: number analyzed (Participants) | 242 | 265 | 265
  DBP:Change at Week 16 | -0.7 (7.85) | -0.6 (8.26) | -1.8 (7.90)
  DBP:Change at Week 24: number analyzed (Participants) | 236 | 255 | 254
  DBP:Change at Week 24 | -0.1 (7.81) | -0.2 (8.42) | -2.0 (7.90)
  DBP:Change at Week 32: number analyzed (Participants) | 228 | 251 | 239
  DBP:Change at Week 32 | -1.2 (8.52) | -0.7 (8.06) | -1.5 (8.64)
  DBP:Change at Week 48 | -0.6 (7.22) | -0.7 (8.32) | -0.9 (8.17)

54. Secondary Outcome: Change From Baseline in Heart Rate at Weeks 2, 4, 8, 12, 16, 24, 32 and 48
Description: Heart rate was measured at sitting position.
Time Frame: Baseline, Weeks 2, 4, 8, 12,16, 24, 32 and 48
Population: The safety population was defined as all participants treated with tanezumab or placebo subcutaneously. Here, 'Number analyzed' = Participants evaluable for this outcome measure for specified time points.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg
Number analyzed (Participants) | 282 | 283 | 284
beats per minute
  Baseline: number analyzed (Participants) | 282 | 283 | 283
  Baseline | 71.1 (8.45) | 70.4 (8.62) | 70.8 (8.33)
  Change at Week 2: number analyzed (Participants) | 275 | 277 | 277
  Change at Week 2 | 0.2 (7.26) | 1.2 (7.25) | 0.2 (8.45)
  Change at Week 4: number analyzed (Participants) | 272 | 280 | 277
  Change at Week 4 | 0.8 (7.92) | 0.9 (7.91) | -0.1 (7.99)
  Change at Week 8: number analyzed (Participants) | 265 | 275 | 274
  Change at Week 8 | 0.5 (7.61) | -0.3 (8.08) | -0.9 (7.54)
  Change at Week 12: number analyzed (Participants) | 255 | 274 | 270
  Change at Week 12 | 0.9 (8.14) | 1.6 (8.28) | 0.5 (8.39)
  Change at Week 16: number analyzed (Participants) | 242 | 265 | 264
  Change at Week 16 | -0.3 (8.13) | -0.4 (8.01) | -0.0 (8.12)
  Change at Week 24: number analyzed (Participants) | 236 | 255 | 253
  Change at Week 24 | -0.5 (8.56) | 0.5 (8.77) | 0.4 (8.86)
  Change at Week 32: number analyzed (Participants) | 228 | 251 | 238
  Change at Week 32 | 1.1 (8.51) | 0.8 (8.19) | 0.6 (9.40)
  Change at Week 48: number analyzed (Participants) | 220 | 242 | 228
  Change at Week 48 | -0.2 (8.13) | 1.4 (9.87) | 0.6 (10.01)

55. Secondary Outcome: Change From Baseline in Electrocardiogram (ECG) Parameters at Weeks 24 and 48
Description: A 12-lead ECG was recorded after participants had rested for at least 5 minutes in the supine position in a quiet environment. All standard intervals (PR, QRS, QT, QTcF, QTcB, QTcF, RR intervals) were collected.
Time Frame: Baseline, Weeks 24 and 48
Population: as for outcome 53
Measure: Mean (Standard Deviation); unit: millisecond
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg
Number analyzed (Participants) | 282 | 283 | 284
millisecond
  RR Interval: Baseline | 923.9 (124.86) | 923.6 (139.69) | 928.3 (126.14)
  RR Interval:Change at Week 24: number analyzed (Participants) | 236 | 254 | 252
  RR Interval:Change at Week 24 | -3.2 (108.30) | -14.6 (119.62) | -16.1 (124.65)
  RR Interval:Change at Week 48: number analyzed (Participants) | 216 | 238 | 224
  RR Interval:Change at Week 48 | -19.0 (118.49) | -16.0 (112.48) | -26.7 (125.81)
  PR Interval: Baseline: number analyzed (Participants) | 276 | 278 | 277
  PR Interval: Baseline | 168.7 (23.95) | 165.6 (21.92) | 168.0 (24.54)
  PR Interval:Change at Week 24: number analyzed (Participants) | 229 | 248 | 240
  PR Interval:Change at Week 24 | 0.1 (14.07) | 0.5 (13.38) | 2.0 (15.43)
  PR Interval:Change at Week 48: number analyzed (Participants) | 209 | 231 | 213
  PR Interval:Change at Week 48 | 1.3 (13.64) | -1.1 (14.38) | -0.4 (14.23)
  QRS Interval: Baseline | 95.7 (12.69) | 95.6 (14.05) | 95.8 (14.48)
  QRS Interval:Change at Week 24: number analyzed (Participants) | 236 | 254 | 252
  QRS Interval:Change at Week 24 | -0.2 (7.22) | 0.2 (7.57) | 0.0 (7.34)
  QRS Interval:Change at Week 48: number analyzed (Participants) | 216 | 238 | 224
  QRS Interval:Change at Week 48 | -0.2 (8.04) | 0.2 (8.33) | 0.8 (8.73)
  QT Interval: Baseline: number analyzed (Participants) | 281 | 282 | 283
  QT Interval: Baseline | 402.0 (28.45) | 403.1 (29.92) | 405.6 (26.84)
  QT Interval:Change at Week 24: number analyzed (Participants) | 234 | 252 | 251
  QT Interval:Change at Week 24 | -2.2 (22.65) | -3.1 (21.78) | -3.8 (25.84)
  QT Interval:Change at Week 48: number analyzed (Participants) | 215 | 237 | 222
  QT Interval:Change at Week 48 | -2.5 (23.27) | -1.6 (24.40) | -4.9 (24.06)
  QTCB Interval: Baseline: number analyzed (Participants) | 281 | 282 | 283
  QTCB Interval: Baseline | 419.8 (22.32) | 421.3 (20.78) | 422.5 (20.57)
  QTCB Interval:Change at Week 24: number analyzed (Participants) | 234 | 252 | 251
  QTCB Interval:Change at Week 24 | -1.5 (17.56) | 0.2 (18.47) | 0.0 (16.26)
  QTCB Interval:Change at Week 48: number analyzed (Participants) | 215 | 237 | 222
  QTCB Interval:Change at Week 48 | 1.5 (16.45) | 1.7 (16.70) | 1.8 (16.80)
  QTCF Interval: Baseline: number analyzed (Participants) | 281 | 282 | 283
  QTCF Interval: Baseline | 413.6 (20.70) | 414.9 (19.23) | 416.6 (18.61)
  QTCF Interval:Change at Week 24: number analyzed (Participants) | 234 | 252 | 251
  QTCF Interval:Change at Week 24 | -1.7 (15.72) | -1.0 (14.94) | -1.3 (15.05)
  QTCF Interval:Change at Week 48: number analyzed (Participants) | 215 | 237 | 222
  QTCF Interval:Change at Week 48 | 0.2 (14.50) | 0.5 (15.58) | -0.5 (13.96)

56. Secondary Outcome: Change From Baseline in Heart Rate (as Assessed by ECG) at Weeks 24 and 48
Description: Heart rate was measured at sitting position.
Time Frame: Baseline, Weeks 24 and 48
Population: The safety population was defined as all participants treated with tanezumab or placebo subcutaneously. Here, 'Number analyzed' = Participants evaluable for this outcome measure at specified time points.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg
Number analyzed (Participants) | 282 | 283 | 284
beats per minute
  Baseline | 66.2 (9.28) | 66.5 (10.69) | 65.9 (9.22)
  change at Week 24: number analyzed (Participants) | 236 | 254 | 252
  change at Week 24 | 0.3 (8.05) | 0.9 (9.15) | 1.4 (10.19)
  Change at Week 48: number analyzed (Participants) | 216 | 238 | 224
  Change at Week 48 | 1.4 (8.59) | 1.1 (8.98) | 2.3 (10.44)

57. Secondary Outcome: Percentage of Participants With Adjudicated Joint Safety Outcomes
Description: Incidence of participants with any of the joint safety adjudication outcomes of primary osteonecrosis, rapidly progressive OA (type 1 and type 2), subchondral insufficiency fracture (or SPONK), or pathological fracture.
Time Frame: Baseline up to Week 48
Population: The safety population was defined as all participants treated with tanezumab or placebo subcutaneously. Here, 'Overall number of participants analyzed' signifies participants analyzed by adjudication committee.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg
Number analyzed (Participants) | 19 | 27 | 33
percentage of participants
  Composite Joint Safety Endpoint | 0 [0.0 to 1.3] | 1.8 [0.6 to 4.1] | 3.2 [1.5 to 5.9]
  Rapidly Progressive OA | 0 [0.0 to 1.3] | 1.4 [0.4 to 3.6] | 2.8 [1.2 to 5.5]
  Rapidly Progressive OA type 1 | 0 [0.0 to 1.3] | 1.1 [0.2 to 3.1] | 1.8 [0.6 to 4.1]
  Rapidly Progressive OA type 2 | 0 [0.0 to 1.3] | 0.4 [0.0 to 2.0] | 1.1 [0.2 to 3.1]
  Primary Osteonecrosis | 0 [0.0 to 1.3] | 0 [0.0 to 1.3] | 0.4 [0.0 to 1.9]
  Pathological Fracture | 0 [0.0 to 1.3] | 0 [0.0 to 1.3] | 0 [0.0 to 1.3]
  Subchondral Insufficiency Fracture | 0 [0.0 to 1.3] | 0.4 [0.0 to 2.0] | 0 [0.0 to 1.3]

58. Secondary Outcome: Percentage of Participants With Total Joint Replacements
Description: Percentage of participants who underwent at least one total knee, hip or shoulder joint replacement surgery.
Time Frame: Baseline up to Week 48
Population: The safety population was defined as all participants treated with tanezumab or placebo subcutaneously.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg
Number analyzed (Participants) | 282 | 283 | 284
percentage of participants | 6.7 [4.1 to 10.3] | 7.8 [4.9 to 11.5] | 7.0 [4.4 to 10.7]

59. Secondary Outcome: Number of Participants With Confirmed Orthostatic Hypotension
Description: Orthostatic hypotension was defined as postural change (supine to standing) that met the following criteria: For systolic BP <=150 mmHg (mean supine): Reduction in systolic BP>=20 mmHg or reduction in diastolic BP>=10 mmHg at the 1 and/or 3 minute standing BP measurements. For systolic BP >150 mmHg (mean supine): Reduction in systolic BP>=30 mmHg or reduction in diastolic BP>=15 mmHg at the 1 and/or 3 minute standing BP measurements. If the 1 minute or 3 minute standing BP in a sequence met the orthostatic hypotension criteria, then that sequence was considered positive. If 2 of 2 or 2 of 3 sequences were positive, then orthostatic hypotension was considered confirmed.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, 24, 32 and 48
Population: The safety population was defined as all participants treated with tanezumab or placebo subcutaneously. Here, 'Overall number of participants analyzed' signifies participants analyzed for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg
Number analyzed (Participants) | 221 | 242 | 228
Participants
  Baseline | 0 | 1 | 0
  Week 2 | 0 | 0 | 0
  Week 4 | 0 | 0 | 1
  Week 8 | 0 | 0 | 1
  Week 12 | 0 | 0 | 0
  Week 16 | 0 | 0 | 1
  Week 24 | 0 | 0 | 0
  Week 32 | 0 | 0 | 0
  Week 48 | 0 | 1 | 1

60. Secondary Outcome: Change From Baseline in Survey of Autonomic Symptom (SAS) Scores at Week 24
Description: The SAS is a 12 item (11 for females) questionnaire, from which the total number of symptoms (0-12 for males and 0-11 for females) is calculated. Each positive symptom is rated from 1 (not at all) to 5 (a lot). The total impact score was the sum of all symptom rating scores, with 0 assigned where the participant did not have the particular symptom. The range for the total impact score is 0-60 for males and 0-55 for females, higher scores indicating higher impact.
Time Frame: Baseline, Week 24
Population: as for outcome 56
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg
Number analyzed (Participants) | 282 | 283 | 284
units on a scale
  Number of symptoms reported: Baseline: number analyzed (Participants) | 280 | 282 | 283
  Number of symptoms reported: Baseline | 0.55 (0.85) | 0.53 (0.85) | 0.55 (0.83)
  Number of symptoms reported: Change at Week 24: number analyzed (Participants) | 232 | 255 | 254
  Number of symptoms reported: Change at Week 24 | 0.03 (1.07) | 0.15 (1.18) | 0.18 (1.22)
  Total Symptom Impact Score: Baseline: number analyzed (Participants) | 280 | 282 | 283
  Total Symptom Impact Score: Baseline | 1.14 (1.94) | 1.11 (1.79) | 1.20 (1.99)
  Total Symptom Impact Score: Change at Week 24: number analyzed (Participants) | 232 | 255 | 254
  Total Symptom Impact Score: Change at Week 24 | 0.32 (2.92) | 0.53 (3.23) | 0.56 (3.11)

61. Secondary Outcome: Change From Baseline in Neuropathy Impairment Score (NIS) at Weeks 2, 4, 8, 12, 16, 24, 32 and 48
Description: NIS is a standardized instrument used to evaluate participant for signs of peripheral neuropathy. NIS is the sum of scores of 37 items, from both the left and right side, where 24 items scored from 0 (normal) to 4 (paralysis), higher score indicated higher abnormality/impairment and 13 items scored from 0 (normal), 1 (decreased) and 2 (absent), higher score indicated higher impairment. NIS possible overall score ranged from 0 (no impairment) to 244 (maximum impairment), higher scores indicated increased impairment.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, 24, 32 and 48
Population: as for outcome 56
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg
Number analyzed (Participants) | 282 | 283 | 284
units on a scale
  Baseline | 1.35 (2.85) | 1.35 (3.72) | 1.48 (3.11)
  Change at Week 2: number analyzed (Participants) | 280 | 280 | 276
  Change at Week 2 | 0.03 (0.92) | -0.09 (0.68) | -0.21 (1.14)
  Change at Week 4: number analyzed (Participants) | 282 | 282 | 281
  Change at Week 4 | 0.01 (1.16) | 0.00 (1.31) | -0.32 (1.24)
  Change at Week 8: number analyzed (Participants) | 282 | 282 | 283
  Change at Week 8 | -0.11 (1.42) | -0.13 (1.20) | -0.41 (1.56)
  Change at Week 12: number analyzed (Participants) | 282 | 282 | 283
  Change at Week 12 | -0.12 (1.38) | -0.03 (1.50) | -0.39 (1.59)
  Change at Week 16: number analyzed (Participants) | 282 | 282 | 283
  Change at Week 16 | -0.17 (1.59) | -0.03 (1.72) | -0.46 (1.53)
  Change at Week 24: number analyzed (Participants) | 282 | 282 | 283
  Change at Week 24 | -0.20 (1.51) | -0.01 (1.85) | -0.47 (1.58)
  Change at Week 32: number analyzed (Participants) | 282 | 282 | 283
  Change at Week 32 | -0.23 (1.69) | 0.00 (1.75) | -0.41 (1.57)
  Change at Week 48: number analyzed (Participants) | 282 | 282 | 283
  Change at Week 48 | -0.22 (1.67) | 0.01 (1.91) | -0.43 (1.57)

62. Secondary Outcome: Number of Participants With Anti Tanezumab Antibodies
Description: Human serum ADA samples were analyzed for the presence or absence of anti-tanezumab antibodies by using a semi quantitative enzyme linked immunosorbent assay (ELISA). Participants listed as having anti-tanezumab antibodies had ADA titer level >=3.32. Less than 3.32 was considered below the limit of quantitation.
Time Frame: Baseline, Weeks 8,16, 24, 32 and 48
Population: as for outcome 56
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg
Number analyzed (Participants) | 282 | 283 | 284
Participants
  Baseline: number analyzed (Participants) | 281 | 282 | 281
  Baseline | 24 | 26 | 36
  Week 8: number analyzed (Participants) | 261 | 275 | 275
  Week 8 | 24 | 27 | 41
  Week 16: number analyzed (Participants) | 242 | 263 | 265
  Week 16 | 25 | 34 | 48
  Week 24: number analyzed (Participants) | 233 | 253 | 251
  Week 24 | 19 | 39 | 49
  Week 32: number analyzed (Participants) | 224 | 247 | 236
  Week 32 | 19 | 38 | 42
  Week 48: number analyzed (Participants) | 216 | 242 | 227
  Week 48 | 18 | 32 | 31

ADVERSE EVENTS:
Time Frame: Baseline up to Week 24
Description: Same event may appear as AE and serious AE, what is presented are distinct events. Event may be categorized as serious in 1 participant and as nonserious in another participant or 1 participant may have experienced both serious and nonserious event during study. One death was accounted as lost to follow-up in participant flow as the death was not confirmed by family nor a doctor, but a follow-up letter to the participant was returned with a note on the envelope that the addressee died.
Arm/Group | Placebo | Tanezumab 2.5 mg | Tanezumab 5 mg
All-Cause Mortality (participants affected / at risk) | 0/282 | 1/283 | 2/284
Serious Adverse Events (participants affected / at risk) | 3/282 | 8/283 | 9/284
Other Adverse Events (participants affected / at risk) | 77/282 | 73/283 | 60/284
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=282) | Tanezumab 2.5 mg (N=283) | Tanezumab 5 mg (N=284)
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 1
Coronary artery stenosis (Cardiac disorders) | 0 | 1 | 0
Cataract (Eye disorders) | 1 | 0 | 0
Ocular vascular disorder (Eye disorders) | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1
Hepatitis (Hepatobiliary disorders) | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 1
Nerve injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Nerve root injury lumbar (Injury, poisoning and procedural complications) | 0 | 1 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0
Lymphatic fistula (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=282) | Tanezumab 2.5 mg (N=283) | Tanezumab 5 mg (N=284)
Nasopharyngitis (Infections and infestations) | 25 | 31 | 21
Arthralgia (Musculoskeletal and connective tissue disorders) | 34 | 27 | 22
Back pain (Musculoskeletal and connective tissue disorders) | 15 | 16 | 17
Headache (Nervous system disorders) | 18 | 15 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2016-02-10): https://cdn.clinicaltrials.gov/large-docs/86/NCT02709486/Prot_000.pdf
  • Statistical Analysis Plan (2018-12-21): https://cdn.clinicaltrials.gov/large-docs/86/NCT02709486/SAP_001.pdf